CLINICAL TRIAL: NCT03945825
Title: A Phase I Study to Assess the Safety, Reactogenicity and Immunogenicity of Two Quadrivalent Seasonal Influenza Vaccines (Fluzone(R) or Flublok(R)) With or Without One of Two Adjuvants (AF03 or Advax-CpG55.2) in Healthy Adults 18-45 Years of Age
Brief Title: Flublok or Fluzone With Advax-CpG55.2 or AF03
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 18-0011; HHSN272201300018I
Record Dates: First submitted 2019-05-09; First posted 2019-05-10 (Actual); Results first posted 2022-01-03 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2021-02-19

CONDITIONS: Influenza; Influenza Immunisation
Keywords: Immunogenicity; Influenza; Influenza Vaccine; Phase 1; Quadrivalent; Safety
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group 1 (Experimental): 0.5 mL of 2018/2019 Fluzone QIV intramuscular injection on Day 1 and 0.5 ml of 2019/2020 Fluzone QIV intramuscular injection on Day 90, n=40
  Interventions: Biological: Influenza Virus Quadrivalent Inactivated Vaccine
- Group 2 (Experimental): 0.5 mL of 2018/2019 Fluzone QIV + 0.25 mL of AF03 (admixed with vaccine) intramuscular injection on Day 1 and 0.5 ml of 2019/2020 Fluzone QIV intramuscular injection on Day 90, n=40
  Interventions: Drug: AF03; Biological: Influenza Virus Quadrivalent Inactivated Vaccine
- Group 3 (Experimental): 0.5 mL of 2018/2019 Fluzone QIV + 0.5 mL of Delta Inulin-CpG55.2 (admixed with vaccine) intramuscular injection on Day 1 and 0.5 2019/2020 of Fluzone QIV intramuscular injection on Day 90, n=40
  Interventions: Biological: Delta Inulin-CpG55.2; Biological: Influenza Virus Quadrivalent Inactivated Vaccine
- Group 4 (Experimental): 0.5 mL of 2018/2019 Flublok QIV intramuscular injection on Day 1 and 0.5 ml of 2019/2020 Flublok QIV intramuscular injection on Day 90, n=40
  Interventions: Biological: Quadrivalent Recombinant Seasonal Influenza Vaccine
- Group 5 (Experimental): 0.5 mL of 2018/2019 Flublok QIV + 0.25 mL AF03 (admixed with vaccine) intramuscular injection on Day 1 and 0.5 ml of 2019/2020 Flublok QIV intramuscular injection on Day 90, n=40
  Interventions: Drug: AF03; Biological: Quadrivalent Recombinant Seasonal Influenza Vaccine
- Group 6 (Experimental): 0.5 mL of 2018/2019 Flublok QIV + 0.5 mL of Delta Inulin-CpG55.2 (admixed with vaccine) intramuscular injection on Day 1 and 0.5 ml of 2019/2020 Flublok QIV intramuscular injection on Day 90, n=40
  Interventions: Biological: Delta Inulin-CpG55.2; Biological: Quadrivalent Recombinant Seasonal Influenza Vaccine

INTERVENTIONS:
Drug: AF03 — A squalene-in-PBS emulsion stabilized by nonionic surfactants, sorbitan oleate and macrogol cetostearyl ether
  Arms: Group 2; Group 5
Biological: Delta Inulin-CpG55.2 — A combination adjuvant supplied as two separate components, Delta Inulin (Sypharma Pty Ltd.) and CpG55.2 (Nikko Denka Avecia and Sypharma Pty Ltd)
  Arms: Group 3; Group 6
Biological: Influenza Virus Quadrivalent Inactivated Vaccine — 2018/2019 Fluzone QIV and 2019/2020 Fluzone QIV vaccines will be given with 90 days interval
  Arms: Group 1; Group 2; Group 3
Biological: Quadrivalent Recombinant Seasonal Influenza Vaccine — 2018/2019 Flublok QIV and 2019/2020 Flublok QIV vaccines will be given with 90 days interval
  Arms: Group 4; Group 5; Group 6

SUMMARY:
This is a Phase I, randomized, double blinded, clinical trial in up to 240 males and non-pregnant females, 18-45 years of age, inclusive, who are in good health and meet all eligibility criteria. This clinical trial is designed to assess the safety, reactogenicity and immunogenicity of either the 2018/2019 seasonal Fluzone or Flublok Quadrivalent Influenza Vaccine (QIV) manufactured by Sanofi Pasteur (SP) given without adjuvant or with one of two adjuvant formulations, AF03 or Advax-CpG55.2. Eight Vaccine and Treatment Evaluation Unit (VTEU) sites will be included in the study. Study duration is approximately 18 months, and subject participation duration is 12 months. The primary objectives of this study are: 1) to assess the safety and reactogenicity of 2018/2019 Fluzone and Flublok with and without AF03 or Advax-CpG55.2 adjuvant; 2) to assess the serum hemagglutination inhibition (HAI) antibody responses against 2018/2019 QIV strains from baseline (Day 1) to approximately Day 29 after receipt of 2018/2019 Fluzone and Flublok with and without AF03 or Advax-CpG55.2 adjuvant; 3) to assess the serum neuraminidase inhibition antibody (NAI) responses by enzyme-linked lectin assay (ELLA) against NA antigens in the 2018/2019 QIV from baseline (Day 1) to approximately Day 29 after receipt of 2018/2019 Fluzone and Flublok with and without AF03 or Advax-CpG55.2 adjuvant; 4) to assess the influenza neutralizing (Neut) antibody titer responses against 2018/2019 QIV strains from baseline (Day 1) to approximately Day 29 after receipt of 2018/2019 Fluzone and Flublok with and without AF03 or Advax- CpG55.2 adjuvant.

DETAILED DESCRIPTION:
This is a Phase I, randomized, double blinded, clinical trial in up to 240 males and non-pregnant females, 18-45 years of age, inclusive, who are in good health and meet all eligibility criteria. This clinical trial is designed to assess the safety, reactogenicity and immunogenicity of either the 2018/2019 seasonal Fluzone or Flublok Quadrivalent Influenza Vaccine (QIV) manufactured by Sanofi Pasteur (SP) given without adjuvant or with one of two adjuvant formulations, AF03 or Advax-CpG55.2. Subjects will be stratified by prior receipt of licensed, seasonal influenza vaccine (defined as receipt of at least one of the 2017/2018 and/or 2018/2019 influenza vaccines) and will be randomly assigned to 1 of 6 treatment arms to receive a single dose of one of the two seasonal 2018/2019 QIV vaccine formulations with or without one of the two adjuvants (Day 1). On approximately Day 90, each subject will receive a single dose of the seasonal 2019/2020 QIV. Groups 1, 2 and 3 will receive 2019/2020 Fluzone QIV and Groups 4, 5 and 6 will receive 2019/2020 Flublok QIV. Eight Vaccine and Treatment Evaluation Unit (VTEU) sites will be included in the study. Study duration is approximately 18 months, and subject participation duration is 12 months. The primary objectives of this study are: 1) to assess the safety and reactogenicity of 2018/2019 Fluzone and Flublok with and without AF03 or Advax-CpG55.2 adjuvant; 2) to assess the serum hemagglutination inhibition (HAI) antibody responses against 2018/2019 QIV strains from baseline (Day 1) to approximately Day 29 after receipt of 2018/2019 Fluzone and Flublok with and without AF03 or Advax-CpG55.2 adjuvant; 3) to assess the serum neuraminidase inhibition antibody (NAI) responses by enzyme-linked lectin assay (ELLA) against NA antigens in the 2018/2019 QIV from baseline (Day 1) to approximately Day 29 after receipt of 2018/2019 Fluzone and Flublok with and without AF03 or Advax-CpG55.2 adjuvant; 4) to assess the influenza neutralizing (Neut) antibody titer responses against 2018/2019 QIV strains from baseline (Day 1) to approximately Day 29 after receipt of 2018/2019 Fluzone and Flublok with and without AF03 or Advax- CpG55.2 adjuvant. The secondary objectives of this study are: 1) to assess protocol specified adverse events of special interest (AESI), medically-attended adverse events (MAAEs), including new-onset chronic medical conditions (NOCMCs) and potentially immune-mediated medical conditions (PIMMCs) that occur after receipt of study product; 2) to assess the HAI, Neut and NAI ELLA responses to the 2019/2020 QIV strains prior to (Day 1) and approximately 28 days after vaccination with the 2019/2020 QIV in all study groups; 3) to assess the HAI antibody responses against heterologous influenza A/H1 and H3 strains from baseline (Day 1) to approximately Days 8, 29, 57, 90 and 118 after receipt of 2018/2019 Fluzone or Flublok with and without AF03 or Advax-CpG55.2 adjuvant; 4) to assess NAI ELLA responses against heterologous N1 and N2 NA antigens from baseline (Day 1) to approximately Days 8, 29, 57, 90 and 118 after administration of 2018/2019 Fluzone with and without AF03 or Advax-CpG55.2 adjuvant; 5) to assess the influenza neutralizing (Neut) antibody titer responses against heterologous influenza A/H1 and H3 strains from baseline (Day 1) to approximately Days 8, 29, 57, 90 and 118 after administration of 2018/2019 Fluzone and Flublok with and without AF03 or Advax-CpG55.2 adjuvant; 6) to assess the longitudinal kinetics and durability of the HAI, NAI, and Neut responses against the 2018/2019 QIV strains on approximately Days 8, 57, 90 and 118 following receipt of the 2018/2019 Fluzone and Flublok with and without AF03 or Advax-CpG55.2 adjuvant.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to initiation of any study procedures.
2. Are able to understand and comply with planned study procedures and be available for all study visits.
3. Must agree to the collection of venous blood per protocol.
4. Are males or non-pregnant females, 18 to 45 years of age, inclusive at time of enrollment.
5. Are in good health*. *As determined by medical history and physical examination to evaluate acute or currently ongoing chronic medical or psychiatric diagnoses or conditions, defined as those that have been present for at least 90 days, which would affect the assessment of the safety of subjects or the immunogenicity of study vaccinations. Chronic medical diagnoses or conditions should be stable for the last 60 days (no hospitalizations, emergency room or urgent care for condition, or invasive medical procedure and no adverse symptoms that need medical intervention such as medication change/supplemental oxygen). This includes no change in chronic prescription medication, dose or in the 60 days prior to enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site PI or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening or treatment of continued symptoms of medical diagnosis or condition. Note: Low dose topical, corticosteroids as outlined in the Subject Exclusion Criteria as well as herbals, vitamins and supplements are permitted.
6. Oral temperature is less than 100.0 degrees Fahrenheit.
7. Pulse is 47 to 100 beats per minute, inclusive.
8. Systolic blood pressure is 85 to 140 mmHg, inclusive.
9. Diastolic blood pressure is 55 to 90 mmHg, inclusive.
10. Screening laboratories (Erythrocyte Sedimentation Rate (ESR), White Blood Cells (WBC), Hemoglobin (Hgb), Platelets (PLTs), Alanine Aminotransferase (ALT), Total Bilirubin (T. Bili), Aspartate Aminotransferase (AST), Gamma-glutamyl Transferase (GGT), Alkaline Phosphatase (ALP) serum lipase, serum amylase and Creatinine (Cr)) are within acceptable parameters*.

    *ESR must be below 30 mm/hr; WBC >3.90 K/MM3 and <10.60 K/MM3; Hgb >/= 11.5 g/dl (women) or >/= 12.5 g/dl (men); PLTs (EDTA) 140-415 K/MM3; PLTs (Citrate) 125-325 K/MM3 ALT </= 43 U/L (women) or </= 60 U/L (men); T Bili </=1.20 mg/dl; Cr < 1.1 mg/dl (women) or < 1.4 mg/dl (men); AST 10-36 U/L (women) or 10-43 U/L (men); GGT 5--32 U/L (women) or 10-49 U/L (men); ALP 30-115 U/L (women) or 43-115 U/L (men); lipase 13-60 U/L; amylase (Total) 35-121 U/L, for subjects to qualify for randomization and vaccination.
11. Women of childbearing potential* must use an acceptable contraception method** from at least 30 days before the first study vaccination until 60 days after the second study vaccination.

    *Not sterilized via bilateral oophorectomy, tubal ligation/ salpingectomy, hysterectomy, or successful Essure(R) placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or <1 year has passed since the last menses if menopausal.
    * Includes non-male sexual relationships, full abstinence from sexual intercourse with a male partner, monogamous relationship with vasectomized partner who has been vasectomized for 180 days or more and shown to be azoospermic prior to the subject receiving the study vaccination, barrier methods such as condoms or diaphragms/cervical cap with spermicide, effective intrauterine devices, NuvaRing(R), and licensed hormonal methods such as implants, injectables or oral contraceptives ("the pill").
12. Women of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to the first study vaccination.
13. For a woman with potential to become pregnant, she understands that in the event of pregnancy during the study she will be approached to enroll in the Sanofi Pregnancy Registry.
14. Must agree to have residual specimens (i.e. residual/excess of per protocol specifications).

Exclusion Criteria:

1. Have an acute illness*, as determined by the site Principal Investigator (PI) or appropriate sub-investigator, within 72 hours prior to study vaccination.

   *An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
2. Have any medical disease or condition that, in the opinion of the site PI or appropriate sub-investigator, is a contraindication to study participation*.

   *Including acute, subacute, intermittent or chronic medical disease or condition that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial.
3. Have immunosuppression as a result of an underlying illness or treatment, a recent history or current use of immunosuppressive or immunomodulating disease therapy.
4. Use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to study vaccination.
5. Have known active or recently active (12 months) neoplastic disease or a history of any hematologic malignancy. Non-melanoma, treated, skin cancers are permitted.
6. Have known human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection.
7. Have known hypersensitivity or allergy to eggs, egg or chicken protein, squalene-based adjuvants, or other components of the study vaccine.
8. Have a history of severe reactions following previous immunization with licensed or unlicensed influenza vaccines.
9. Have a history of Guillain-Barré Syndrome (GBS).
10. Have a history of convulsions or encephalomyelitis within 90 days prior to study vaccination.
11. Have a history of Potentially Immune-Mediated Medical Conditions (PIMMCs).
12. Have a history of alcohol or drug abuse within 5 years prior to study vaccination.
13. Have any diagnosis, current or past, of schizophrenia, bipolar disease or other psychiatric diagnosis that may interfere* with subject compliance or safety evaluations.

    *As determined by the site PI or appropriate sub-investigator.
14. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 5 years prior to study vaccination.
15. Have taken oral or parenteral (including intra-articular) corticosteroids of any dose within 30 days prior to study vaccination.
16. Have taken high-dose inhaled corticosteroids* within 30 days prior to study vaccination.

    *High-dose defined as per age as using inhaled high-dose per reference chart in the National Heart, Lung and Blood Institute Guidelines for the Diagnosis and Management of Asthma (EPR-3) or other lists published in UPTODATE.
17. Received or plan to receive a licensed, live vaccine (excluding all licensed, seasonal LAIVs) within 30 days before or after the study vaccination.
18. Received or plan to receive a licensed, inactivated vaccine (excluding all licensed, seasonal IIVs) within 14 days before or after each study vaccination.
19. Have received any 2018/2019 seasonal influenza vaccine within the 6 months prior to enrollment.
20. Plans to receive any 2019/2020 seasonal influenza vaccine within approximately 90 days of receipt of the first study vaccination.
21. Have a known history of documented influenza infection within the past 6 months.
22. Received immunoglobulin or other blood products (except Rho D immunoglobulin) within 90 days prior to study vaccination.
23. Received an experimental agent* within 30 days prior to the study vaccination or expect to receive another experimental agent* during the trial-reporting period*.

    *Including vaccine, drug, biologic, device, blood product, or medication.

    **Other than from participation in this trial.

    ***Approximately 12 months after the first study vaccination.
24. Are participating or plan to participate in another clinical trial with an interventional agent* that will be received during the trial-reporting period**.

    *Including licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication.

    **Approximately 12 months after the first study vaccination.
25. Female subjects who are breastfeeding or plan to breastfeed from the time of the first study vaccination through 30 days after the last study vaccination.
26. Plan to travel outside the US (continental US, Hawaii and Alaska) from the time of study vaccination through approximately 90 days after the first study vaccination.
27. Planning to donate blood within 4 months following first vaccination.

Exclusion Criteria for Second Study Vaccination:

All study participants will be expected to receive the second study vaccination except under the circumstances listed below. The second study vaccination will not be administered to a subject if any of the following criteria are met:

* Meets the contraindication on the package insert to receipt of licensed influenza vaccine.
* As deemed necessary by the site principal investigator or appropriate sub-investigator for noncompliance or other reasons.
* Subject refusal of further study vaccination.
* Withdrawal of consent.
* Subject is lost to follow-up.
* Termination of this trial.
* New information becomes available that makes further participation unsafe.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 241 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-09-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Iowa - Vaccine Research and Education Unit, Iowa City, Iowa
  - University of Maryland Baltimore - School of Medicine - Medicine, Baltimore, Maryland
  - Saint Louis University Center for Vaccine Development, St Louis, Missouri
  - Duke Vaccine and Trials Unit, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center Vaccine Research Center, Cincinnati, Ohio
  - Vanderbilt University - Pediatric - Vanderbilt Vaccine Research Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Derived] Hegmann TE, Walter EB, Smith MJ, Campbell J, El Sahly HM, Whitaker JA, Creech CB, Ustyugova IV, Goncalvez AP, Pandey A, Alefantis T, Sridhar S, Honda-Okubo Y, Petrovsky N, Frey SE, Abate G, Paulsen G, Anderson EJ, Rostad CA, Rouphael N, Makhene M, Roberts PC, Tuyishimire B, Bryant C, Winokur P. A phase I study of the safety, reactogenicity and immunogenicity of two quadrivalent seasonal influenza vaccines (Fluzone(R) or Flublok(R)) with or without one of two adjuvants (AF03 or Advax-CpG55.2) in healthy adults 18-45 years of age. Vaccine. 2025 Apr 30;54:126991. doi: 10.1016/j.vaccine.2025.126991. Epub 2025 Mar 18. PMID 40107003

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy males and non-pregnant females aged 18 to 45 years old recruited from existing volunteer populations and from the communities at large around the clinical sites. Participants were enrolled between 18JUN2019 and 27AUG2019.
Groups:
- Fluzone: 0.5 mL of 2018/2019 Fluzone QIV intramuscular injection on Day 1 and 0.5 ml of 2019/2020 Fluzone QIV intramuscular injection on Day 90.
  Influenza Virus Quadrivalent Inactivated Vaccine: unadjuvanted 2018/2019 Fluzone QIV and 2019/2020 Fluzone QIV vaccines will be given with 90 days interval
- Fluzone + AF03: 0.5 mL of 2018/2019 Fluzone QIV + 0.25 mL of AF03 (admixed with vaccine) intramuscular injection on Day 1 and 0.5 ml of 2019/2020 Fluzone QIV intramuscular injection on Day 90.
  AF03: A squalene-in-PBS emulsion stabilized by nonionic surfactants, sorbitan oleate and macrogol cetostearyl ether
  Influenza Virus Quadrivalent Inactivated Vaccine: 2018/2019 Fluzone QIV and 2019/2020 Fluzone QIV vaccines will be given with 90 days interval
- Fluzone + CpG55: 0.5 mL of 2018/2019 Fluzone QIV + 0.5 mL of Delta Inulin-CpG55.2 (admixed with vaccine) intramuscular injection on Day 1 and 0.5 mL 2019/2020 of Fluzone QIV intramuscular injection on Day 90.
  Delta Inulin-CpG55.2 (referred to as CpG55): A combination adjuvant supplied as two separate components, Delta Inulin (Sypharma Pty Ltd.) and CpG55.2 (Nikko Denka Avecia and Sypharma Pty Ltd)
  Influenza Virus Quadrivalent Inactivated Vaccine: 2018/2019 Fluzone QIV and 2019/2020 Fluzone QIV vaccines will be given with 90 days interval
- Flublok: 0.5 mL of 2018/2019 Flublok QIV intramuscular injection on Day 1 and 0.5 ml of 2019/2020 Flublok QIV intramuscular injection on Day 90.
  Quadrivalent Recombinant Seasonal Influenza Vaccine: unadjuvanted 2018/2019 Flublok QIV and 2019/2020 Flublok QIV vaccines will be given with 90 days interval
- Flublok + AF03: 0.5 mL of 2018/2019 Flublok QIV + 0.25 mL AF03 (admixed with vaccine) intramuscular injection on Day 1 and 0.5 ml of 2019/2020 Flublok QIV intramuscular injection on Day 90.
  AF03: A squalene-in-PBS emulsion stabilized by nonionic surfactants, sorbitan oleate and macrogol cetostearyl ether
  Quadrivalent Recombinant Seasonal Influenza Vaccine: 2018/2019 Flublok QIV and 2019/2020 Flublok QIV vaccines will be given with 90 days interval
- Flublok + CpG55: 0.5 mL of 2018/2019 Flublok QIV + 0.5 mL of Delta Inulin-CpG55.2 (admixed with vaccine) intramuscular injection on Day 1 and 0.5 ml of 2019/2020 Flublok QIV intramuscular injection on Day 90.
  Delta Inulin-CpG55.2 (referred to as CpG55): A combination adjuvant supplied as two separate components, Delta Inulin (Sypharma Pty Ltd.) and CpG55.2 (Nikko Denka Avecia and Sypharma Pty Ltd)
  Quadrivalent Recombinant Seasonal Influenza Vaccine: 2018/2019 Flublok QIV and 2019/2020 Flublok QIV vaccines will be given with 90 days interval
Period: Overall Study
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Started | 41 | 37 | 40 | 41 | 39 | 43
Completed | 39 | 32 | 39 | 39 | 36 | 40
Not Completed | 2 | 5 | 1 | 2 | 3 | 3
Not completed — Enrolled but treatment not administered | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 5 | 0 | 1 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all participants that were enrolled.
Groups:
- Fluzone: 0.5 mL of 2018/2019 Fluzone QIV intramuscular injection on Day 1 and 0.5 ml of 2019/2020 Fluzone QIV intramuscular injection on Day 90.
- Fluzone + AF03: 0.5 mL of 2018/2019 Fluzone QIV + 0.25 mL of AF03 (admixed with vaccine) intramuscular injection on Day 1 and 0.5 ml of 2019/2020 Fluzone QIV intramuscular injection on Day 90.
- Fluzone + CpG55: 0.5 mL of 2018/2019 Fluzone QIV + 0.5 mL of Delta Inulin-CpG55.2 (admixed with vaccine) intramuscular injection on Day 1 and 0.5 mL of 2019/2020 of Fluzone QIV intramuscular injection on Day 90.
- Flublok: 0.5 mL of 2018/2019 Flublok QIV intramuscular injection on Day 1 and 0.5 ml of 2019/2020 Flublok QIV intramuscular injection on Day 90.
- Flublok + AF03: 0.5 mL of 2018/2019 Flublok QIV + 0.25 mL AF03 (admixed with vaccine) intramuscular injection on Day 1 and 0.5 ml of 2019/2020 Flublok QIV intramuscular injection on Day 90.
- Flublok + CpG55: 0.5 mL of 2018/2019 Flublok QIV + 0.5 mL of Delta Inulin-CpG55.2 (admixed with vaccine) intramuscular injection on Day 1 and 0.5 ml of 2019/2020 Flublok QIV intramuscular injection on Day 90.
- Total: Total of all reporting groups
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55 | Total
Number analyzed (Participants) | 41 | 37 | 40 | 41 | 39 | 43 | 241
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 41 | 37 | 40 | 41 | 39 | 43 | 241
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (7.2) | 29.6 (6.2) | 28.2 (7.0) | 30.2 (7.6) | 29.7 (6.8) | 28.7 (6.5) | 29.5 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 26 | 28 | 27 | 23 | 26 | 152
  Male | 19 | 11 | 12 | 14 | 16 | 17 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 3 | 7 | 5 | 3 | 23
  Not Hispanic or Latino | 40 | 33 | 36 | 34 | 34 | 40 | 217
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 1 | 2 | 4 | 5 | 5 | 5 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 4 | 2 | 7 | 8 | 2 | 30
  White | 33 | 28 | 32 | 26 | 24 | 34 | 177
  More than one race | 0 | 2 | 2 | 1 | 2 | 2 | 9
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 41 | 37 | 40 | 41 | 39 | 43 | 241
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.73 (5.37) | 26.87 (6.29) | 24.82 (4.64) | 26.91 (6.55) | 26.25 (6.81) | 25.79 (5.67) | 26.22 (5.91)
Prior Seasonal Influenza Vaccination [Count of Participants; unit: Participants]
  Either 2017-2018 or 2018-2019 | 36 | 29 | 32 | 32 | 30 | 36 | 195
  Neither 2017-2018 or 2018-2019 | 5 | 7 | 8 | 8 | 9 | 7 | 44
  Unknown | 0 | 1 | 0 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local and Systemic Solicited Reactogenicity Events Post First Vaccination
Description: Local adverse events (AEs) solicited on a memory aid provided to participants included Pain, Tenderness, Itching/Pruritus, Ecchymosis/Bruising (functional grade based on interference with daily activities), Ecchymosis/Bruising (any measured value >0mm), Erythema/Redness (functional grade), Erythema/ Redness (any measured value >0mm), Induration/Swelling (functional grade), and Induration/Swelling (any measured value >0mm).
  Systemic AEs solicited on a memory aid provided to participants included Elevated Oral Temperature, Feverishness, Fatigue, Malaise, Myalgia, Arthralgia, Headache, and Nausea. Participants are considered reporting the local or systemic AE if they reported mild or greater severity at any time during the 8 days at or following the first vaccination.
Time Frame: Day 1 through Day 8
Population: The Safety Analysis population includes all participants who received the first study vaccination. Analyses for the safety population are based on vaccine actually received. One participant randomized to Flublok + AF03 group received Flublok due to a pharmacy error and is analyzed in the Flublok group.
Measure: Count of Participants; unit: Participants
Groups:
- Flublok: 0.5 mL of 2018/2019 Flublok QIV intramuscular injection on Day 1 and 0.5 ml of 2019/2020 Flublok QIV intramuscular injection on Day 90.
  One participant randomized to the Flublok + AF03 arm received Flublok due to a pharmacy error and is analyzed in the Flublok group for safety-related analyses.
- Flublok + AF03: 0.5 mL of 2018/2019 Flublok QIV + 0.25 mL AF03 (admixed with vaccine) intramuscular injection on Day 1 and 0.5 ml of 2019/2020 Flublok QIV intramuscular injection on Day 90.
  One participant randomized to the Flublok + AF03 arm received Flublok due to a pharmacy error and is analyzed in the Flublok group for safety-related analyses.
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 42 | 37 | 43
Participants
  Any Systemic Symptom | 24 | 25 | 23 | 23 | 18 | 26
  Any Local Symptom | 35 | 36 | 40 | 32 | 33 | 43

2. Primary Outcome: Number of Participants Reporting Serious and Non-serious Adverse Events (AE) Through Day 29
Description: Adverse events were defined as any untoward medical occurrence in a participant administered a pharmaceutical product regardless of its causal relationship to the study treatment. Non-serious AEs were collected from participants at follow up visits through 28 days after the first study vaccination while serious adverse events (SAEs) were collected at follow up visits through approximately 12 months after the first study vaccination. Adverse events were MedDRA coded and are summarized by MedDRA System Organ Class (SOC).
Time Frame: Day 1 through Day 29
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 42 | 37 | 43
Participants
  AEs | 12 | 11 | 8 | 14 | 10 | 15
  SAEs | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: SAEs included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation or a congenital anomaly/birth defect. All SAEs were reported from time of first study vaccination through approximately 12 months after the first study vaccination.
Time Frame: Day 1 through Day 365
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Flublok + CpG55: 0.5 mL of 2018/2019 Flublok QIV + 0.5 mL of Delta Inulin-CpG55.2 (admixed with vaccine) intramuscular injection on Day 1 and 0.5 mL of of 2019/2020 Flublok QIV intramuscular injection on Day 90.
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 42 | 37 | 43
Participants | 0 | 1 | 0 | 0 | 0 | 1

4. Primary Outcome: Number of Participants Reporting Clinical Safety Laboratory Adverse Events (AEs) Post First Vaccination
Description: Laboratory parameters include white blood cells (WBC), hemoglobin, platelets, alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin, Gamma-Glutamyl Transferase (GGT), alkaline phosphatase (ALP), amylase, lipase, and creatinine. Thresholds for adverse events were considered WBC of 3.90 x10^3/uL or lower or 10.60 x10^3/uL or higher; hemoglobin 11.4 g/dL or lower (female) or 12.4 g/dL or lower (male); platelets 139 x10^3/uL or below or 416 x10^3/uL or greater when using EDTA tubes or platelets 124 x10^3/uL or below or 550 x10^3/uL or greater when using Citrate tubes; ALT 44 IU/L or greater (female) or 61 IU/L or greater (male); AST 37 IU/L or greater (female) or 44 IU/L or greater (male); bilirubin 1.30 mg/dL or greater; GGT 33 IU/L or greater (female) or 50 IU/L or greater (male); ALP 116 IU/L or greater; amylase 122 IU/L or greater; lipase 61 IU/L or greater; creatinine 1.1 mg/dL or greater (female) or 1.4 mg/dL or greater (male).
Time Frame: Day 1 through Day 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 42 | 37 | 43
Participants
  WBCs | 6 | 2 | 3 | 2 | 3 | 0
  Hemoglobin | 1 | 1 | 2 | 3 | 0 | 0
  Platelets | 0 | 0 | 0 | 4 | 0 | 0
  ALT | 1 | 1 | 0 | 1 | 1 | 1
  AST | 0 | 1 | 0 | 1 | 2 | 1
  Bilirubin | 0 | 0 | 1 | 0 | 1 | 0
  GGT | 2 | 0 | 0 | 0 | 0 | 2
  ALP | 0 | 0 | 0 | 0 | 1 | 1
  Amylase | 1 | 0 | 1 | 0 | 0 | 0
  Lipase | 0 | 1 | 1 | 0 | 0 | 0
  Creatinine | 1 | 0 | 0 | 0 | 0 | 1

5. Primary Outcome: Geometric Mean Titers (GMTs) of Serum Hemagglutination Inhibition (HAI) Against the 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains
Description: Blood was collected for HAI assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at Day 1 and Day 29 post first study vaccination.
Time Frame: Day 1, Day 29
Population: The modified intent-to-treat (mITT) population includes all randomized participants who received the first study vaccination and contributed at least one post-first study vaccination venous blood sample for immunogenicity testing (HAI, NAI or Neut antibody assays) for which valid HAI results were reported. For analyses using the mITT population, participants were grouped based on randomized study arm.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 41 | 38 | 42
titer
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 1 | 114.1 [72.7 to 179.1] | 193.0 [129.8 to 286.8] | 96.8 [60.4 to 155.0] | 164.1 [106.4 to 253.0] | 129.7 [81.1 to 207.5] | 108.6 [74.2 to 158.9]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 1 | 140.9 [88.5 to 224.6] | 149.8 [101.2 to 221.9] | 120.2 [75.7 to 190.8] | 248.3 [156.0 to 395.2] | 107.1 [70.4 to 162.9] | 131.3 [90.6 to 190.2]
  A/Michigan/45/2015 X-275 (H1N1) - Day 1 | 242.1 [164.8 to 355.7] | 196.6 [139.2 to 277.6] | 174.5 [108.2 to 281.2] | 296.6 [194.9 to 451.3] | 186.8 [117.1 to 298.2] | 237.8 [156.9 to 360.3]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 1 | 366.3 [262.9 to 510.4] | 478.7 [311.3 to 736.1] | 489.3 [355.3 to 673.7] | 618.7 [397.9 to 962.2] | 331.9 [208.7 to 527.8] | 390.1 [296.2 to 513.7]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 29 | 270.2 [195.9 to 372.8] | 538.2 [414.7 to 698.5] | 340.5 [257.1 to 451.0] | 634.5 [478.4 to 841.4] | 516.0 [357.5 to 744.6] | 492.5 [359.4 to 674.8]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 29 | 423.0 [323.1 to 553.7] | 456.9 [338.5 to 616.7] | 349.7 [253.3 to 482.9] | 515.4 [355.0 to 748.3] | 416.0 [281.3 to 615.2] | 388.7 [278.7 to 542.1]
  A/Michigan/45/2015 X-275 (H1N1) - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Michigan/45/2015 X-275 (H1N1) - Day 29 | 488.3 [363.2 to 656.6] | 474.9 [354.3 to 636.4] | 365.6 [259.8 to 514.5] | 680.0 [479.4 to 964.5] | 722.9 [516.0 to 1012.7] | 522.5 [371.6 to 734.6]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 29 | 952.2 [721.6 to 1256.5] | 1356.1 [1006.0 to 1828.1] | 1081.1 [828.3 to 1411.2] | 1645.6 [1252.9 to 2161.4] | 1280.0 [969.6 to 1689.8] | 1280.0 [995.0 to 1646.6]

6. Primary Outcome: Ratio of Geometric Mean Titers (GMTs) of Serum Hemagglutination Inhibition (HAI) Against the 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains Between Adjuvanted and Unadjuvanted Study Arms
Description: Blood was collected for HAI assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at Day 1 and Day 29 post first study vaccination and the ratio of these GMTs between adjuvanted and unadjuvanted study arms were calculated.
  Unadjuvanted Fluzone and Flublok study arms are considered as reference groups for the analysis of ratio of GMTs.
  Ratio of GMTs is defined as the ratio of the GMT from the adjuvanted group divided by the GMT from the corresponding unadjuvanted group.
Time Frame: Day 1, Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: ratio of GMT
Arm/Group | Fluzone + AF03 | Fluzone + CpG55 | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 37 | 40 | 38 | 42
ratio of GMT
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 1 | 1.7 [0.9 to 3.1] | 0.8 [0.4 to 1.6] | 0.8 [0.4 to 1.5] | 0.7 [0.4 to 1.2]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 1 | 1.1 [0.6 to 1.9] | 0.9 [0.4 to 1.6] | 0.4 [0.2 to 0.8] | 0.5 [0.3 to 0.9]
  A/Michigan/45/2015 X-275 (H1N1) - Day 1 | 0.8 [0.5 to 1.4] | 0.7 [0.4 to 1.3] | 0.6 [0.3 to 1.2] | 0.8 [0.4 to 1.4]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 1 | 1.3 [0.8 to 2.2] | 1.3 [0.8 to 2.1] | 0.5 [0.3 to 1.0] | 0.6 [0.4 to 1.1]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 29: number analyzed (Participants) | 36 | 39 | 37 | 41
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 29 | 2.0 [1.3 to 3.0] | 1.3 [0.8 to 1.9] | 0.8 [0.5 to 1.3] | 0.8 [0.5 to 1.2]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 29: number analyzed (Participants) | 36 | 39 | 37 | 41
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 29 | 1.1 [0.7 to 1.6] | 0.8 [0.5 to 1.3] | 0.8 [0.5 to 1.4] | 0.8 [0.5 to 1.2]
  A/Michigan/45/2015 X-275 (H1N1) - Day 29: number analyzed (Participants) | 36 | 39 | 37 | 41
  A/Michigan/45/2015 X-275 (H1N1) - Day 29 | 1.0 [0.6 to 1.5] | 0.7 [0.5 to 1.2] | 1.1 [0.7 to 1.7] | 0.8 [0.5 to 1.2]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 29: number analyzed (Participants) | 36 | 39 | 37 | 41
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 29 | 1.4 [1.0 to 2.1] | 1.1 [0.8 to 1.7] | 0.8 [0.5 to 1.1] | 0.8 [0.5 to 1.1]

7. Primary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Titer Seroconversion Against 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains
Description: Blood was collected for HAI assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. HAI seroconversion was defined as either a pre-vaccination titer < 1:10 and a post-vaccination titer >= 1:40 or a pre-vaccination titer >= 1:10 and a minimum four-fold rise in post-vaccination antibody titer.
Time Frame: Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
percentage of participants
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) | 27 [14 to 43] | 33 [19 to 51] | 36 [21 to 53] | 45 [29 to 62] | 46 [29 to 63] | 56 [40 to 72]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) | 29 [16 to 46] | 36 [21 to 54] | 31 [17 to 48] | 23 [11 to 38] | 41 [25 to 58] | 32 [18 to 48]
  A/Michigan/45/2015 X-275 (H1N1) | 24 [12 to 40] | 19 [8 to 36] | 18 [8 to 34] | 23 [11 to 38] | 46 [29 to 63] | 32 [18 to 48]
  B/Phuket/3073/2013 (B Yamagata lineage) | 24 [12 to 40] | 25 [12 to 42] | 23 [11 to 39] | 28 [15 to 44] | 30 [16 to 47] | 34 [20 to 51]

8. Primary Outcome: Percentage of Participants With Hemagglutination Inhibition (HAI) Titer of 1:40 or Greater Against the 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains
Description: Blood was collected for HAI assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result.
Time Frame: Day 1, Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 41 | 38 | 42
percentage of participants
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 1 | 85 [71 to 94] | 95 [82 to NA] — Value is NA because it's >99 but <100 | 75 [59 to 87] | 93 [80 to 98] | 76 [60 to 89] | 88 [74 to 96]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 1 | 80 [65 to 91] | 89 [75 to 97] | 80 [64 to 91] | 90 [77 to 97] | 79 [63 to 90] | 90 [77 to 97]
  A/Michigan/45/2015 X-275 (H1N1) - Day 1 | 93 [80 to 98] | 95 [82 to NA] — Value is NA because it's >99 but <100 | 88 [73 to 96] | 93 [80 to 98] | 89 [75 to 97] | 95 [84 to NA] — Value is NA because it's >99 but <100
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 1 | 98 [87 to NA] — Value is NA because it's >99 but <100 | 95 [82 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 95 [83 to NA] — Value is NA because it's >99 but <100 | 92 [79 to 98] | 100 [92 to 100]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 29 | 100 [91 to 100] | 100 [90 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 29 | 100 [91 to 100] | 100 [90 to 100] | 97 [87 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 97 [86 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100]
  A/Michigan/45/2015 X-275 (H1N1) - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Michigan/45/2015 X-275 (H1N1) - Day 29 | 100 [91 to 100] | 100 [90 to 100] | 97 [87 to NA] — Value is NA because it's >99 but <100 | 98 [87 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 100 [91 to 100]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 29 | 100 [91 to 100] | 100 [90 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100]

9. Primary Outcome: Geometric Mean Fold Rise (GMFR) in Hemagglutination Inhibition (HAI) Titers Against the 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains
Description: Blood was collected for HAI assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. Fold-rises from baseline were calculated as the Day 29 titer divided by the baseline titers for each participant. The geometric mean of these fold rises was then calculated to obtain the GMFR.
Time Frame: Day 29
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
fold rise
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) | 2.4 [1.6 to 3.6] | 2.6 [1.8 to 3.7] | 3.6 [2.4 to 5.5] | 3.8 [2.5 to 5.7] | 3.8 [2.7 to 5.3] | 4.3 [2.9 to 6.3]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) | 3.0 [2.0 to 4.5] | 3.2 [2.1 to 4.8] | 2.9 [2.0 to 4.4] | 2.1 [1.5 to 2.7] | 3.7 [2.5 to 5.4] | 2.9 [2.1 to 4.0]
  A/Michigan/45/2015 X-275 (H1N1) | 2.0 [1.4 to 3.0] | 2.3 [1.5 to 3.5] | 2.2 [1.5 to 3.2] | 2.1 [1.7 to 2.8] | 3.7 [2.4 to 5.8] | 2.1 [1.5 to 3.0]
  B/Phuket/3073/2013 (B Yamagata lineage) | 2.6 [1.9 to 3.6] | 2.7 [1.8 to 4.0] | 2.3 [1.7 to 3.0] | 2.6 [1.9 to 3.7] | 4.0 [2.6 to 6.0] | 3.2 [2.4 to 4.2]

10. Primary Outcome: Geometric Mean Titers (GMTs) of Serum Neuraminidase Inhibition (NAI) Against the 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains
Description: Blood was collected for NAI assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at Day 1 and Day 29 post first study vaccination.
Time Frame: Day 1, Day 29
Population: The modified intent-to-treat (mITT) population includes all randomized participants who received the first study vaccination and contributed at least one post-first study vaccination venous blood sample for immunogenicity testing (HAI, NAI or Neut antibody assays) for which valid NAI results were reported. For analyses using the mITT population, participants were grouped based on randomized study arm.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 41 | 38 | 42
titer
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 1 | 123.1 [85.1 to 178.1] | 116.4 [82.3 to 164.5] | 91.9 [60.3 to 140.1] | 140.9 [91.1 to 218.0] | 129.7 [92.5 to 181.8] | 105.9 [73.8 to 152.0]
  B/Colorado/06/2017 (B Victoria lineage) - Day 1 | 178.6 [142.4 to 223.9] | 211.9 [156.5 to 286.9] | 213.0 [160.3 to 282.9] | 256.9 [183.1 to 360.4] | 226.3 [170.3 to 300.6] | 166.7 [131.3 to 211.7]
  A/Michigan/45/2015 X-275 (H1N1) - Day 1 | 118.0 [81.6 to 170.6] | 108.0 [75.4 to 154.7] | 96.8 [63.7 to 147.0] | 143.3 [92.8 to 221.5] | 127.4 [89.8 to 180.7] | 100.8 [69.2 to 146.7]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 1 | 63.1 [49.9 to 79.9] | 89.5 [69.6 to 115.1] | 91.1 [72.5 to 114.5] | 88.5 [65.8 to 119.1] | 81.5 [62.8 to 105.7] | 66.7 [54.0 to 82.5]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 29 | 259.0 [197.1 to 340.5] | 293.4 [213.9 to 402.6] | 224.3 [164.5 to 305.7] | 157.3 [105.7 to 234.0] | 129.0 [94.0 to 177.1] | 107.5 [74.7 to 154.8]
  B/Colorado/06/2017 (B Victoria lineage) - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  B/Colorado/06/2017 (B Victoria lineage) - Day 29 | 402.0 [333.4 to 484.8] | 538.2 [409.8 to 706.8] | 464.8 [367.3 to 588.1] | 346.0 [258.6 to 462.8] | 243.9 [186.7 to 318.5] | 211.5 [167.6 to 266.8]
  A/Michigan/45/2015 X-275 (H1N1) - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Michigan/45/2015 X-275 (H1N1) - Day 29 | 250.4 [191.5 to 327.5] | 264.0 [195.8 to 355.8] | 216.4 [160.6 to 291.7] | 161.4 [111.1 to 234.5] | 129.0 [95.7 to 173.9] | 105.7 [73.0 to 153.3]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 29 | 116.0 [98.2 to 137.1] | 188.5 [147.0 to 241.6] | 143.8 [117.2 to 176.5] | 112.2 [87.8 to 143.3] | 92.1 [72.7 to 116.6] | 82.1 [66.9 to 100.6]

11. Primary Outcome: Ratio of Geometric Mean Titers (GMTs) of Serum Neuraminidase Inhibition (NAI) Against the 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains Between Adjuvanted and Unadjuvanted Study Arms
Description: Blood was collected for NAI assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at Day 1 and Day 29 post first study vaccination and the ratio of these GMTs between adjuvanted and unadjuvanted study arms were calculated.
  Unadjuvanted Fluzone and Flublok study arms are considered as reference groups for the analysis of ratio of GMTs.
  Ratio of GMTs is defined as the ratio of the GMT from the adjuvanted group divided by the GMT from the corresponding unadjuvanted group.
Time Frame: Day 1, Day 29
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: ratio of GMT
Arm/Group | Fluzone + AF03 | Fluzone + CpG55 | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 37 | 40 | 38 | 42
ratio of GMT
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 1 | 0.9 [0.6 to 1.6] | 0.7 [0.4 to 1.3] | 0.9 [0.5 to 1.6] | 0.8 [0.4 to 1.3]
  B/Colorado/06/2017 (B Victoria lineage) - Day 1 | 1.2 [0.8 to 1.7] | 1.2 [0.8 to 1.7] | 0.9 [0.6 to 1.4] | 0.6 [0.4 to 1.0]
  A/Michigan/45/2015 X-275 (H1N1) - Day 1 | 0.9 [0.6 to 1.5] | 0.8 [0.5 to 1.4] | 0.9 [0.5 to 1.5] | 0.7 [0.4 to 1.2]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 1 | 1.4 [1.0 to 2.0] | 1.4 [1.0 to 2.0] | 0.9 [0.6 to 1.4] | 0.8 [0.5 to 1.1]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 29: number analyzed (Participants) | 36 | 39 | 37 | 41
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 29 | 1.1 [0.8 to 1.7] | 0.9 [0.6 to 1.3] | 0.8 [0.5 to 1.4] | 0.7 [0.4 to 1.2]
  B/Colorado/06/2017 (B Victoria lineage) - Day 29: number analyzed (Participants) | 36 | 39 | 37 | 41
  B/Colorado/06/2017 (B Victoria lineage) - Day 29 | 1.3 [1.0 to 1.9] | 1.2 [0.9 to 1.6] | 0.7 [0.5 to 1.0] | 0.6 [0.4 to 0.9]
  A/Michigan/45/2015 X-275 (H1N1) - Day 29: number analyzed (Participants) | 36 | 39 | 37 | 41
  A/Michigan/45/2015 X-275 (H1N1) - Day 29 | 1.1 [0.7 to 1.6] | 0.9 [0.6 to 1.3] | 0.8 [0.5 to 1.3] | 0.7 [0.4 to 1.1]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 29: number analyzed (Participants) | 36 | 39 | 37 | 41
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 29 | 1.6 [1.2 to 2.2] | 1.2 [1.0 to 1.6] | 0.8 [0.6 to 1.1] | 0.7 [0.5 to 1.0]

12. Primary Outcome: Percentage of Participants Achieving Neuraminidase Inhibition (NAI) Titer Seroconversion Against 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains
Description: Blood was collected for NAI assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. NAI seroconversion was defined as >4 four-fold rise in post-vaccination antibody titer at Day 29.
Time Frame: Day 29
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
percentage of participants
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) | 27 [14 to 43] | 36 [21 to 54] | 36 [21 to 53] | 3 [NA to 13] — Value is NA because it's >0 but <1 | 0 [0 to 9] | 2 [NA to 13] — Value is NA because it's >0 but <1
  B/Colorado/06/2017 (B Victoria lineage) | 27 [14 to 43] | 25 [12 to 42] | 18 [8 to 34] | 0 [0 to 9] | 0 [0 to 9] | 5 [NA to 17] — Value is NA because it's >0 but <1
  A/Michigan/45/2015 X-275 (H1N1) | 27 [14 to 43] | 31 [16 to 48] | 36 [21 to 53] | 3 [NA to 13] — Value is NA because it's >0 but <1 | 0 [0 to 9] | 2 [NA to 13] — Value is NA because it's >0 but <1
  B/Phuket/3073/2013 (B Yamagata lineage) | 20 [9 to 35] | 22 [10 to 39] | 10 [3 to 24] | 3 [NA to 13] — Value is NA because it's >0 but <1 | 0 [0 to 9] | 2 [NA to 13] — Value is NA because it's >0 but <1

13. Primary Outcome: Geometric Mean Fold Rise (GMFR) in Neuraminidase Inhibition (NAI) Titers Against the 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains
Description: Blood was collected for NAI assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. Fold-rises from baseline were calculated as the Day 29 titer divided by the baseline titers for each participant. The geometric mean of these fold rises was then calculated to obtain the GMFR.
Time Frame: Day 29
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
fold rise
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) | 2.1 [1.6 to 2.7] | 2.5 [2.0 to 3.3] | 2.6 [2.0 to 3.2] | 1.0 [0.9 to 1.2] | 1.0 [0.9 to 1.1] | 1.0 [0.9 to 1.3]
  B/Colorado/06/2017 (B Victoria lineage) | 2.3 [1.9 to 2.7] | 2.6 [2.0 to 3.3] | 2.2 [1.8 to 2.7] | 1.2 [1.1 to 1.4] | 1.1 [1.0 to 1.2] | 1.2 [1.0 to 1.5]
  A/Michigan/45/2015 X-275 (H1N1) | 2.1 [1.7 to 2.7] | 2.5 [1.9 to 3.2] | 2.4 [1.9 to 3.0] | 1.0 [0.9 to 1.2] | 1.0 [0.9 to 1.2] | 1.1 [0.9 to 1.3]
  B/Phuket/3073/2013 (B Yamagata lineage | 1.8 [1.5 to 2.3] | 2.1 [1.7 to 2.6] | 1.6 [1.3 to 2.0] | 1.2 [1.0 to 1.3] | 1.2 [1.0 to 1.3] | 1.2 [1.0 to 1.4]

14. Primary Outcome: Geometric Mean Titers (GMTs) of Serum Neutralizing (Neut) Titers Against the 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains
Description: Blood was collected for Neut assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, but only one result which a geometric mean titer of the replicates was reported by the lab. The geometric mean titer was calculated for each study arm from the available results at Day 1 and Day 29 post first study vaccination.
Time Frame: Day 1, Day 29
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 41 | 38 | 42
titer
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 1 | 106.8 [78.0 to 146.1] | 147.7 [111.1 to 196.3] | 101.9 [75.5 to 137.6] | 151.6 [109.9 to 209.2] | 121.2 [87.6 to 167.7] | 118.5 [88.4 to 158.8]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 1 | 108.9 [63.1 to 187.9] | 113.4 [68.8 to 186.9] | 94.0 [53.9 to 164.0] | 199.4 [115.0 to 345.9] | 81.9 [49.7 to 134.9] | 101.0 [65.3 to 156.4]
  A/Michigan/45/2015 X-275 (H1N1) - Day 1 | 3141.7 [2145.9 to 4599.4] | 2697.5 [1756.2 to 4143.2] | 2147.8 [1271.7 to 3627.5] | 3703.3 [2937.7 to 5719.6] | 2214.0 [1337.5 to 3664.9] | 2764.2 [1667.7 to 4581.7]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 1 | 479.4 [320.1 to 717.9] | 577.8 [383.2 to 871.1] | 630.3 [447.0 to 889.0] | 860.1 [562.1 to 1316.1] | 447.8 [281.3 to 712.9] | 539.2 [394.8 to 736.5]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 29 | 379.1 [285.4 to 503.4] | 671.9 [497.1 to 908.2] | 456.5 [334.5 to 622.9] | 848.9 [667.6 to 1079.4] | 741.9 [536.1 to 1026.7] | 567.0 [422.5 to 760.9]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 29 | 302.2 [207.7 to 439.8] | 305.1 [219.1 to 424.9] | 248.4 [169.4 to 364.3] | 463.3 [279.2 to 768.9] | 304.8 [188.2 to 493.7] | 291.6 [191.2 to 444.7]
  A/Michigan/45/2015 X-275 (H1N1) - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Michigan/45/2015 X-275 (H1N1) - Day 29 | 5639.5 [3958.0 to 8035.2] | 5435.2 [3627.9 to 8142.8] | 4455.8 [2877.2 to 6900.5] | 8539.5 [5785.7 to 12603.9] | 9197.6 [5941.1 to 14239.1] | 6021.9 [4138.3 to 8762.7]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 29 | 1162.7 [860.0 to 1572.0] | 1437.4 [1053.1 to 1962.0] | 1152.1 [873.2 to 1520.1] | 2053.5 [1509.7 to 2793.3] | 1473.1 [1049.7 to 2067.5] | 1291.7 [940.6 to 1774.0]

15. Primary Outcome: Ratio of Serum Neutralizing (Neut) Geometric Mean Titers (GMT) Against the 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains Between Adjuvanted and Unadjuvanted Study Arms
Description: Blood was collected for Neut assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, but only one result which a geometric mean titer of the replicates was reported by the lab. The geometric mean titer was calculated for each study arm from the available results at Day 1 and Day 29 post first study vaccination and the ratio of these GMTs between adjuvanted and unadjuvanted study arms were calculated.
  Unadjuvanted Fluzone and Flublok study arms are considered as reference groups for the analysis of ratio of GMTs.
  Ratio of GMTs is defined as the ratio of the GMT from the adjuvanted group divided by the GMT from the corresponding unadjuvanted group.
Time Frame: Day 1, Day 29
Population: The modified intent-to-treat (mITT) population includes all randomized participants who received the first study vaccination and contributed at least one post-first study vaccination venous blood sample for immunogenicity testing (HAI, NAI or Neut antibody assays) for which valid Neut results were reported. For analyses using the mITT population, participants were grouped based on randomized study arm.
Measure: Number (95% Confidence Interval); unit: ratio of GMT
Arm/Group | Fluzone + AF03 | Fluzone + CpG55 | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 37 | 40 | 38 | 42
ratio of GMT
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 1 | 1.4 [0.9 to 2.1] | 1.0 [0.6 to 1.5] | 0.8 [0.5 to 1.3] | 0.8 [0.5 to 1.2]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 1 | 1.0 [0.5 to 2.2] | 0.9 [0.4 to 1.9] | 0.4 [0.2 to 0.9] | 0.5 [0.3 to 1.0]
  A/Michigan/45/2015 X-275 (H1N1) - Day 1 | 0.9 [0.5 to 1.5] | 0.7 [0.4 to 1.3] | 0.6 [0.3 to 1.2] | 0.7 [0.4 to 1.4]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 1 | 1.2 [0.7 to 2.1] | 1.3 [0.8 to 2.2] | 0.5 [0.3 to 1.0] | 0.6 [0.4 to 1.1]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 29: number analyzed (Participants) | 36 | 39 | 37 | 41
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 29 | 1.8 [1.2 to 2.7] | 1.2 [0.8 to 1.8] | 0.9 [0.6 to 1.3] | 0.7 [0.5 to 1.0]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 29: number analyzed (Participants) | 36 | 39 | 37 | 41
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 29 | 1.0 [0.6 to 1.7] | 0.8 [0.5 to 1.4] | 0.7 [0.3 to 1.3] | 0.6 [0.3 to 1.2]
  A/Michigan/45/2015 X-275 (H1N1) - Day 29: number analyzed (Participants) | 36 | 39 | 37 | 41
  A/Michigan/45/2015 X-275 (H1N1) - Day 29 | 1.0 [0.6 to 1.6] | 0.8 [0.5 to 1.4] | 1.1 [0.6 to 1.9] | 0.7 [0.4 to 1.2]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 29: number analyzed (Participants) | 36 | 39 | 37 | 41
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 29 | 1.2 [0.8 to 1.9] | 1.0 [0.7 to 1.5] | 0.7 [0.5 to 1.1] | 0.6 [0.4 to 1.0]

16. Primary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Titer Seroconversion Against 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains
Description: Blood was collected for Neut assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, but only one result which a geometric mean titer of the replicates was reported by the lab. Neut seroconversion was defined as either a pre-vaccination titer < 1:10 and a post-vaccination titer >= 1:40 or a pre-vaccination titer >= 1:10 and a minimum four-fold rise in post-vaccination antibody titer.
Time Frame: Day 29
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
percentage of participants
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) | 37 [22 to 53] | 42 [26 to 59] | 38 [23 to 55] | 60 [43 to 75] | 65 [47 to 80] | 56 [40 to 72]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) | 22 [11 to 38] | 19 [8 to 36] | 28 [15 to 45] | 20 [9 to 36] | 30 [16 to 47] | 34 [20 to 51]
  A/Michigan/45/2015 X-275 (H1N1) | 15 [6 to 29] | 11 [3 to 26] | 21 [9 to 36] | 20 [9 to 36] | 41 [25 to 58] | 20 [9 to 35]
  B/Phuket/3073/2013 (B Yamagata lineage) | 24 [12 to 40] | 14 [5 to 29] | 18 [8 to 34] | 18 [7 to 33] | 30 [16 to 47] | 22 [11 to 38]

17. Primary Outcome: Percentage of Participants With Neutralizing (Neut) Titer of 1:40 or Greater Against the 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains
Description: Blood was collected for Neut assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, but only one result which a geometric mean titer of the replicates was reported by the lab.
Time Frame: Day 1, Day 29
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 41 | 38 | 42
percentage of participants
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 1 | 88 [74 to 96] | 95 [82 to NA] — Value is NA because it's >99 but <100 | 75 [59 to 87] | 90 [77 to 97] | 89 [75 to 97] | 90 [77 to 97]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 1 | 78 [62 to 89] | 78 [62 to 90] | 68 [51 to 81] | 83 [68 to 93] | 71 [54 to 85] | 76 [61 to 88]
  A/Michigan/45/2015 X-275 (H1N1) - Day 1 | 100 [91 to 100] | 97 [86 to NA] — Value is NA because it's >99 but <100 | 98 [87 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 97 [86 to NA] — Value is NA because it's >99 but <100 | 98 [87 to NA] — Value is NA because it's >99 but <100
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 1 | 100 [91 to 100] | 97 [86 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 95 [83 to NA] — Value is NA because it's >99 but <100 | 92 [79 to 98] | 100 [92 to 100]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 29 | 100 [91 to 100] | 100 [90 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 29 | 95 [83 to NA] — Value is NA because it's >99 but <100 | 97 [85 to NA] — Value is NA because it's >99 but <100 | 95 [83 to NA] — Value is NA because it's >99 but <100 | 90 [76 to 97] | 92 [78 to 98] | 95 [83 to NA] — Value is NA because it's >99 but <100
  A/Michigan/45/2015 X-275 (H1N1) - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Michigan/45/2015 X-275 (H1N1) - Day 29 | 100 [91 to 100] | 100 [90 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 29 | 100 [91 to 100] | 100 [90 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100]

18. Primary Outcome: Geometric Mean Fold Rise (GMFR) in Neutralizing (Neut) Titers Against the 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains
Description: Blood was collected for Neut assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, but only one result which a geometric mean titer of the replicates was reported by the lab. Fold-rises from baseline were calculated as the Day 29 titer divided by the baseline titers for each participant. The geometric mean of these fold rises was then calculated to obtain the GMFR.
Time Frame: Day 29
Population: The modified intent-to-treat (mITT) population includes all randomized participants who received the first study vaccination and contributed at least one post-first study vaccination venous blood samples for immunogenicity testing (HAI, NAI or Neut antibody assays) for which valid Neut results were reported. For analyses using the mITT population, participants were grouped based on randomized study arm.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Groups:
- Fluzone + CpG55: 0.5 mL of 2018/2019 Fluzone QIV + 0.5 mL of Delta Inulin-CpG55.2 (admixed with vaccine) intramuscular injection on Day 1 and 0.5 2019/2020 of Fluzone QIV intramuscular injection on Day 90.
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
fold rise
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) | 3.6 [2.7 to 4.7] | 4.3 [3.1 to 6.1] | 4.6 [3.2 to 6.7] | 5.5 [3.9 to 7.7] | 5.9 [4.6 to 7.5] | 4.6 [3.4 to 6.3]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) | 2.8 [1.7 to 4.5] | 2.8 [1.6 to 4.8] | 2.7 [1.6 to 4.3] | 2.3 [1.6 to 3.3] | 3.5 [2.4 to 5.3] | 2.8 [1.9 to 4.2]
  A/Michigan/45/2015 X-275 (H1N1) | 1.8 [1.1 to 2.8] | 1.9 [1.1 to 3.3] | 2.2 [1.3 to 3.6] | 2.1 [1.6 to 2.8] | 4.2 [2.4 to 7.2] | 2.1 [1.4 to 3.2]
  B/Phuket/3073/2013 (B Yamagata lineage) | 2.4 [1.6 to 3.6] | 2.4 [1.6 to 3.6] | 1.9 [1.4 to 2.6] | 2.4 [1.7 to 3.4] | 3.4 [2.0 to 5.5] | 2.3 [1.7 to 3.3]

19. Secondary Outcome: Number of Participants Reporting Protocol Specified Adverse Events of Special Interest (AESIs)
Description: Participants were queried at each visit for the occurrence of adverse events of special interest (AESIs) through approximately 12 months following the first study vaccination. AESIs include reports of tearing, dry mouth, and dry eyes.
Time Frame: Day 1 through Day 365
Population: The Safety Analysis population includes all participants who received study vaccination. Analyses for the safety population are based on vaccine actually received. One participant randomized to Flublok + AF03 group received Flublok due to a pharmacy error and is analyzed in the Flublok group.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 42 | 37 | 43
Participants | 0 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Participants Reporting Medically-Attended Adverse Events (MAAEs), New-Onset Chronic Medical Conditions (NOCMCs), and Potentially Immune-Mediated Medical Conditions (PIMMCs)
Description: Participants were queried at each visit for the occurrence of medically-attended adverse events (MAAEs), including new-onset chronic medical conditions (NOCMCs) and potentially immune-mediated medical conditions (PIMMCs) through approximately 12 months following the first study vaccination.
Time Frame: Day 1 through Day 365
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 42 | 37 | 43
Participants
  MAAEs | 9 | 13 | 7 | 8 | 7 | 10
  NOCMCs | 1 | 0 | 0 | 1 | 1 | 0
  PIMMCs | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Hemagglutination Inhibition (HAI) Against the 2019/2020 Quadrivalent Influenza Vaccine (QIV) Strains
Description: Blood was collected for HAI assay which was conducted with the 2019/2020 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at Day 90 and Day 118 post first study vaccination.
Time Frame: Day 90 through Day 118
Population: The modified intent-to-treat (mITT) population includes all randomized participants who received the first study vaccination and contributed at least one post-first study vaccination venous blood samples for immunogenicity testing (HAI, NAI or Neut antibody assays) for which valid HAI results were reported. For analyses using the mITT population, participants were grouped based on randomized study arm.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 41 | 38 | 42
titer
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 90 | 325.5 [242.9 to 436.0] | 326.2 [237.6 to 447.9] | 234.7 [157.8 to 349.1] | 456.6 [314.7 to 662.4] | 408.2 [278.0 to 599.4] | 355.1 [246.5 to 511.4]
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 118 | 387.9 [281.0 to 535.6] | 367.6 [254.7 to 530.6] | 269.1 [173.3 to 417.7] | 627.1 [430.9 to 912.7] | 509.8 [330.5 to 786.5] | 491.0 [343.5 to 701.9]
  A/Kansas/14/2017 (H3N2) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Kansas/14/2017 (H3N2) - Day 90 | 33.8 [23.2 to 49.2] | 67.9 [44.6 to 103.4] | 38.2 [25.8 to 56.6] | 69.4 [47.0 to 102.4] | 50.1 [32.5 to 77.2] | 62.2 [41.8 to 92.5]
  A/Kansas/14/2017 (H3N2) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Kansas/14/2017 (H3N2) - Day 118 | 203.5 [132.1 to 313.6] | 213.6 [136.9 to 333.1] | 274.6 [198.4 to 380.1] | 369.1 [238.5 to 571.2] | 254.9 [154.2 to 421.3] | 212.8 [135.9 to 333.5]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90 | 797.3 [595.9 to 1066.9] | 1129.4 [853.2 to 1495.2] | 849.1 [644.1 to 1119.4] | 1502.0 [1132.8 to 1991.7] | 1041.6 [747.5 to 1451.6] | 995.6 [752.0 to 1318.1]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118 | 665.1 [499.2 to 886.2] | 874.3 [647.1 to 1181.1] | 792.8 [615.8 to 1020.6] | 1228.9 [924.0 to 1634.4] | 905.1 [649.8 to 1260.7] | 1065.4 [836.2 to 1357.5]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90 | 312.0 [231.6 to 420.3] | 339.0 [241.2 to 476.5] | 245.6 [170.6 to 353.7] | 410.4 [270.4 to 622.8] | 323.0 [219.2 to 475.9] | 303.8 [215.8 to 427.6]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118 | 323.1 [235.1 to 443.9] | 281.8 [196.2 to 404.8] | 255.7 [170.6 to 383.3] | 404.5 [255.1 to 641.4] | 320.0 [224.4 to 456.3] | 329.9 [233.6 to 465.9]

22. Secondary Outcome: Ratio of Geometric Mean Titers (GMTs) of Serum Hemagglutination Inhibition (HAI) Against the 2019/2020 Quadrivalent Influenza Vaccine (QIV) Strains Between Adjuvanted and Unadjuvanted Study Arms
Description: Blood was collected for HAI assay which was conducted with the 2019/2020 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at Day 90 and Day 118 post first study vaccination and the ratio of these GMTs between adjuvanted and unadjuvanted study arms were calculated.
  Unadjuvanted Fluzone and Flublok study arms are considered as reference groups for the analysis of ratio of GMTs.
  Ratio of GMTs is defined as the ratio of the GMT from the adjuvanted group divided by the GMT from the corresponding unadjuvanted group.
Time Frame: Day 90 through Day 118
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: ratio of GMT
Arm/Group | Fluzone + AF03 | Fluzone + CpG55 | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 37 | 40 | 38 | 42
ratio of GMT
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 90: number analyzed (Participants) | 36 | 38 | 37 | 40
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 90 | 1.0 [0.7 to 1.5] | 0.7 [0.4 to 1.2] | 0.9 [0.5 to 1.5] | 0.8 [0.5 to 1.3]
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 118: number analyzed (Participants) | 30 | 34 | 32 | 34
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 118 | 0.9 [0.6 to 1.5] | 0.7 [0.4 to 1.2] | 0.8 [0.5 to 1.4] | 0.8 [0.5 to 1.3]
  A/Kansas/14/2017 (H3N2) - Day 90: number analyzed (Participants) | 36 | 38 | 37 | 40
  A/Kansas/14/2017 (H3N2) - Day 90 | 2.0 [1.2 to 3.5] | 1.1 [0.7 to 1.9] | 0.7 [0.4 to 1.3] | 0.9 [0.5 to 1.5]
  A/Kansas/14/2017 (H3N2) - Day 118: number analyzed (Participants) | 30 | 34 | 32 | 34
  A/Kansas/14/2017 (H3N2) - Day 118 | 1.0 [0.6 to 1.9] | 1.3 [0.8 to 2.3] | 0.7 [0.4 to 1.3] | 0.6 [0.3 to 1.1]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90: number analyzed (Participants) | 36 | 38 | 37 | 40
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90 | 1.4 [1.0 to 2.1] | 1.1 [0.7 to 1.6] | 0.7 [0.5 to 1.1] | 0.7 [0.4 to 1.0]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118: number analyzed (Participants) | 30 | 34 | 32 | 34
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118 | 1.3 [0.9 to 2.0] | 1.2 [0.8 to 1.7] | 0.7 [0.5 to 1.1] | 0.9 [0.6 to 1.3]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90: number analyzed (Participants) | 36 | 38 | 37 | 40
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90 | 1.1 [0.7 to 1.7] | 0.8 [0.5 to 1.3] | 0.8 [0.4 to 1.4] | 0.7 [0.4 to 1.3]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118: number analyzed (Participants) | 30 | 34 | 32 | 34
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118 | 0.9 [0.5 to 1.4] | 0.8 [0.5 to 1.3] | 0.8 [0.4 to 1.4] | 0.8 [0.5 to 1.4]

23. Secondary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Titer Seroconversion Against 2019/2020 Quadrivalent Influenza Vaccine (QIV) Strains
Description: Blood was collected for HAI assay which was conducted with the 2019/2020 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. HAI seroconversion was defined as either a pre-second vaccination titer < 1:10 and a post- second vaccination titer >= 1:40 or a pre-second vaccination titer >= 1:10 and a minimum four-fold rise in post-vaccination antibody titer.
Time Frame: Day 118
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
percentage of participants
  A/Brisbane/02/2018 IVR-190 (H1N1) | 0 [0 to 10] | 0 [0 to 12] | 0 [0 to 10] | 6 [NA to 20] — Value is NA because it is >0 but <1 | 0 [0 to 11] | 6 [NA to 20] — Value is NA because it is >0 but <1
  A/Kansas/14/2017 (H3N2) | 67 [49 to 81] | 43 [25 to 63] | 74 [56 to 87] | 56 [38 to 73] | 53 [35 to 71] | 53 [35 to 70]
  B/Phuket/3073/2013 (B Yamagata lineage) | 0 [0 to 10] | 0 [0 to 12] | 0 [0 to 10] | 0 [0 to 10] | 0 [0 to 11] | 0 [0 to 10]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) | 0 [0 to 10] | 0 [0 to 12] | 0 [0 to 10] | 0 [0 to 10] | 0 [0 to 11] | 0 [0 to 10]

24. Secondary Outcome: Percentage of Participants With Hemagglutination Inhibition (HAI) Titer of 1:40 or Greater Against the 2019/2020 Quadrivalent Influenza Vaccine (QIV) Strains
Description: Blood was collected for HAI assay which was conducted with the 2019/2020 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result.
Time Frame: Day 90 through Day 118
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 41 | 38 | 42
percentage of participants
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 90 | 100 [91 to 100] | 100 [90 to 100] | 92 [79 to 98] | 95 [83 to NA] — Value is NA because it is >99 but <100 | 95 [82 to NA] — Value is NA because it is >99 but <100 | 95 [83 to NA] — Value is NA because it is >99 but <100
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 118 | 100 [90 to 100] | 100 [88 to 100] | 91 [76 to 98] | 97 [85 to NA] — Value is NA because it is >99 but <100 | 97 [84 to NA] — Value is NA because it is >99 but <100 | 97 [85 to NA] — Value is NA because it is >99 but <100
  A/Kansas/14/2017 (H3N2) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Kansas/14/2017 (H3N2) - Day 90 | 41 [26 to 58] | 67 [49 to 81] | 50 [33 to 67] | 77 [61 to 89] | 59 [42 to 75] | 73 [56 to 85]
  A/Kansas/14/2017 (H3N2) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Kansas/14/2017 (H3N2) - Day 118 | 92 [78 to 98] | 93 [78 to NA] — Value is NA because it is >99 but <100 | 94 [80 to NA] — Value is NA because it is >99 but <100 | 100 [90 to 100] | 91 [75 to 98] | 94 [80 to NA] — Value is NA because it is >99 but <100
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90 | 100 [91 to 100] | 100 [90 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118 | 100 [90 to 100] | 100 [88 to 100] | 100 [90 to 100] | 100 [90 to 100] | 100 [89 to 100] | 100 [90 to 100]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90 | 98 [87 to NA] — Value is NA because it is >99 but <100 | 100 [90 to 100] | 97 [86 to NA] — Value is NA because it is >99 but <100 | 97 [87 to NA] — Value is NA because it is >99 but <100 | 97 [86 to NA] — Value is NA because it is >99 but <100 | 100 [91 to 100]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118 | 100 [90 to 100] | 100 [88 to 100] | 97 [85 to NA] — Value is NA because it is >99 but <100 | 100 [90 to 100] | 94 [79 to NA] — Value is NA because it is >99 but <100 | 100 [90 to 100]

25. Secondary Outcome: Geometric Mean Fold Rise in Hemagglutination Inhibition (HAI) Titers Against the 2019/2020 Quadrivalent Influenza Vaccine (QIV) Strains
Description: Blood was collected for HAI assay which was conducted with the 2019/2020 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. Fold-rises at Day 118 were calculated as the Day 118 titer divided by the Day 90 titers for each participant. The geometric mean of these fold rises was then calculated to obtain the GMFR.
Time Frame: Day 90 through Day 118
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 41 | 38 | 42
fold rise
  A/Brisbane/02/2018 IVR-190 (H1N1): number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Brisbane/02/2018 IVR-190 (H1N1) | 1.1 [1.0 to 1.2] | 1.1 [1.0 to 1.2] | 1.2 [1.1 to 1.4] | 1.3 [1.1 to 1.6] | 1.3 [1.1 to 1.4] | 1.4 [1.2 to 1.7]
  A/Kansas/14/2017 (H3N2): number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Kansas/14/2017 (H3N2) | 7.1 [4.8 to 10.6] | 3.3 [2.3 to 4.6] | 6.9 [4.7 to 10.0] | 5.4 [3.4 to 8.4] | 5.5 [3.4 to 8.7] | 3.6 [2.7 to 4.9]
  B/Phuket/3073/2013 (B Yamagata lineage): number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  B/Phuket/3073/2013 (B Yamagata lineage) | 0.8 [0.8 to 0.9] | 0.8 [0.7 to 0.9] | 1.0 [0.8 to 1.1] | 0.8 [0.7 to 1.0] | 0.9 [0.8 to 1.0] | 1.1 [0.9 to 1.3]
  B/Maryland/15/2016 BX-69A (B Victoria lineage): number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  B/Maryland/15/2016 BX-69A (B Victoria lineage) | 1.1 [0.9 to 1.2] | 0.9 [0.8 to 1.0] | 1.0 [0.9 to 1.2] | 1.0 [0.9 to 1.1] | 1.0 [0.9 to 1.2] | 1.1 [1.0 to 1.3]

26. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Neuraminidase Inhibition (NAI) Against the 2019/2020 Quadrivalent Influenza Vaccine (QIV) Strains for the Fluzone Study Arms
Description: Blood was collected for NAI assay which was conducted with the 2019/2020 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at Day 90 and Day 118 post first study vaccination.
Time Frame: Day 90 through Day 118
Population: The modified intent-to-treat (mITT) population includes all randomized participants who received the first study vaccination and contributed at least one post-first study vaccination venous blood samples for immunogenicity testing (HAI, NAI or Neut antibody assays) for which valid NAI results were reported. For analyses using the mITT population, participants were grouped based on randomized study arm.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55
Number analyzed (Participants) | 41 | 37 | 40
titer
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 90 | 90.1 [65.0 to 124.8] | 91.5 [65.8 to 127.3] | 72.4 [50.1 to 104.5]
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 118 | 107.8 [76.8 to 151.3] | 111.8 [79.4 to 157.5] | 79.2 [55.6 to 112.7]
  A/Kansas/14/2017 (H3N2) - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Kansas/14/2017 (H3N2) - Day 90 | 35.8 [28.9 to 44.5] | 49.0 [38.6 to 62.1] | 36.5 [28.1 to 47.5]
  A/Kansas/14/2017 (H3N2) - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Kansas/14/2017 (H3N2) - Day 118 | 48.5 [38.2 to 61.6] | 51.0 [41.0 to 63.4] | 45.7 [34.8 to 59.9]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90 | 104.0 [86.2 to 125.4] | 156.9 [120.1 to 205.0] | 137.0 [113.1 to 166.1]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118 | 115.3 [97.5 to 136.4] | 158.2 [117.3 to 213.3] | 150.5 [120.1 to 188.6]
  B/Colorado/06/2017 (B Victoria lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38
  B/Colorado/06/2017 (B Victoria lineage) - Day 90 | 286.7 [241.4 to 340.5] | 391.7 [285.8 to 536.8] | 294.8 [234.2 to 371.0]
  B/Colorado/06/2017 (B Victoria lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34
  B/Colorado/06/2017 (B Victoria lineage) - Day 118 | 373.3 [305.9 to 455.5] | 474.0 [351.9 to 638.3] | 400.4 [313.3 to 511.8]

27. Secondary Outcome: Ratio of Geometric Mean Titers (GMTs) of Serum Neuraminidase Inhibition (NAI) Against the 2019/2020 Quadrivalent Influenza Vaccine (QIV) Strains Between Adjuvanted and Unadjuvanted Study Arms for the Fluzone Study Arms
Description: Blood was collected for NAI assay which was conducted with the 2019/2020 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at Day 90 and Day 118 post first study vaccination and the ratio of these GMTs between adjuvanted and unadjuvanted study arms were calculated.
  The unadjuvanted Fluzone study arm is considered a reference group for the analysis of ratio of GMTs.
  Ratio of GMTs is defined as the ratio of the GMT from the adjuvanted group divided by the GMT from the corresponding unadjuvanted group.
Time Frame: Day 90 through Day 118
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: ratio of GMT
Arm/Group | Fluzone + AF03 | Fluzone + CpG55
Number analyzed (Participants) | 37 | 40
ratio of GMT
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 90: number analyzed (Participants) | 36 | 38
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 90 | 1.0 [0.6 to 1.6] | 0.8 [0.5 to 1.3]
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 118: number analyzed (Participants) | 30 | 34
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 118 | 1.0 [0.6 to 1.7] | 0.7 [0.5 to 1.2]
  A/Kansas/14/2017 (H3N2) - Day 90: number analyzed (Participants) | 36 | 38
  A/Kansas/14/2017 (H3N2) - Day 90 | 1.4 [1.0 to 1.9] | 1.0 [0.7 to 1.4]
  A/Kansas/14/2017 (H3N2) - Day 118: number analyzed (Participants) | 30 | 34
  A/Kansas/14/2017 (H3N2) - Day 118 | 1.1 [0.8 to 1.4] | 0.9 [0.7 to 1.3]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90: number analyzed (Participants) | 36 | 38
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90 | 1.5 [1.1 to 2.1] | 1.3 [1.0 to 1.7]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118: number analyzed (Participants) | 30 | 34
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118 | 1.4 [1.0 to 1.9] | 1.3 [1.0 to 1.7]
  B/Colorado/06/2017 (B Victoria lineage) - Day 90: number analyzed (Participants) | 36 | 38
  B/Colorado/06/2017 (B Victoria lineage) - Day 90 | 1.4 [1.0 to 1.9] | 1.0 [0.8 to 1.4]
  B/Colorado/06/2017 (B Victoria lineage) - Day 118: number analyzed (Participants) | 30 | 34
  B/Colorado/06/2017 (B Victoria lineage) - Day 118 | 1.3 [0.9 to 1.8] | 1.1 [0.8 to 1.5]

28. Secondary Outcome: Percentage of Participants Achieving Neuraminidase Inhibition (NAI) Titer Seroconversion Against 2019/2020 Quadrivalent Influenza Vaccine (QIV) Strains for the Fluzone Study Arms
Description: Blood was collected for NAI assay which was conducted with the 2019/2020 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. NAI seroconversion was defined as >4 four-fold rise in post-vaccination antibody titer at Day 90 through Day 118.
Time Frame: Day 118
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55
Number analyzed (Participants) | 36 | 30 | 34
percentage of participants
  A/Brisbane/02/2018 IVR-190 (H1N1) | 6 [NA to 19] — Value is NA because it is >0 but <1 | 0 [0 to 12] | 0 [0 to 10]
  A/Kansas/14/2017 (H3N2) | 8 [2 to 22] | 0 [0 to 12] | 0 [0 to 10]
  B/Phuket/3073/2013 (B Yamagata lineage) | 3 [NA to 15] — Value is NA because it is >0 but <1 | 0 [0 to 12] | 0 [0 to 10]
  B/Colorado/06/2017 (B Victoria lineage) | 8 [2 to 22] | 0 [0 to 12] | 0 [0 to 10]

29. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in Neuraminidase Inhibition (NAI) Titers Against the 2019/2020 Quadrivalent Influenza Vaccine (QIV) Strains for the Fluzone Study Arms
Description: Blood was collected for NAI assay which was conducted with the 2019/2020 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. Fold-rises at Day 118 were calculated as the Day 118 titer divided by the Day 90 titers for each participant. The geometric mean of these fold rises was then calculated to obtain the GMFR.
Time Frame: Day 118
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55
Number analyzed (Participants) | 36 | 30 | 34
Fold Rise
  A/Brisbane/02/2018 IVR-190 (H1N1) | 1.3 [1.1 to 1.5] | 1.2 [1.0 to 1.3] | 1.2 [1.1 to 1.4]
  A/Kansas/14/2017 (H3N2) | 1.4 [1.2 to 1.7] | 1.1 [1.0 to 1.2] | 1.3 [1.1 to 1.5]
  B/Phuket/3073/2013 (B Yamagata lineage) | 1.2 [1.0 to 1.3] | 1.0 [0.9 to 1.2] | 1.1 [1.0 to 1.2]
  B/Colorado/06/2017 (B Victoria lineage) | 1.3 [1.2 to 1.6] | 1.3 [1.2 to 1.5] | 1.3 [1.2 to 1.5]

30. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Neutralizing (Neut) Titers Against the 2019/2020 Quadrivalent Influenza Vaccine (QIV) Strains
Description: Blood was collected for Neut assay which was conducted with the 2019/2020 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, but only one result which a geometric mean titer of the replicates was reported by the lab. The geometric mean titer was calculated for each study arm from the available results at Day 90 and Day 118 post first study vaccination.
Time Frame: Day 90 through Day 118
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 41 | 38 | 42
titer
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 90 | 3375.3 [2416.0 to 4715.5] | 3727.3 [2736.7 to 5076.5] | 2488.0 [1582.9 to 3910.7] | 4850.2 [3042.7 to 7731.4] | 5622.8 [3362.1 to 9403.6] | 3899.5 [2623.1 to 5796.9]
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 118 | 3891.7 [2737.9 to 5531.8] | 3613.3 [2494.4 to 5234.0] | 2895.1 [1881.9 to 4453.8] | 6618.8 [4313.1 to 10157.2] | 5654.7 [3513.2 to 9101.6] | 4983.6 [3408.9 to 7285.6]
  A/Kansas/14/2017 (H3N2) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Kansas/14/2017 (H3N2) - Day 90 | 50.7 [41.0 to 62.5] | 81.4 [63.0 to 105.3] | 57.2 [45.0 to 72.7] | 90.7 [65.0 to 126.7] | 72.3 [56.8 to 92.2] | 79.1 [60.9 to 102.8]
  A/Kansas/14/2017 (H3N2) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Kansas/14/2017 (H3N2) - Day 118 | 238.1 [164.2 to 345.2] | 198.0 [140.0 to 280.2] | 225.6 [173.2 to 293.9] | 396.6 [262.7 to 598.7] | 266.5 [178.4 to 398.2] | 251.9 [168.1 to 377.3]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90 | 681.0 [490.3 to 945.9] | 909.3 [638.8 to 1294.5] | 766.9 [541.3 to 1086.4] | 1371.5 [981.9 to 1915.7] | 953.5 [638.6 to 1423.7] | 754.8 [533.9 to 1066.9]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118 | 1087.2 [762.1 to 1551.2] | 1031.7 [703.9 to 1512.2] | 1086.9 [798.5 to 1479.6] | 1920.9 [1351.2 to 2730.8] | 1234.9 [710.6 to 2146.0] | 1284.8 [914.5 to 1805.0]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90 | 255.4 [173.2 to 376.7] | 235.4 [164.9 to 335.9] | 178.3 [110.1 to 288.7] | 362.6 [208.1 to 632.0] | 234.1 [140.7 to 389.6] | 232.4 [151.2 to 357.3]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118 | 202.2 [127.2 to 321.4] | 180.7 [113.0 to 288.9] | 151.5 [85.9 to 267.2] | 312.0 [160.1 to 607.8] | 212.1 [127.1 to 354.2] | 211.7 [136.9 to 327.2]

31. Secondary Outcome: Ratio of Serum Neutralizing (Neut) Geometric Mean Titers (GMT) Against the 2019/2020 Quadrivalent Influenza Vaccine (QIV) Strains Between Adjuvanted and Unadjuvanted Study Arms
Description: Blood was collected for Neut assay which was conducted with the 2019/2020 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, but only one result which a geometric mean titer of the replicates was reported by the lab. The geometric mean titer was calculated for each study arm from the available results at Day 90 and Day 118 post first study vaccination and the ratio of these GMTs between adjuvanted and unadjuvanted study arms were calculated.
  Unadjuvanted Fluzone and Flublok study arms are considered as reference groups for the analysis of ratio of GMTs.
  Ratio of GMTs is defined as the ratio of the GMT from the adjuvanted group divided by the GMT from the corresponding unadjuvanted group.
Time Frame: Day 90 through Day 118
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: ratio of GMT
Arm/Group | Fluzone + AF03 | Fluzone + CpG55 | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 37 | 40 | 38 | 42
ratio of GMT
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 90: number analyzed (Participants) | 36 | 38 | 37 | 40
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 90 | 1.1 [0.7 to 1.7] | 0.7 [0.4 to 1.3] | 1.2 [0.6 to 2.3] | 0.8 [0.4 to 1.5]
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 118: number analyzed (Participants) | 30 | 34 | 32 | 34
  A/Brisbane/02/2018 IVR-190 (H1N1) - Day 118 | 0.9 [0.6 to 1.5] | 0.7 [0.4 to 1.3] | 0.9 [0.5 to 1.6] | 0.8 [0.4 to 1.3]
  A/Kansas/14/2017 (H3N2) - Day 90: number analyzed (Participants) | 36 | 38 | 37 | 40
  A/Kansas/14/2017 (H3N2) - Day 90 | 1.6 [1.2 to 2.2] | 1.1 [0.8 to 1.5] | 0.8 [0.5 to 1.2] | 0.9 [0.6 to 1.3]
  A/Kansas/14/2017 (H3N2) - Day 118: number analyzed (Participants) | 30 | 34 | 32 | 34
  A/Kansas/14/2017 (H3N2) - Day 118 | 0.8 [0.5 to 1.4] | 0.9 [0.6 to 1.5] | 0.7 [0.4 to 1.2] | 0.6 [0.4 to 1.1]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90: number analyzed (Participants) | 36 | 38 | 37 | 40
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90 | 1.3 [0.8 to 2.1] | 1.1 [0.7 to 1.8] | 0.7 [0.4 to 1.2] | 0.6 [0.3 to 0.9]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118: number analyzed (Participants) | 30 | 34 | 32 | 34
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118 | 0.9 [0.6 to 1.6] | 1.0 [0.6 to 1.6] | 0.6 [0.3 to 1.2] | 0.7 [0.4 to 1.1]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90: number analyzed (Participants) | 36 | 38 | 37 | 40
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90 | 0.9 [0.5 to 1.5] | 0.7 [0.4 to 1.3] | 0.6 [0.3 to 1.4] | 0.6 [0.3 to 1.3]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118: number analyzed (Participants) | 30 | 34 | 32 | 34
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118 | 0.9 [0.5 to 1.7] | 0.7 [0.4 to 1.5] | 0.7 [0.3 to 1.6] | 0.7 [0.3 to 1.5]

32. Secondary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Titer Seroconversion Against 2019/2020 Quadrivalent Influenza Vaccine (QIV) Strains
Description: Blood was collected for Neut assay which was conducted with the 2019/2020 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, but only one result which a geometric mean titer of the replicates was reported by the lab. Neut seroconversion was defined as either a pre-second vaccination titer < 1:10 and a post-second vaccination titer >= 1:40 or a pre-second vaccination titer >= 1:10 and a minimum four-fold rise in post-vaccination antibody titer.
Time Frame: Day 118
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
percentage of participants
  A/Brisbane/02/2018 IVR-190 (H1N1) | 0 [0 to 10] | 0 [0 to 12] | 0 [0 to 10] | 9 [2 to 24] | 6 [NA to 21] — Value is NA because it is >0 but <1 | 3 [NA to 15] — Value is NA because it is >0 but <1
  A/Kansas/14/2017 (H3N2) | 58 [41 to 74] | 30 [15 to 49] | 44 [27 to 62] | 56 [38 to 73] | 38 [21 to 56] | 26 [13 to 44]
  B/Phuket/3073/2013 (B Yamagata lineage) | 8 [2 to 22] | 3 [NA to 17] — Value is NA because it is >0 but <1 | 3 [NA to 15] — Value is NA because it is >0 but <1 | 0 [0 to 10] | 9 [2 to 25] | 12 [3 to 27]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) | 3 [NA to 15] — Value is NA because it is >0 but <1 | 0 [0 to 12] | 0 [0 to 10] | 0 [0 to 10] | 0 [0 to 11] | 0 [0 to 10]

33. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in Neutralizing (Neut) Titers Against the 2019/2020 Quadrivalent Influenza Vaccine (QIV) Strains
Description: Blood was collected for Neut assay which was conducted with the 2019/2020 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, but only one result which a geometric mean titer of the replicates was reported by the lab. Fold-rises at Day 118 were calculated as the Day 118 titer divided by the Day 90 titers for each participant. The geometric mean of these fold rises was then calculated to obtain the GMFR.
Time Frame: Day 118
Population: as for outcome 18
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
Fold Rise
  A/Brisbane/02/2018 IVR-190 (H1N1) | 1.0 [0.9 to 1.2] | 1.0 [0.8 to 1.2] | 1.3 [1.1 to 1.5] | 1.4 [1.0 to 1.9] | 1.1 [0.8 to 1.4] | 1.3 [1.1 to 1.6]
  A/Kansas/14/2017 (H3N2) | 5.1 [3.7 to 6.9] | 2.5 [1.9 to 3.3] | 3.9 [2.9 to 5.2] | 4.5 [2.9 to 7.0] | 3.9 [2.7 to 5.6] | 3.1 [2.3 to 4.3]
  B/Phuket/3073/2013 (B Yamagata lineage) | 1.7 [1.3 to 2.2] | 1.2 [0.9 to 1.6] | 1.5 [1.2 to 1.7] | 1.5 [1.3 to 1.8] | 1.3 [0.9 to 1.8] | 1.7 [1.4 to 2.0]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) | 0.8 [0.7 to 0.9] | 0.9 [0.7 to 1.0] | 0.9 [0.7 to 1.0] | 0.9 [0.7 to 1.0] | 0.9 [0.8 to 1.1] | 0.9 [0.8 to 1.1]

34. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Hemagglutination Inhibition (HAI) Against the 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains
Description: Blood was collected for HAI assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at Day 8, Day 57, Day 90, and Day 118 Post first study vaccination.
Time Frame: Day 8, Day 57, Day 90, Day 118
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 41 | 38 | 42
titer
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 8 | 296.6 [215.3 to 408.5] | 582.8 [421.4 to 805.9] | 343.0 [256.2 to 459.2] | 398.7 [294.9 to 538.8] | 469.4 [314.4 to 700.6] | 347.5 [255.9 to 472.0]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57 | 248.9 [175.2 to 353.7] | 520.8 [386.2 to 702.3] | 266.6 [184.4 to 385.5] | 602.3 [451.0 to 804.5] | 506.4 [354.6 to 723.1] | 408.9 [301.2 to 555.1]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90 | 224.4 [162.3 to 310.2] | 456.9 [338.1 to 617.5] | 245.6 [169.1 to 356.7] | 565.1 [426.9 to 748.2] | 444.1 [314.1 to 628.1] | 383.9 [272.1 to 541.5]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118 | 320.0 [224.7 to 455.7] | 570.2 [409.2 to 794.5] | 404.5 [264.2 to 619.4] | 962.2 [698.8 to 1324.9] | 839.0 [585.3 to 1202.7] | 554.9 [356.8 to 863.0]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 8 | 441.2 [335.5 to 580.2] | 525.7 [389.4 to 709.8] | 400.9 [290.8 to 552.6] | 480.1 [333.2 to 691.8] | 402.0 [278.4 to 580.3] | 344.7 [247.1 to 480.7]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 57 | 322.8 [241.0 to 432.3] | 338.5 [243.7 to 470.2] | 254.8 [177.6 to 365.3] | 422.2 [285.7 to 624.0] | 311.1 [216.9 to 446.3] | 286.7 [201.2 to 408.5]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90 | 312.0 [231.6 to 420.3] | 339.0 [241.2 to 476.5] | 245.6 [170.6 to 353.7] | 410.4 [270.4 to 622.8] | 323.0 [219.2 to 475.9] | 303.8 [215.8 to 427.6]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118 | 323.1 [235.1 to 443.9] | 281.8 [196.2 to 404.8] | 255.7 [170.6 to 383.3] | 404.5 [255.1 to 641.4] | 320.0 [224.4 to 456.3] | 329.9 [233.6 to 465.9]
  A/Michigan/45/2015 X-275 (H1N1) - Day 8 | 603.2 [442.7 to 821.9] | 561.3 [409.9 to 768.8] | 472.6 [340.3 to 656.3] | 673.3 [476.6 to 951.2] | 701.1 [471.8 to 1041.9] | 542.6 [382.1 to 770.6]
  A/Michigan/45/2015 X-275 (H1N1) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Michigan/45/2015 X-275 (H1N1) - Day 57 | 629.0 [472.5 to 837.4] | 582.8 [431.6 to 787.0] | 440.3 [305.5 to 634.6] | 897.3 [648.4 to 1241.7] | 771.9 [527.9 to 1128.6] | 645.4 [460.9 to 903.8]
  A/Michigan/45/2015 X-275 (H1N1) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Michigan/45/2015 X-275 (H1N1) - Day 90 | 526.9 [390.9 to 710.3] | 548.6 [401.8 to 749.1] | 366.9 [252.9 to 532.4] | 757.7 [550.4 to 1043.2] | 689.8 [476.7 to 998.2] | 571.8 [401.5 to 814.3]
  A/Michigan/45/2015 X-275 (H1N1) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Michigan/45/2015 X-275 (H1N1) - Day 118 | 586.9 [436.0 to 790.0] | 519.8 [351.0 to 770.0] | 361.6 [242.1 to 540.3] | 868.9 [610.4 to 1237.0] | 697.9 [457.5 to 1064.6] | 715.9 [502.3 to 1020.4]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 8 | 714.3 [553.7 to 921.6] | 1061.3 [844.2 to 1334.2] | 889.5 [727.8 to 1087.3] | 1045.0 [801.2 to 1363.0] | 1019.0 [794.5 to 1306.9] | 875.7 [690.0 to 1111.4]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57 | 629.0 [478.4 to 827.1] | 905.1 [688.4 to 1190.1] | 740.6 [584.7 to 938.0] | 1133.8 [887.1 to 1449.1] | 839.8 [617.7 to 1141.6] | 817.8 [638.6 to 1047.3]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90 | 797.3 [595.9 to 1066.9] | 1129.4 [853.2 to 1495.2] | 849.1 [644.1 to 1119.4] | 1502.0 [1132.8 to 1991.7] | 1041.6 [747.5 to 1451.6] | 995.6 [752.0 to 1318.1]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118 | 665.1 [499.2 to 886.2] | 874.3 [647.1 to 1181.1] | 792.8 [615.8 to 1020.6] | 1228.9 [924.0 to 1634.4] | 905.1 [649.8 to 1260.7] | 1065.4 [836.2 to 1357.5]

35. Secondary Outcome: Ratio of Geometric Mean Titers (GMTs) of Serum Hemagglutination Inhibition (HAI) Against the 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains Between Adjuvanted and Unadjuvanted Study Arms
Description: Blood was collected for HAI assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at Day 8, Day 57, Day 90, and Day 118 Post first study vaccination and the ratio of these GMTs between adjuvanted and unadjuvanted study arms were calculated.
  Unadjuvanted Fluzone and Flublok study arms are considered as reference groups for the analysis of ratio of GMTs.
  Ratio of GMTs is defined as the ratio of the GMT from the adjuvanted group divided by the GMT from the corresponding unadjuvanted group.
Time Frame: Day 8, Day 57, Day 90, Day 118
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: ratio of GMT
Arm/Group | Fluzone + AF03 | Fluzone + CpG55 | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 37 | 40 | 38 | 42
ratio of GMT
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 8 | 2.0 [1.3 to 3.1] | 1.2 [0.8 to 1.8] | 1.2 [0.7 to 1.9] | 0.9 [0.6 to 1.3]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57: number analyzed (Participants) | 37 | 38 | 37 | 41
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57 | 2.1 [1.3 to 3.3] | 1.1 [0.6 to 1.8] | 0.8 [0.5 to 1.3] | 0.7 [0.4 to 1.0]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90: number analyzed (Participants) | 36 | 38 | 37 | 40
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90 | 2.0 [1.3 to 3.1] | 1.1 [0.7 to 1.8] | 0.8 [0.5 to 1.2] | 0.7 [0.4 to 1.1]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118: number analyzed (Participants) | 30 | 34 | 32 | 34
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118 | 1.8 [1.1 to 2.9] | 1.3 [0.7 to 2.2] | 0.9 [0.5 to 1.4] | 0.6 [0.3 to 1.0]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 8 | 1.2 [0.8 to 1.8] | 0.9 [0.6 to 1.4] | 0.8 [0.5 to 1.4] | 0.7 [0.4 to 1.2]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 57: number analyzed (Participants) | 37 | 38 | 37 | 41
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 57 | 1.0 [0.7 to 1.6] | 0.8 [0.5 to 1.2] | 0.7 [0.4 to 1.2] | 0.7 [0.4 to 1.1]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90: number analyzed (Participants) | 36 | 38 | 37 | 40
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90 | 1.1 [0.7 to 1.7] | 0.8 [0.5 to 1.3] | 0.8 [0.4 to 1.4] | 0.7 [0.4 to 1.3]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118: number analyzed (Participants) | 30 | 34 | 32 | 34
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118 | 0.9 [0.5 to 1.4] | 0.8 [0.5 to 1.3] | 0.8 [0.4 to 1.4] | 0.8 [0.5 to 1.4]
  A/Michigan/45/2015 X-275 (H1N1) - Day 8 | 0.9 [0.6 to 1.4] | 0.8 [0.5 to 1.2] | 1.0 [0.6 to 1.7] | 0.8 [0.5 to 1.3]
  A/Michigan/45/2015 X-275 (H1N1) - Day 57: number analyzed (Participants) | 37 | 38 | 37 | 41
  A/Michigan/45/2015 X-275 (H1N1) - Day 57 | 0.9 [0.6 to 1.4] | 0.7 [0.4 to 1.1] | 0.9 [0.5 to 1.4] | 0.7 [0.5 to 1.1]
  A/Michigan/45/2015 X-275 (H1N1) - Day 90: number analyzed (Participants) | 36 | 38 | 37 | 40
  A/Michigan/45/2015 X-275 (H1N1) - Day 90 | 1.0 [0.7 to 1.6] | 0.7 [0.4 to 1.1] | 0.9 [0.6 to 1.5] | 0.8 [0.5 to 1.2]
  A/Michigan/45/2015 X-275 (H1N1) - Day 118: number analyzed (Participants) | 30 | 34 | 32 | 34
  A/Michigan/45/2015 X-275 (H1N1) - Day 118 | 0.9 [0.5 to 1.4] | 0.6 [0.4 to 1.0] | 0.8 [0.5 to 1.4] | 0.8 [0.5 to 1.3]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 8 | 1.5 [1.1 to 2.1] | 1.2 [0.9 to 1.7] | 1.0 [0.7 to 1.4] | 0.8 [0.6 to 1.2]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57: number analyzed (Participants) | 37 | 38 | 37 | 41
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57 | 1.4 [1.0 to 2.1] | 1.2 [0.8 to 1.7] | 0.7 [0.5 to 1.1] | 0.7 [0.5 to 1.0]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90: number analyzed (Participants) | 36 | 38 | 37 | 40
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90 | 1.4 [1.0 to 2.1] | 1.1 [0.7 to 1.6] | 0.7 [0.5 to 1.1] | 0.7 [0.4 to 1.0]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118: number analyzed (Participants) | 30 | 34 | 32 | 34
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118 | 1.3 [0.9 to 2.0] | 1.2 [0.8 to 1.7] | 0.7 [0.5 to 1.1] | 0.9 [0.6 to 1.3]

36. Secondary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Titer Seroconversion Against 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains
Description: as for outcome 7
Time Frame: Day 8, Day 57, Day 90, Day 118
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 41 | 38 | 42
percentage of participants
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 8 | 27 [14 to 43] | 35 [20 to 53] | 30 [17 to 47] | 29 [16 to 46] | 47 [31 to 64] | 43 [28 to 59]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57 | 25 [13 to 41] | 30 [16 to 47] | 32 [18 to 49] | 43 [27 to 59] | 54 [37 to 71] | 44 [28 to 60]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90 | 24 [12 to 40] | 25 [12 to 42] | 32 [18 to 49] | 41 [26 to 58] | 41 [25 to 58] | 43 [27 to 59]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118 | 42 [26 to 59] | 37 [20 to 56] | 50 [32 to 68] | 71 [53 to 85] | 72 [53 to 86] | 56 [38 to 73]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 8 | 27 [14 to 43] | 35 [20 to 53] | 35 [21 to 52] | 22 [11 to 38] | 47 [31 to 64] | 26 [14 to 42]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 57 | 20 [9 to 36] | 22 [10 to 38] | 24 [11 to 40] | 15 [6 to 30] | 35 [20 to 53] | 22 [11 to 38]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90 | 22 [11 to 38] | 22 [10 to 39] | 24 [11 to 40] | 15 [6 to 31] | 35 [20 to 53] | 23 [11 to 38]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118 | 22 [10 to 39] | 17 [6 to 35] | 26 [13 to 44] | 15 [5 to 31] | 31 [16 to 50] | 29 [15 to 47]
  A/Michigan/45/2015 X-275 (H1N1) - Day 8 | 22 [11 to 38] | 19 [8 to 35] | 23 [11 to 38] | 24 [12 to 40] | 39 [24 to 57] | 24 [12 to 39]
  A/Michigan/45/2015 X-275 (H1N1) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Michigan/45/2015 X-275 (H1N1) - Day 57 | 23 [11 to 38] | 24 [12 to 41] | 24 [11 to 40] | 33 [19 to 49] | 46 [29 to 63] | 24 [12 to 40]
  A/Michigan/45/2015 X-275 (H1N1) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Michigan/45/2015 X-275 (H1N1) - Day 90 | 20 [9 to 35] | 17 [6 to 33] | 16 [6 to 31] | 28 [15 to 45] | 38 [22 to 55] | 23 [11 to 38]
  A/Michigan/45/2015 X-275 (H1N1) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Michigan/45/2015 X-275 (H1N1) - Day 118 | 22 [10 to 39] | 10 [2 to 27] | 24 [11 to 41] | 32 [17 to 51] | 47 [29 to 65] | 44 [27 to 62]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 8 | 20 [9 to 35] | 16 [6 to 32] | 20 [9 to 36] | 12 [4 to 26] | 29 [15 to 46] | 21 [10 to 37]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57 | 15 [6 to 30] | 19 [8 to 35] | 16 [6 to 31] | 18 [7 to 33] | 30 [16 to 47] | 22 [11 to 38]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90 | 22 [11 to 38] | 14 [5 to 29] | 13 [4 to 28] | 26 [13 to 42] | 27 [14 to 44] | 30 [17 to 47]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118 | 17 [6 to 33] | 13 [4 to 31] | 15 [5 to 31] | 15 [5 to 31] | 16 [5 to 33] | 35 [20 to 54]

37. Secondary Outcome: Percentage of Participants With Hemagglutination Inhibition (HAI) Titer of 1:40 or Greater Against the 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains
Description: as for outcome 8
Time Frame: Day 8, Day 57, Day 90, Day 118
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 41 | 38 | 42
percentage of participants
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 8 | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 97 [86 to NA] — Value is NA because it's >99 but <100 | 100 [92 to 100]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57 | 100 [91 to 100] | 100 [91 to 100] | 97 [86 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90 | 98 [87 to NA] — Value is NA because it's >99 but <100 | 100 [90 to 100] | 97 [86 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 100 [91 to 100] | 98 [87 to NA] — Value is NA because it's >99 but <100
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118 | 100 [90 to 100] | 100 [88 to 100] | 97 [85 to NA] — Value is NA because it's >99 but <100 | 100 [90 to 100] | 100 [89 to 100] | 100 [90 to 100]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 8 | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 97 [86 to NA] — Value is NA because it's >99 but <100 | 100 [92 to 100]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 57 | 100 [91 to 100] | 100 [91 to 100] | 97 [86 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 97 [86 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90 | 98 [87 to NA] — Value is NA because it's >99 but <100 | 100 [90 to 100] | 97 [86 to NA] — Value is NA because it's >99 but <100 | 97 [87 to NA] — Value is NA because it's >99 but <100 | 97 [86 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118 | 100 [90 to 100] | 100 [88 to 100] | 97 [85 to NA] — Value is NA because it's >99 but <100 | 100 [90 to 100] | 94 [79 to NA] — Value is NA because it's >99 but <100 | 100 [90 to 100]
  A/Michigan/45/2015 X-275 (H1N1) - Day 8 | 100 [91 to 100] | 100 [91 to 100] | 98 [87 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 97 [86 to NA] — Value is NA because it's >99 but <100 | 98 [87 to NA] — Value is NA because it's >99 but <100
  A/Michigan/45/2015 X-275 (H1N1) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Michigan/45/2015 X-275 (H1N1) - Day 57 | 100 [91 to 100] | 100 [91 to 100] | 95 [82 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 97 [86 to NA] — Value is NA because it's >99 but <100 | 98 [87 to NA] — Value is NA because it's >99 but <100
  A/Michigan/45/2015 X-275 (H1N1) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Michigan/45/2015 X-275 (H1N1) - Day 90 | 100 [91 to 100] | 100 [90 to 100] | 95 [82 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 97 [86 to NA] — Value is NA because it's >99 but <100 | 98 [87 to NA] — Value is NA because it's >99 but <100
  A/Michigan/45/2015 X-275 (H1N1) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Michigan/45/2015 X-275 (H1N1) - Day 118 | 100 [90 to 100] | 100 [88 to 100] | 94 [80 to NA] — Value is NA because it's >99 but <100 | 100 [90 to 100] | 97 [84 to NA] — Value is NA because it's >99 but <100 | 100 [90 to 100]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 8 | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [92 to 100]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57 | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90 | 100 [91 to 100] | 100 [90 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118 | 100 [90 to 100] | 100 [88 to 100] | 100 [90 to 100] | 100 [90 to 100] | 100 [89 to 100] | 100 [90 to 100]

38. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in Hemagglutination Inhibition (HAI) Titers Against the 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains
Description: Blood was collected for HAI assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. Fold-rises from baseline were calculated as the Day 8 (or Day 57, Day 90, Day 118) titer divided by the baseline titers for each participant. The geometric mean of these fold rises was then calculated to obtain the GMFR.
Time Frame: Day 8, Day 57, Day 90, Day 118
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 41 | 38 | 42
fold rise
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 8 | 2.6 [1.7 to 3.9] | 3.0 [1.9 to 4.8] | 3.5 [2.1 to 5.9] | 2.4 [1.8 to 3.3] | 3.6 [2.6 to 5.1] | 3.2 [2.2 to 4.6]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57 | 2.2 [1.5 to 3.1] | 2.7 [1.8 to 4.0] | 3.0 [2.0 to 4.5] | 3.6 [2.5 to 5.2] | 3.8 [2.7 to 5.3] | 3.6 [2.5 to 5.0]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90 | 2.0 [1.4 to 2.7] | 2.2 [1.6 to 3.1] | 2.8 [1.9 to 4.1] | 3.4 [2.4 to 4.8] | 3.3 [2.4 to 4.6] | 3.3 [2.3 to 4.7]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118 | 3.1 [2.2 to 4.5] | 2.8 [2.0 to 3.9] | 5.0 [3.3 to 7.7] | 6.1 [4.2 to 8.8] | 6.7 [4.3 to 10.2] | 5.3 [3.7 to 7.7]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 8 | 3.1 [2.0 to 5.0] | 3.5 [2.4 to 5.2] | 3.3 [2.2 to 5.1] | 1.9 [1.5 to 2.5] | 3.8 [2.5 to 5.6] | 2.6 [1.9 to 3.6]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 57 | 2.2 [1.5 to 3.2] | 2.3 [1.5 to 3.3] | 2.2 [1.5 to 3.2] | 1.7 [1.3 to 2.2] | 2.8 [2.0 to 4.0] | 2.1 [1.6 to 2.8]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90 | 2.2 [1.5 to 3.3] | 2.4 [1.6 to 3.5] | 2.1 [1.5 to 2.9] | 1.7 [1.3 to 2.2] | 2.9 [2.1 to 4.1] | 2.3 [1.7 to 3.0]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118 | 2.3 [1.5 to 3.5] | 2.1 [1.4 to 3.2] | 2.3 [1.7 to 3.1] | 1.6 [1.3 to 2.2] | 2.9 [2.0 to 4.2] | 2.6 [1.9 to 3.7]
  A/Michigan/45/2015 X-275 (H1N1) - Day 8 | 2.5 [1.6 to 3.8] | 2.9 [1.9 to 4.4] | 2.7 [1.8 to 4.2] | 2.3 [1.7 to 3.0] | 3.8 [2.4 to 5.8] | 2.3 [1.7 to 3.1]
  A/Michigan/45/2015 X-275 (H1N1) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Michigan/45/2015 X-275 (H1N1) - Day 57 | 2.4 [1.7 to 3.5] | 3.0 [1.9 to 4.6] | 2.7 [1.9 to 3.9] | 2.8 [2.2 to 3.6] | 4.2 [2.9 to 6.3] | 2.6 [2.0 to 3.5]
  A/Michigan/45/2015 X-275 (H1N1) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Michigan/45/2015 X-275 (H1N1) - Day 90 | 2.2 [1.6 to 3.0] | 2.7 [1.8 to 4.1] | 2.3 [1.6 to 3.2] | 2.4 [1.9 to 3.0] | 3.8 [2.5 to 5.7] | 2.4 [1.8 to 3.0]
  A/Michigan/45/2015 X-275 (H1N1) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Michigan/45/2015 X-275 (H1N1) - Day 118 | 2.2 [1.5 to 3.2] | 2.2 [1.4 to 3.7] | 2.5 [1.8 to 3.6] | 2.7 [2.1 to 3.4] | 3.8 [2.5 to 5.7] | 3.0 [2.2 to 4.2]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 8 | 1.9 [1.4 to 2.8] | 2.2 [1.6 to 3.1] | 1.8 [1.4 to 2.3] | 1.7 [1.2 to 2.4] | 3.1 [2.0 to 4.8] | 2.2 [1.8 to 2.8]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57 | 1.7 [1.3 to 2.3] | 1.9 [1.3 to 2.8] | 1.5 [1.1 to 2.1] | 1.8 [1.3 to 2.5] | 2.5 [1.6 to 3.9] | 2.1 [1.6 to 2.7]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90 | 2.2 [1.7 to 2.8] | 2.2 [1.5 to 3.3] | 1.8 [1.4 to 2.3] | 2.5 [1.7 to 3.5] | 3.1 [2.0 to 4.7] | 2.5 [2.0 to 3.2]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118 | 1.8 [1.4 to 2.3] | 1.8 [1.1 to 2.7] | 1.8 [1.4 to 2.4] | 2.0 [1.4 to 2.9] | 2.6 [1.7 to 3.9] | 2.8 [2.2 to 3.5]

39. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Neuraminidase Inhibition (NAI) Against the 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains for the Fluzone Study Arms
Description: Blood was collected for NAI assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at Day 8, Day 57, Day 90, and Day 118 Post first study vaccination.
Time Frame: Day 8, Day 57, Day 90, Day 118
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: titer
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55
Number analyzed (Participants) | 41 | 37 | 40
titer
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 8 | 441.2 [330.9 to 588.3] | 501.7 [383.2 to 656.8] | 394.0 [291.6 to 532.3]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57: number analyzed (Participants) | 40 | 37 | 38
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57 | 262.2 [190.5 to 360.8] | 260.4 [195.3 to 347.2] | 202.8 [145.2 to 283.3]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90 | 201.0 [143.3 to 282.0] | 201.6 [145.0 to 280.2] | 148.7 [103.3 to 214.1]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118 | 258.9 [191.1 to 350.8] | 242.5 [170.2 to 345.5] | 200.2 [144.3 to 277.8]
  B/Colorado/06/2017 (B Victoria lineage) - Day 8 | 385.4 [306.3 to 484.9] | 566.6 [432.0 to 743.2] | 415.0 [326.7 to 527.1]
  B/Colorado/06/2017 (B Victoria lineage) - Day 57: number analyzed (Participants) | 40 | 37 | 38
  B/Colorado/06/2017 (B Victoria lineage) - Day 57 | 309.1 [261.3 to 365.6] | 427.8 [313.8 to 583.3] | 311.4 [243.8 to 397.7]
  B/Colorado/06/2017 (B Victoria lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38
  B/Colorado/06/2017 (B Victoria lineage) - Day 90 | 286.7 [241.4 to 340.5] | 391.7 [285.8 to 536.8] | 294.8 [234.2 to 371.0]
  B/Colorado/06/2017 (B Victoria lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34
  B/Colorado/06/2017 (B Victoria lineage) - Day 118 | 373.3 [305.9 to 455.5] | 474.0 [351.9 to 638.3] | 400.4 [313.3 to 511.8]
  A/Michigan/45/2015 X-275 (H1N1) - Day 8 | 398.7 [303.7 to 523.3] | 419.9 [318.0 to 554.4] | 352.0 [265.0 to 467.6]
  A/Michigan/45/2015 X-275 (H1N1) - Day 57: number analyzed (Participants) | 40 | 37 | 38
  A/Michigan/45/2015 X-275 (H1N1) - Day 57 | 218.6 [160.9 to 296.9] | 220.0 [161.6 to 299.5] | 155.7 [113.5 to 213.5]
  A/Michigan/45/2015 X-275 (H1N1) - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Michigan/45/2015 X-275 (H1N1) - Day 90 | 189.5 [139.3 to 257.7] | 176.2 [127.9 to 242.7] | 125.1 [89.7 to 174.5]
  A/Michigan/45/2015 X-275 (H1N1) - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Michigan/45/2015 X-275 (H1N1) - Day 118 | 261.4 [186.5 to 366.5] | 218.6 [156.0 to 306.2] | 177.2 [126.8 to 247.6]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 8 | 137.4 [111.7 to 169.1] | 208.0 [164.2 to 263.5] | 174.5 [143.5 to 212.2]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57: number analyzed (Participants) | 40 | 37 | 38
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57 | 117.1 [96.2 to 142.7] | 177.4 [140.3 to 224.1] | 157.1 [126.5 to 195.1]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90 | 104.0 [86.2 to 125.4] | 156.9 [120.1 to 205.0] | 137.0 [113.1 to 166.1]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118 | 115.3 [97.5 to 136.4] | 158.2 [117.3 to 213.3] | 150.5 [120.1 to 188.6]

40. Secondary Outcome: Ratio of Geometric Mean Titers (GMTs) of Serum Neuraminidase Inhibition (NAI) Against the 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains Between Adjuvanted and Unadjuvanted Study Arms for the Fluzone Study Arms
Description: Blood was collected for NAI assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at Day 8, Day 57, Day 90, and Day 118 Post first study vaccination and the ratio of these GMTs between adjuvanted and unadjuvanted study arms were calculated.
  The unadjuvanted Fluzone study arm is considered a reference group for the analysis of ratio of GMTs.
  Ratio of GMTs is defined as the ratio of the GMT from the adjuvanted group divided by the GMT from the corresponding unadjuvanted group.
Time Frame: Day 8, Day 57, Day 90, Day 118
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: ratio of GMT
Arm/Group | Fluzone + AF03 | Fluzone + CpG55
Number analyzed (Participants) | 37 | 40
ratio of GMT
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 8 | 1.1 [0.8 to 1.7] | 0.9 [0.6 to 1.3]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57: number analyzed (Participants) | 37 | 38
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57 | 1.0 [0.7 to 1.5] | 0.8 [0.5 to 1.2]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90: number analyzed (Participants) | 36 | 38
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90 | 1.0 [0.6 to 1.6] | 0.7 [0.5 to 1.2]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118: number analyzed (Participants) | 30 | 34
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118 | 0.9 [0.6 to 1.5] | 0.8 [0.5 to 1.2]
  B/Colorado/06/2017 (B Victoria lineage) - Day 8 | 1.5 [1.0 to 2.1] | 1.1 [0.8 to 1.5]
  B/Colorado/06/2017 (B Victoria lineage) - Day 57: number analyzed (Participants) | 37 | 38
  B/Colorado/06/2017 (B Victoria lineage) - Day 57 | 1.4 [1.0 to 2.0] | 1.0 [0.8 to 1.3]
  B/Colorado/06/2017 (B Victoria lineage) - Day 90: number analyzed (Participants) | 36 | 38
  B/Colorado/06/2017 (B Victoria lineage) - Day 90 | 1.4 [1.0 to 1.9] | 1.0 [0.8 to 1.4]
  B/Colorado/06/2017 (B Victoria lineage) - Day 118: number analyzed (Participants) | 30 | 34
  B/Colorado/06/2017 (B Victoria lineage) - Day 118 | 1.3 [0.9 to 1.8] | 1.1 [0.8 to 1.5]
  A/Michigan/45/2015 X-275 (H1N1) - Day 8 | 1.1 [0.7 to 1.5] | 0.9 [0.6 to 1.3]
  A/Michigan/45/2015 X-275 (H1N1) - Day 57: number analyzed (Participants) | 37 | 38
  A/Michigan/45/2015 X-275 (H1N1) - Day 57 | 1.0 [0.7 to 1.5] | 0.7 [0.5 to 1.1]
  A/Michigan/45/2015 X-275 (H1N1) - Day 90: number analyzed (Participants) | 36 | 38
  A/Michigan/45/2015 X-275 (H1N1) - Day 90 | 0.9 [0.6 to 1.4] | 0.7 [0.4 to 1.0]
  A/Michigan/45/2015 X-275 (H1N1) - Day 118: number analyzed (Participants) | 30 | 34
  A/Michigan/45/2015 X-275 (H1N1) - Day 118 | 0.8 [0.5 to 1.3] | 0.7 [0.4 to 1.1]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 8 | 1.5 [1.1 to 2.1] | 1.3 [1.0 to 1.7]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57: number analyzed (Participants) | 37 | 38
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57 | 1.5 [1.1 to 2.0] | 1.3 [1.0 to 1.8]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90: number analyzed (Participants) | 36 | 38
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90 | 1.5 [1.1 to 2.1] | 1.3 [1.0 to 1.7]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118: number analyzed (Participants) | 30 | 34
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118 | 1.4 [1.0 to 1.9] | 1.3 [1.0 to 1.7]

41. Secondary Outcome: Percentage of Participants Achieving Neuraminidase Inhibition (NAI) Titer Seroconversion Against 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains for the Fluzone Study Arms
Description: Blood was collected for NAI assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. NAI seroconversion was defined as >4 four-fold rise in post-vaccination antibody titer at Day 8, 57, 90, and 118.
Time Frame: Day 8, Day 57, Day 90, Day 118
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55
Number analyzed (Participants) | 41 | 37 | 40
percentage of participants
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 8 | 49 [33 to 65] | 62 [45 to 78] | 50 [34 to 66]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57: number analyzed (Participants) | 40 | 37 | 38
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57 | 20 [9 to 36] | 22 [10 to 38] | 24 [11 to 40]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90 | 12 [4 to 26] | 8 [2 to 22] | 13 [4 to 28]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118 | 28 [14 to 45] | 23 [10 to 42] | 32 [17 to 51]
  B/Colorado/06/2017 (B Victoria lineage) - Day 8 | 20 [9 to 35] | 30 [16 to 47] | 13 [4 to 27]
  B/Colorado/06/2017 (B Victoria lineage) - Day 57: number analyzed (Participants) | 40 | 37 | 38
  B/Colorado/06/2017 (B Victoria lineage) - Day 57 | 18 [7 to 33] | 16 [6 to 32] | 8 [2 to 21]
  B/Colorado/06/2017 (B Victoria lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38
  B/Colorado/06/2017 (B Victoria lineage) - Day 90 | 10 [3 to 23] | 8 [2 to 22] | 5 [NA to 18] — Value is NA because it's >0 but <1
  B/Colorado/06/2017 (B Victoria lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34
  B/Colorado/06/2017 (B Victoria lineage) - Day 118 | 19 [8 to 36] | 20 [8 to 39] | 9 [2 to 24]
  A/Michigan/45/2015 X-275 (H1N1) - Day 8 | 46 [31 to 63] | 57 [39 to 73] | 50 [34 to 66]
  A/Michigan/45/2015 X-275 (H1N1) - Day 57: number analyzed (Participants) | 40 | 37 | 38
  A/Michigan/45/2015 X-275 (H1N1) - Day 57 | 15 [6 to 30] | 22 [10 to 38] | 11 [3 to 25]
  A/Michigan/45/2015 X-275 (H1N1) - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Michigan/45/2015 X-275 (H1N1) - Day 90 | 10 [3 to 23] | 11 [3 to 26] | 3 [NA to 14] — Value is NA because it's >0 but <1
  A/Michigan/45/2015 X-275 (H1N1) - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Michigan/45/2015 X-275 (H1N1) - Day 118 | 25 [12 to 42] | 13 [4 to 31] | 24 [11 to 41]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 8 | 27 [14 to 43] | 30 [16 to 47] | 20 [9 to 36]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57: number analyzed (Participants) | 40 | 37 | 38
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57 | 18 [7 to 33] | 16 [6 to 32] | 8 [2 to 21]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90 | 12 [4 to 26] | 11 [3 to 26] | 5 [NA to 18] — Value is NA because it's >0 but <1
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118 | 17 [6 to 33] | 10 [2 to 27] | 6 [NA to 20] — Value is NA because it's >0 but <1

42. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in Neuraminidase Inhibition (NAI) Titers Against the 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains for the Fluzone Study Arms
Description: Blood was collected for NAI assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. Fold-rises from baseline were calculated as the Day 8 (or Day 57, Day 90, Day 118) titer divided by the baseline titers for each participant. The geometric mean of these fold rises was then calculated to obtain the GMFR.
Time Frame: Day 8, Day 57, Day 90, Day 118
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55
Number analyzed (Participants) | 41 | 37 | 40
fold rise
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 8 | 3.6 [2.6 to 4.9] | 4.3 [3.3 to 5.7] | 4.3 [3.2 to 5.8]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57: number analyzed (Participants) | 40 | 37 | 38
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57 | 2.0 [1.7 to 2.4] | 2.2 [1.8 to 2.8] | 2.4 [1.9 to 3.0]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90 | 1.6 [1.4 to 1.9] | 1.7 [1.4 to 2.1] | 1.8 [1.5 to 2.1]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118 | 2.2 [1.7 to 2.7] | 2.1 [1.6 to 2.8] | 2.7 [2.2 to 3.4]
  B/Colorado/06/2017 (B Victoria lineage) - Day 8 | 2.2 [1.7 to 2.8] | 2.7 [2.0 to 3.6] | 1.9 [1.5 to 2.5]
  B/Colorado/06/2017 (B Victoria lineage) - Day 57: number analyzed (Participants) | 40 | 37 | 38
  B/Colorado/06/2017 (B Victoria lineage) - Day 57 | 1.8 [1.5 to 2.1] | 2.0 [1.6 to 2.6] | 1.5 [1.3 to 1.8]
  B/Colorado/06/2017 (B Victoria lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38
  B/Colorado/06/2017 (B Victoria lineage) - Day 90 | 1.6 [1.3 to 1.9] | 1.9 [1.5 to 2.4] | 1.5 [1.2 to 1.8]
  B/Colorado/06/2017 (B Victoria lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34
  B/Colorado/06/2017 (B Victoria lineage) - Day 118 | 2.2 [1.8 to 2.7] | 2.5 [1.9 to 3.3] | 2.0 [1.6 to 2.3]
  A/Michigan/45/2015 X-275 (H1N1) - Day 8 | 3.4 [2.6 to 4.5] | 3.9 [2.8 to 5.3] | 3.6 [2.7 to 4.9]
  A/Michigan/45/2015 X-275 (H1N1) - Day 57: number analyzed (Participants) | 40 | 37 | 38
  A/Michigan/45/2015 X-275 (H1N1) - Day 57 | 1.8 [1.5 to 2.1] | 2.0 [1.6 to 2.6] | 1.8 [1.4 to 2.2]
  A/Michigan/45/2015 X-275 (H1N1) - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Michigan/45/2015 X-275 (H1N1) - Day 90 | 1.6 [1.4 to 1.9] | 1.6 [1.2 to 2.0] | 1.4 [1.2 to 1.7]
  A/Michigan/45/2015 X-275 (H1N1) - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Michigan/45/2015 X-275 (H1N1) - Day 118 | 2.4 [1.9 to 2.9] | 2.0 [1.5 to 2.6] | 2.2 [1.8 to 2.8]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 8 | 2.2 [1.6 to 3.0] | 2.3 [1.8 to 2.9] | 1.9 [1.5 to 2.4]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57: number analyzed (Participants) | 40 | 37 | 38
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57 | 1.8 [1.5 to 2.3] | 2.0 [1.6 to 2.5] | 1.7 [1.5 to 2.1]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90 | 1.6 [1.3 to 2.0] | 1.7 [1.4 to 2.2] | 1.5 [1.3 to 1.8]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118 | 1.9 [1.5 to 2.5] | 1.7 [1.3 to 2.2] | 1.7 [1.4 to 2.0]

43. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Neutralizing (Neut) Titers Against the 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains
Description: Blood was collected for Neut assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, but only one result which is a geometric mean titer of the replicates was reported by the lab. The geometric mean titer was calculated for each study arm from the available results at Day 8, Day 57, Day 90, and Day 118 Post first study vaccination.
Time Frame: Day 8, Day 57, Day 90, Day 118
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 41 | 38 | 42
titer
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 8 | 140.6 [106.7 to 185.4] | 271.9 [201.0 to 367.9] | 154.0 [113.7 to 208.6] | 168.8 [129.9 to 219.5] | 210.6 [149.7 to 296.3] | 148.5 [111.9 to 196.9]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57 | 150.2 [114.2 to 197.5] | 312.9 [243.1 to 402.6] | 195.6 [142.1 to 269.1] | 354.4 [264.8 to 474.5] | 309.0 [219.9 to 434.1] | 259.3 [189.4 to 355.0]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90 | 132.1 [102.0 to 171.1] | 244.2 [177.7 to 335.6] | 152.8 [107.1 to 217.9] | 273.4 [185.7 to 402.6] | 265.7 [184.9 to 381.8] | 202.7 [144.5 to 284.3]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118 | 161.8 [113.5 to 230.7] | 257.6 [188.3 to 352.4] | 224.1 [156.4 to 321.3] | 446.6 [300.1 to 664.6] | 409.5 [286.6 to 585.1] | 276.8 [178.2 to 430.0]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 8 | 309.6 [203.4 to 471.4] | 333.9 [223.3 to 499.3] | 261.6 [165.7 to 413.0] | 369.0 [227.9 to 597.7] | 243.2 [148.5 to 398.4] | 255.4 [169.9 to 383.8]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 57 | 365.7 [238.0 to 561.8] | 358.1 [231.2 to 554.8] | 232.1 [147.8 to 364.6] | 439.5 [255.9 to 755.0] | 300.2 [178.1 to 506.3] | 306.0 [198.5 to 471.7]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90 | 255.4 [173.2 to 376.7] | 235.4 [164.9 to 335.9] | 178.3 [110.1 to 288.7] | 362.6 [208.1 to 632.0] | 234.1 [140.7 to 389.6] | 232.4 [151.2 to 357.3]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118 | 202.2 [127.2 to 321.4] | 180.7 [113.0 to 288.9] | 151.5 [85.9 to 267.2] | 312.0 [160.1 to 607.8] | 212.1 [127.1 to 354.2] | 211.7 [136.9 to 327.2]
  A/Michigan/45/2015 X-275 (H1N1) - Day 8 | 6824.7 [5245.8 to 8878.7] | 7795.4 [5275.0 to 11520.0] | 5604.4 [3894.9 to 8064.2] | 6666.4 [4657.5 to 9541.7] | 8444.6 [5590.8 to 12755.0] | 5925.2 [4184.9 to 8389.3]
  A/Michigan/45/2015 X-275 (H1N1) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Michigan/45/2015 X-275 (H1N1) - Day 57 | 3437.4 [2218.8 to 5325.2] | 4437.2 [3179.4 to 6192.8] | 3335.0 [2194.5 to 5068.3] | 8293.9 [5358.8 to 12836.6] | 6502.7 [4251.4 to 9946.1] | 5791.6 [3915.1 to 8567.5]
  A/Michigan/45/2015 X-275 (H1N1) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Michigan/45/2015 X-275 (H1N1) - Day 90 | 4623.9 [3377.1 to 6331.0] | 4965.3 [3475.0 to 7094.9] | 3255.1 [2163.5 to 4897.5] | 6518.8 [4528.7 to 9383.4] | 6113.7 [4061.6 to 9202.6] | 4837.8 [3410.7 to 6862.1]
  A/Michigan/45/2015 X-275 (H1N1) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Michigan/45/2015 X-275 (H1N1) - Day 118 | 5094.4 [3714.6 to 6986.7] | 5393.5 [3578.0 to 8130.2] | 3153.9 [2145.3 to 4636.8] | 8037.0 [5516.3 to 11709.7] | 6631.4 [4338.9 to 10135.2] | 6168.6 [4323.8 to 8800.5]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 8 | 1126.1 [727.4 to 1743.5] | 1049.1 [645.4 to 1705.3] | 1095.1 [817.4 to 1467.1] | 1515.8 [1031.0 to 2228.7] | 1154.5 [747.1 to 1784.0] | 824.8 [495.5 to 1372.9]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57 | 859.6 [592.8 to 1246.6] | 1225.3 [851.4 to 1763.2] | 1037.6 [759.5 to 1417.5] | 1959.7 [1398.2 to 2746.6] | 1243.1 [834.1 to 1852.8] | 1173.0 [816.8 to 1684.5]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90 | 681.0 [490.3 to 945.9] | 909.3 [638.8 to 1294.5] | 766.9 [541.3 to 1086.4] | 1371.5 [981.9 to 1915.7] | 953.5 [638.6 to 1423.7] | 754.8 [533.9 to 1066.9]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118 | 1087.2 [762.1 to 1551.2] | 1031.7 [703.9 to 1512.2] | 1086.9 [798.5 to 1479.6] | 1920.9 [1351.2 to 2730.8] | 1234.9 [710.6 to 2146.0] | 1284.8 [914.5 to 1805.0]

44. Secondary Outcome: Ratio of Serum Neutralizing (Neut) Geometric Mean Titers (GMT) Against the 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains Between Adjuvanted and Unadjuvanted Study Arms
Description: Blood was collected for Neut assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, but only one result which is a geometric mean titer of the replicates was reported by the lab. The geometric mean titer was calculated for each study arm from the available results at Day 8, Day 57, Day 90, and Day 118 Post first study vaccination and the ratio of these GMTs between adjuvanted and unadjuvanted study arms were calculated.
  Unadjuvanted Fluzone and Flublok study arms are considered as reference groups for the analysis of ratio of GMTs.
  Ratio of GMTs is defined as the ratio of the GMT from the adjuvanted group divided by the GMT from the corresponding unadjuvanted group.
Time Frame: Day 8, Day 57, Day 90, Day 118
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: ratio of GMT
Arm/Group | Fluzone + AF03 | Fluzone + CpG55 | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 37 | 40 | 38 | 42
ratio of GMT
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 8 | 1.9 [1.3 to 2.9] | 1.1 [0.7 to 1.6] | 1.2 [0.8 to 1.9] | 0.9 [0.6 to 1.3]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57: number analyzed (Participants) | 37 | 38 | 37 | 41
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57 | 2.1 [1.4 to 3.0] | 1.3 [0.9 to 2.0] | 0.9 [0.6 to 1.4] | 0.7 [0.5 to 1.1]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90: number analyzed (Participants) | 36 | 38 | 37 | 40
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90 | 1.8 [1.2 to 2.8] | 1.2 [0.8 to 1.8] | 1.0 [0.6 to 1.6] | 0.7 [0.4 to 1.2]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118: number analyzed (Participants) | 30 | 34 | 32 | 34
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118 | 1.6 [1.0 to 2.5] | 1.4 [0.8 to 2.3] | 0.9 [0.5 to 1.5] | 0.6 [0.3 to 1.1]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 8 | 1.1 [0.6 to 1.9] | 0.8 [0.5 to 1.6] | 0.7 [0.3 to 1.3] | 0.7 [0.4 to 1.3]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 57: number analyzed (Participants) | 37 | 38 | 37 | 41
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 57 | 1.0 [0.5 to 1.8] | 0.6 [0.3 to 1.2] | 0.7 [0.3 to 1.4] | 0.7 [0.4 to 1.4]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90: number analyzed (Participants) | 36 | 38 | 37 | 40
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90 | 0.9 [0.5 to 1.5] | 0.7 [0.4 to 1.3] | 0.6 [0.3 to 1.4] | 0.6 [0.3 to 1.3]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118: number analyzed (Participants) | 30 | 34 | 32 | 34
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118 | 0.9 [0.5 to 1.7] | 0.7 [0.4 to 1.5] | 0.7 [0.3 to 1.6] | 0.7 [0.3 to 1.5]
  A/Michigan/45/2015 X-275 (H1N1) - Day 8 | 1.1 [0.7 to 1.8] | 0.8 [0.5 to 1.3] | 1.3 [0.7 to 2.2] | 0.9 [0.5 to 1.5]
  A/Michigan/45/2015 X-275 (H1N1) - Day 57: number analyzed (Participants) | 37 | 38 | 37 | 41
  A/Michigan/45/2015 X-275 (H1N1) - Day 57 | 1.3 [0.8 to 2.2] | 1.0 [0.5 to 1.8] | 0.8 [0.4 to 1.4] | 0.7 [0.4 to 1.2]
  A/Michigan/45/2015 X-275 (H1N1) - Day 90: number analyzed (Participants) | 36 | 38 | 37 | 40
  A/Michigan/45/2015 X-275 (H1N1) - Day 90 | 1.1 [0.7 to 1.7] | 0.7 [0.4 to 1.2] | 0.9 [0.5 to 1.6] | 0.7 [0.5 to 1.2]
  A/Michigan/45/2015 X-275 (H1N1) - Day 118: number analyzed (Participants) | 30 | 34 | 32 | 34
  A/Michigan/45/2015 X-275 (H1N1) - Day 118 | 1.1 [0.6 to 1.8] | 0.6 [0.4 to 1.0] | 0.8 [0.5 to 1.4] | 0.8 [0.5 to 1.3]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 8 | 0.9 [0.5 to 1.8] | 1.0 [0.6 to 1.6] | 0.8 [0.4 to 1.3] | 0.5 [0.3 to 1.0]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57: number analyzed (Participants) | 37 | 38 | 37 | 41
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57 | 1.4 [0.9 to 2.4] | 1.2 [0.7 to 1.9] | 0.6 [0.4 to 1.1] | 0.6 [0.4 to 1.0]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90: number analyzed (Participants) | 36 | 38 | 37 | 40
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90 | 1.3 [0.8 to 2.1] | 1.1 [0.7 to 1.8] | 0.7 [0.4 to 1.2] | 0.6 [0.3 to 0.9]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118: number analyzed (Participants) | 30 | 34 | 32 | 34
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118 | 0.9 [0.6 to 1.6] | 1.0 [0.6 to 1.6] | 0.6 [0.3 to 1.2] | 0.7 [0.4 to 1.1]

45. Secondary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Titer Seroconversion Against 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains
Description: Blood was collected for Neut assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, but only one result which is a geometric mean titer of the replicates was reported by the lab. Neut seroconversion was defined as either a pre-vaccination titer < 1:10 and a post-vaccination titer >= 1:40 or a pre-vaccination titer >= 1:10 and a minimum four-fold rise in post-vaccination antibody titer.
Time Frame: Day 8, Day 57, Day 90, Day 118
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 41 | 38 | 42
percentage of participants
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 8 | 10 [3 to 23] | 16 [6 to 32] | 20 [9 to 36] | 15 [6 to 29] | 11 [3 to 25] | 7 [1 to 19]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57 | 10 [3 to 24] | 22 [10 to 38] | 18 [8 to 34] | 38 [23 to 54] | 27 [14 to 44] | 24 [12 to 40]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90 | 12 [4 to 26] | 11 [3 to 26] | 13 [4 to 28] | 23 [11 to 39] | 22 [10 to 38] | 10 [3 to 24]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118 | 14 [5 to 29] | 10 [2 to 27] | 24 [11 to 41] | 32 [17 to 51] | 38 [21 to 56] | 24 [11 to 41]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 8 | 15 [6 to 29] | 24 [12 to 41] | 30 [17 to 47] | 15 [6 to 29] | 34 [20 to 51] | 31 [18 to 47]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 57 | 25 [13 to 41] | 27 [14 to 44] | 32 [18 to 49] | 25 [13 to 41] | 35 [20 to 53] | 34 [20 to 51]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90 | 17 [7 to 32] | 19 [8 to 36] | 18 [8 to 34] | 13 [4 to 27] | 30 [16 to 47] | 25 [13 to 41]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118 | 14 [5 to 29] | 17 [6 to 35] | 18 [7 to 35] | 9 [2 to 24] | 28 [14 to 47] | 26 [13 to 44]
  A/Michigan/45/2015 X-275 (H1N1) - Day 8 | 17 [7 to 32] | 24 [12 to 41] | 20 [9 to 36] | 20 [9 to 35] | 37 [22 to 54] | 24 [12 to 39]
  A/Michigan/45/2015 X-275 (H1N1) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Michigan/45/2015 X-275 (H1N1) - Day 57 | 13 [4 to 27] | 11 [3 to 25] | 8 [2 to 21] | 23 [11 to 38] | 27 [14 to 44] | 17 [7 to 32]
  A/Michigan/45/2015 X-275 (H1N1) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Michigan/45/2015 X-275 (H1N1) - Day 90 | 12 [4 to 26] | 11 [3 to 26] | 11 [3 to 25] | 8 [2 to 21] | 30 [16 to 47] | 13 [4 to 27]
  A/Michigan/45/2015 X-275 (H1N1) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Michigan/45/2015 X-275 (H1N1) - Day 118 | 11 [3 to 26] | 10 [2 to 27] | 18 [7 to 35] | 18 [7 to 35] | 31 [16 to 50] | 21 [9 to 38]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 8 | 32 [18 to 48] | 11 [3 to 25] | 23 [11 to 38] | 24 [12 to 40] | 24 [11 to 40] | 19 [9 to 34]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57 | 28 [15 to 44] | 16 [6 to 32] | 21 [10 to 37] | 18 [7 to 33] | 22 [10 to 38] | 27 [14 to 43]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90 | 15 [6 to 29] | 11 [3 to 26] | 8 [2 to 21] | 15 [6 to 31] | 22 [10 to 38] | 15 [6 to 30]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118 | 22 [10 to 39] | 13 [4 to 31] | 18 [7 to 35] | 18 [7 to 35] | 16 [5 to 33] | 21 [9 to 38]

46. Secondary Outcome: Percentage of Participants With Neutralizing (Neut) Titer of 1:40 or Greater Against the 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains
Description: Blood was collected for Neut assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, but only one result which is a geometric mean titer of the replicates was reported by the lab.
Time Frame: Day 8, Day 57, Day 90, Day 118
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 41 | 38 | 42
percentage of participants
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 8 | 95 [83 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 95 [83 to NA] — Value is NA because it's >99 but <100 | 95 [83 to NA] — Value is NA because it's >99 but <100 | 95 [82 to NA] — Value is NA because it's >99 but <100 | 93 [81 to 99]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57 | 98 [87 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 97 [86 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90 | 95 [83 to NA] — Value is NA because it's >99 but <100 | 100 [90 to 100] | 89 [75 to 97] | 97 [87 to NA] — Value is NA because it's >99 but <100 | 95 [82 to NA] — Value is NA because it's >99 but <100 | 93 [80 to 98]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118 | 94 [81 to NA] — Value is NA because it's >99 but <100 | 100 [88 to 100] | 97 [85 to NA] — Value is NA because it's >99 but <100 | 100 [90 to 100] | 97 [84 to NA] — Value is NA because it's >99 but <100 | 97 [85 to NA] — Value is NA because it's >99 but <100
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 8 | 93 [80 to 98] | 97 [86 to NA] — Value is NA because it's >99 but <100 | 90 [76 to 97] | 95 [83 to NA] — Value is NA because it's >99 but <100 | 87 [72 to 96] | 98 [87 to NA] — Value is NA because it's >99 but <100
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 57 | 95 [83 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 95 [82 to NA] — Value is NA because it's >99 but <100 | 90 [76 to 97] | 89 [75 to 97] | 98 [87 to NA] — Value is NA because it's >99 but <100
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90 | 95 [83 to NA] — Value is NA because it's >99 but <100 | 100 [90 to 100] | 82 [66 to 92] | 87 [73 to 96] | 89 [75 to 97] | 93 [80 to 98]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118 | 89 [74 to 97] | 90 [73 to 98] | 71 [53 to 85] | 85 [69 to 95] | 91 [75 to 98] | 94 [80 to NA] — Value is NA because it's >99 but <100
  A/Michigan/45/2015 X-275 (H1N1) - Day 8 | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [92 to 100]
  A/Michigan/45/2015 X-275 (H1N1) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Michigan/45/2015 X-275 (H1N1) - Day 57 | 98 [87 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100]
  A/Michigan/45/2015 X-275 (H1N1) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Michigan/45/2015 X-275 (H1N1) - Day 90 | 100 [91 to 100] | 100 [90 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100]
  A/Michigan/45/2015 X-275 (H1N1) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Michigan/45/2015 X-275 (H1N1) - Day 118 | 100 [90 to 100] | 100 [88 to 100] | 100 [90 to 100] | 100 [90 to 100] | 100 [89 to 100] | 100 [90 to 100]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 8 | 98 [87 to NA] — Value is NA because it's >99 but <100 | 97 [86 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 100 [91 to 100] | 97 [86 to NA] — Value is NA because it's >99 but <100 | 95 [84 to NA] — Value is NA because it's >99 but <100
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57 | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90 | 100 [91 to 100] | 100 [90 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118 | 100 [90 to 100] | 100 [88 to 100] | 100 [90 to 100] | 100 [90 to 100] | 97 [84 to NA] — Value is NA because it's >99 but <100 | 100 [90 to 100]

47. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in Neutralizing (Neut) Titers Against the 2018/2019 Quadrivalent Influenza Vaccine (QIV) Strains
Description: Blood was collected for Neut assay which was conducted with the 2018/2019 QIV viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, but only one result which a geometric mean titer of the replicates was reported by the lab. Fold-rises from baseline were calculated as the Day 8 (or Day 57, Day 90, Day 118) titer divided by the baseline titers for each participant. The geometric mean of these fold rises was then calculated to obtain the GMFR.
Time Frame: Day 8, Day 57, Day 90, Day 118
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 41 | 38 | 42
fold rise
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 8 | 1.3 [1.0 to 1.8] | 1.8 [1.3 to 2.6] | 1.5 [1.1 to 2.1] | 1.1 [0.8 to 1.5] | 1.7 [1.3 to 2.3] | 1.3 [0.9 to 1.7]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 57 | 1.4 [1.1 to 1.8] | 2.1 [1.5 to 2.9] | 2.0 [1.4 to 2.9] | 2.3 [1.7 to 3.1] | 2.5 [1.9 to 3.3] | 2.1 [1.5 to 2.9]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 90 | 1.2 [0.9 to 1.6] | 1.6 [1.1 to 2.2] | 1.6 [1.2 to 2.2] | 1.8 [1.3 to 2.5] | 2.1 [1.5 to 3.0] | 1.7 [1.2 to 2.2]
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Singapore/INFIMH-16-0019/2016 IVR-186 (H3N2) - Day 118 | 1.7 [1.3 to 2.2] | 1.7 [1.3 to 2.3] | 2.4 [1.7 to 3.5] | 3.0 [2.3 to 4.1] | 3.5 [2.5 to 4.9] | 2.4 [1.8 to 3.3]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 8 | 2.8 [1.6 to 5.0] | 2.9 [1.8 to 4.9] | 2.8 [1.6 to 4.9] | 1.9 [1.3 to 2.6] | 3.0 [1.9 to 4.5] | 2.5 [1.8 to 3.6]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 57 | 3.2 [1.9 to 5.3] | 3.2 [1.7 to 5.8] | 2.5 [1.6 to 4.0] | 2.2 [1.5 to 3.2] | 3.6 [2.2 to 5.7] | 2.9 [2.0 to 4.4]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 90 | 2.3 [1.6 to 3.5] | 2.1 [1.3 to 3.6] | 2.0 [1.3 to 2.9] | 1.8 [1.3 to 2.5] | 2.8 [1.9 to 4.0] | 2.3 [1.6 to 3.2]
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  B/Maryland/15/2016 BX-69A (B Victoria lineage) - Day 118 | 1.8 [1.2 to 2.9] | 1.7 [0.9 to 3.2] | 1.7 [1.1 to 2.8] | 1.5 [1.1 to 2.1] | 2.5 [1.6 to 3.8] | 2.2 [1.4 to 3.4]
  A/Michigan/45/2015 X-275 (H1N1) - Day 8 | 2.2 [1.4 to 3.4] | 2.9 [1.7 to 4.8] | 2.6 [1.6 to 4.4] | 1.8 [1.3 to 2.4] | 3.8 [2.3 to 6.2] | 2.1 [1.5 to 3.1]
  A/Michigan/45/2015 X-275 (H1N1) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Michigan/45/2015 X-275 (H1N1) - Day 57 | 1.0 [0.6 to 1.6] | 1.6 [1.0 to 2.8] | 1.7 [1.0 to 2.7] | 2.1 [1.5 to 2.9] | 3.0 [1.9 to 4.8] | 2.0 [1.4 to 3.1]
  A/Michigan/45/2015 X-275 (H1N1) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Michigan/45/2015 X-275 (H1N1) - Day 90 | 1.5 [1.0 to 2.2] | 1.7 [1.1 to 2.9] | 1.6 [1.0 to 2.6] | 1.6 [1.3 to 2.1] | 2.9 [1.8 to 4.4] | 1.7 [1.2 to 2.5]
  A/Michigan/45/2015 X-275 (H1N1) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Michigan/45/2015 X-275 (H1N1) - Day 118 | 1.5 [1.0 to 2.2] | 1.7 [0.9 to 3.2] | 1.8 [1.1 to 2.9] | 2.0 [1.5 to 2.6] | 3.0 [1.8 to 4.9] | 2.3 [1.6 to 3.5]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 8 | 2.3 [1.4 to 4.0] | 1.8 [1.2 to 2.9] | 1.7 [1.2 to 2.4] | 1.8 [1.2 to 2.6] | 2.6 [1.6 to 4.3] | 1.5 [0.9 to 2.5]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 57 | 1.8 [1.2 to 2.6] | 2.1 [1.3 to 3.4] | 1.6 [1.1 to 2.4] | 2.2 [1.6 to 3.1] | 2.7 [1.7 to 4.3] | 2.1 [1.4 to 3.1]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 90 | 1.4 [1.0 to 1.9] | 1.5 [1.0 to 2.3] | 1.2 [0.9 to 1.7] | 1.6 [1.1 to 2.3] | 2.1 [1.3 to 3.4] | 1.4 [1.0 to 2.0]
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  B/Phuket/3073/2013 (B Yamagata lineage) - Day 118 | 2.2 [1.5 to 3.3] | 1.7 [1.0 to 2.8] | 1.9 [1.3 to 2.6] | 2.3 [1.6 to 3.3] | 2.4 [1.5 to 4.1] | 2.6 [1.9 to 3.5]

48. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Hemagglutination Inhibition (HAI) Against Heterologous H1 and H3 Influenza Strains
Description: Blood was collected for HAI assay which was conducted with the heterologous H1 and H3 influenza viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at Day 1, Day 8, Day 29, Day 57, Day 90, and Day 118 post first study vaccination.
Time Frame: Day 1, Day 8, Day 29, Day 57, Day 90, Day 118
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 41 | 38 | 42
titer
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 1 | 59.5 [39.7 to 89.3] | 113.1 [71.1 to 180.0] | 70.3 [44.2 to 111.6] | 87.8 [53.7 to 143.5] | 78.6 [49.2 to 125.4] | 63.5 [41.2 to 97.8]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 8 | 189.5 [138.6 to 259.0] | 440.0 [307.1 to 630.5] | 296.0 [210.3 to 416.6] | 261.2 [176.8 to 386.1] | 357.0 [223.6 to 570.0] | 299.6 [209.6 to 428.2]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 29 | 184.7 [126.9 to 269.0] | 415.0 [299.9 to 574.3] | 282.6 [195.5 to 408.5] | 400.9 [272.9 to 588.8] | 440.0 [279.1 to 693.7] | 366.3 [249.2 to 538.4]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 57 | 116.1 [78.6 to 171.5] | 272.9 [193.9 to 384.1] | 167.5 [113.0 to 248.1] | 314.5 [212.0 to 466.6] | 317.0 [204.6 to 491.2] | 281.9 [194.6 to 408.4]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 90 | 112.2 [75.4 to 167.0] | 264.0 [182.7 to 381.4] | 155.7 [102.6 to 236.3] | 272.7 [179.6 to 414.1] | 288.7 [182.3 to 457.1] | 244.6 [163.5 to 365.9]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 118 | 215.6 [137.9 to 337.1] | 351.0 [232.5 to 529.9] | 291.9 [197.3 to 432.0] | 583.9 [360.2 to 946.5] | 580.6 [362.1 to 930.8] | 388.4 [246.3 to 612.5]
  A/Aksaray/4048/2016 [H3N2] - Day 1 | 72.9 [48.1 to 110.6] | 141.7 [87.1 to 230.3] | 76.6 [48.8 to 120.4] | 112.2 [72.3 to 174.1] | 80.0 [50.7 to 126.2] | 87.6 [60.5 to 126.8]
  A/Aksaray/4048/2016 [H3N2] - Day 8 | 178.6 [133.9 to 238.1] | 452.5 [337.9 to 606.1] | 259.9 [188.5 to 358.4] | 314.6 [230.5 to 429.5] | 394.7 [264.7 to 588.5] | 339.0 [251.7 to 456.7]
  A/Aksaray/4048/2016 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Aksaray/4048/2016 [H3N2] - Day 29 | 174.1 [124.2 to 244.1] | 415.0 [298.8 to 576.4] | 222.3 [157.8 to 313.2] | 433.4 [326.5 to 575.2] | 456.8 [322.1 to 647.8] | 402.0 [295.2 to 547.6]
  A/Aksaray/4048/2016 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Aksaray/4048/2016 [H3N2] - Day 57 | 146.7 [102.2 to 210.7] | 338.5 [250.4 to 457.6] | 188.5 [131.5 to 270.2] | 407.9 [303.0 to 549.0] | 423.8 [299.4 to 600.0] | 366.3 [269.9 to 497.2]
  A/Aksaray/4048/2016 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Aksaray/4048/2016 [H3N2] - Day 90 | 140.9 [95.5 to 207.9] | 299.1 [212.8 to 420.6] | 157.1 [104.7 to 235.8] | 331.6 [241.6 to 455.0] | 323.0 [222.9 to 468.1] | 293.4 [214.1 to 402.2]
  A/Aksaray/4048/2016 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Aksaray/4048/2016 [H3N2] - Day 118 | 320.0 [226.8 to 451.6] | 496.4 [336.9 to 731.2] | 438.9 [300.0 to 642.1] | 877.8 [610.8 to 1261.5] | 812.2 [548.2 to 1203.4] | 578.0 [394.5 to 846.7]
  A/Kenya/105/2017 [H3N2] - Day 1 | 63.7 [44.3 to 91.6] | 123.1 [79.5 to 190.5] | 67.3 [42.7 to 106.1] | 105.7 [71.6 to 156.1] | 69.8 [44.7 to 108.9] | 78.0 [56.6 to 107.6]
  A/Kenya/105/2017 [H3N2] - Day 8 | 184.7 [140.7 to 242.6] | 483.2 [349.8 to 667.6] | 251.1 [184.4 to 341.8] | 312.0 [233.7 to 416.4] | 405.6 [273.8 to 600.9] | 374.3 [281.9 to 497.0]
  A/Kenya/105/2017 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Kenya/105/2017 [H3N2] - Day 29 | 265.7 [186.9 to 377.8] | 646.2 [472.1 to 884.6] | 311.6 [225.0 to 431.4] | 656.9 [480.9 to 897.3] | 709.5 [494.9 to 1017.1] | 650.9 [494.7 to 856.5]
  A/Kenya/105/2017 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Kenya/105/2017 [H3N2] - Day 57 | 182.2 [132.9 to 249.7] | 435.9 [311.3 to 610.4] | 216.2 [153.0 to 305.4] | 452.5 [339.2 to 603.8] | 416.0 [302.6 to 571.7] | 405.5 [309.0 to 532.1]
  A/Kenya/105/2017 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Kenya/105/2017 [H3N2] - Day 90 | 202.7 [141.1 to 291.3] | 508.0 [357.5 to 721.7] | 226.3 [156.5 to 327.2] | 545.4 [404.8 to 734.9] | 516.0 [365.8 to 727.7] | 460.5 [335.9 to 631.2]
  A/Kenya/105/2017 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Kenya/105/2017 [H3N2] - Day 118 | 269.1 [191.2 to 378.7] | 417.4 [275.4 to 632.6] | 301.0 [204.3 to 443.5] | 784.7 [546.9 to 1126.0] | 661.1 [445.1 to 982.0] | 543.7 [372.1 to 794.4]
  A/Louisiana/13/2017 [H3N2] - Day 1 | 29.8 [20.7 to 42.8] | 61.5 [38.4 to 98.6] | 29.8 [19.6 to 45.4] | 43.5 [28.8 to 65.8] | 33.0 [23.0 to 47.4] | 34.8 [25.0 to 48.4]
  A/Louisiana/13/2017 [H3N2] - Day 8 | 103.1 [74.2 to 143.1] | 248.5 [168.5 to 366.5] | 121.3 [85.8 to 171.4] | 130.6 [94.3 to 181.0] | 148.7 [100.1 to 220.9] | 117.9 [83.2 to 167.0]
  A/Louisiana/13/2017 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Louisiana/13/2017 [H3N2] - Day 29 | 113.1 [80.3 to 159.5] | 271.7 [188.0 to 392.6] | 129.3 [90.5 to 184.7] | 226.3 [160.7 to 318.6] | 196.6 [133.3 to 290.0] | 180.1 [125.1 to 259.2]
  A/Louisiana/13/2017 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Louisiana/13/2017 [H3N2] - Day 57 | 74.6 [53.1 to 104.8] | 169.2 [115.9 to 247.2] | 86.8 [58.7 to 128.6] | 177.5 [128.0 to 246.3] | 132.7 [89.1 to 197.5] | 127.4 [89.8 to 180.5]
  A/Louisiana/13/2017 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Louisiana/13/2017 [H3N2] - Day 90 | 72.3 [50.9 to 102.7] | 163.1 [107.8 to 246.7] | 77.1 [51.5 to 115.4] | 176.4 [124.7 to 249.5] | 129.0 [84.6 to 196.6] | 124.5 [86.1 to 180.0]
  A/Louisiana/13/2017 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Louisiana/13/2017 [H3N2] - Day 118 | 256.4 [174.2 to 377.5] | 278.6 [178.3 to 435.4] | 253.1 [168.2 to 381.0] | 673.5 [445.3 to 1018.6] | 521.0 [334.9 to 810.5] | 365.3 [239.0 to 558.4]
  A/Michigan/84/2016 [H3N2] - Day 1 | 82.1 [59.7 to 112.7] | 98.3 [67.6 to 143.0] | 62.8 [44.4 to 88.8] | 98.0 [69.8 to 137.5] | 58.1 [41.0 to 82.4] | 74.9 [54.8 to 102.3]
  A/Michigan/84/2016 [H3N2] - Day 8 | 115.1 [89.1 to 148.5] | 169.2 [120.6 to 237.4] | 96.8 [72.2 to 129.8] | 129.5 [91.8 to 182.7] | 100.5 [68.7 to 147.0] | 106.8 [76.0 to 150.0]
  A/Michigan/84/2016 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Michigan/84/2016 [H3N2] - Day 29 | 124.2 [94.8 to 162.7] | 152.5 [105.7 to 220.0] | 94.7 [68.5 to 130.9] | 168.5 [119.0 to 238.8] | 108.0 [71.8 to 162.3] | 121.1 [85.0 to 172.4]
  A/Michigan/84/2016 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Michigan/84/2016 [H3N2] - Day 57 | 95.1 [70.5 to 128.4] | 131.4 [92.0 to 187.8] | 75.7 [54.4 to 105.4] | 154.5 [108.1 to 221.0] | 81.5 [53.3 to 124.6] | 106.6 [74.1 to 153.4]
  A/Michigan/84/2016 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Michigan/84/2016 [H3N2] - Day 90 | 99.7 [73.2 to 135.8] | 137.2 [95.0 to 198.0] | 79.3 [56.0 to 112.3] | 162.9 [113.8 to 233.2] | 78.5 [51.8 to 119.1] | 111.2 [74.2 to 166.5]
  A/Michigan/84/2016 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Michigan/84/2016 [H3N2] - Day 118 | 129.5 [93.9 to 178.5] | 183.8 [122.3 to 276.2] | 121.5 [83.7 to 176.4] | 323.3 [231.3 to 451.8] | 153.2 [97.5 to 240.8] | 180.8 [118.8 to 275.2]

49. Secondary Outcome: Ratio of Geometric Mean Titers (GMTs) of Serum Hemagglutination Inhibition (HAI) Against Heterologous H1 and H3 Influenza Strains Between Adjuvanted and Unadjuvanted Study Arms
Description: Blood was collected for HAI assay which was conducted with the heterologous H1 and H3 influenza viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at Day 1, Day 8, Day 29, Day 57, Day 90, and Day 118 post first study vaccination and the ratio of these GMTs between adjuvanted and unadjuvanted study arms was calculated.
  Unadjuvanted Fluzone and Flublok study arms are considered as reference groups for the analysis of ratio of GMTs.
  Ratio of GMTs is defined as the ratio of the GMT from the adjuvanted group divided by the GMT from the corresponding unadjuvanted group.
Time Frame: Day 1, Day 8, Day 29, Day 57, Day 90, Day 118
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: ratio of GMT
Arm/Group | Fluzone + AF03 | Fluzone + CpG55 | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 37 | 40 | 38 | 42
ratio of GMT
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 1 | 1.9 [1.0 to 3.5] | 1.2 [0.6 to 2.2] | 0.9 [0.5 to 1.7] | 0.7 [0.4 to 1.4]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 8 | 2.3 [1.5 to 3.7] | 1.6 [1.0 to 2.5] | 1.4 [0.7 to 2.5] | 1.1 [0.7 to 1.9]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 29: number analyzed (Participants) | 36 | 39 | 37 | 41
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 29 | 2.2 [1.4 to 3.7] | 1.5 [0.9 to 2.6] | 1.1 [0.6 to 2.0] | 0.9 [0.5 to 1.6]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 57: number analyzed (Participants) | 37 | 38 | 37 | 41
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 57 | 2.4 [1.4 to 3.9] | 1.4 [0.8 to 2.5] | 1.0 [0.6 to 1.8] | 0.9 [0.5 to 1.5]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 90: number analyzed (Participants) | 36 | 38 | 37 | 40
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 90 | 2.4 [1.4 to 4.0] | 1.4 [0.8 to 2.4] | 1.1 [0.6 to 2.0] | 0.9 [0.5 to 1.6]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 118: number analyzed (Participants) | 30 | 34 | 32 | 34
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 118 | 1.6 [0.9 to 3.0] | 1.4 [0.8 to 2.4] | 1.0 [0.5 to 1.9] | 0.7 [0.3 to 1.3]
  A/Aksaray/4048/2016 [H3N2] - Day 1 | 1.9 [1.0 to 3.6] | 1.1 [0.6 to 1.9] | 0.7 [0.4 to 1.3] | 0.8 [0.4 to 1.4]
  A/Aksaray/4048/2016 [H3N2] - Day 8 | 2.5 [1.7 to 3.8] | 1.5 [1.0 to 2.2] | 1.3 [0.8 to 2.1] | 1.1 [0.7 to 1.6]
  A/Aksaray/4048/2016 [H3N2] - Day 29: number analyzed (Participants) | 36 | 39 | 37 | 41
  A/Aksaray/4048/2016 [H3N2] - Day 29 | 2.4 [1.5 to 3.8] | 1.3 [0.8 to 2.1] | 1.1 [0.7 to 1.6] | 0.9 [0.6 to 1.4]
  A/Aksaray/4048/2016 [H3N2] - Day 57: number analyzed (Participants) | 37 | 38 | 37 | 41
  A/Aksaray/4048/2016 [H3N2] - Day 57 | 2.3 [1.5 to 3.7] | 1.3 [0.8 to 2.1] | 1.0 [0.7 to 1.6] | 0.9 [0.6 to 1.4]
  A/Aksaray/4048/2016 [H3N2] - Day 90: number analyzed (Participants) | 36 | 38 | 37 | 40
  A/Aksaray/4048/2016 [H3N2] - Day 90 | 2.1 [1.3 to 3.5] | 1.1 [0.6 to 1.9] | 1.0 [0.6 to 1.6] | 0.9 [0.6 to 1.4]
  A/Aksaray/4048/2016 [H3N2] - Day 118: number analyzed (Participants) | 30 | 34 | 32 | 34
  A/Aksaray/4048/2016 [H3N2] - Day 118 | 1.6 [0.9 to 2.6] | 1.4 [0.8 to 2.3] | 0.9 [0.5 to 1.6] | 0.7 [0.4 to 1.1]
  A/Kenya/105/2017 [H3N2] - Day 1 | 1.9 [1.1 to 3.4] | 1.1 [0.6 to 1.9] | 0.7 [0.4 to 1.2] | 0.7 [0.4 to 1.2]
  A/Kenya/105/2017 [H3N2] - Day 8 | 2.6 [1.7 to 4.0] | 1.4 [0.9 to 2.0] | 1.3 [0.8 to 2.1] | 1.2 [0.8 to 1.8]
  A/Kenya/105/2017 [H3N2] - Day 29: number analyzed (Participants) | 36 | 39 | 37 | 41
  A/Kenya/105/2017 [H3N2] - Day 29 | 2.4 [1.5 to 3.9] | 1.2 [0.7 to 1.9] | 1.1 [0.7 to 1.7] | 1.0 [0.7 to 1.5]
  A/Kenya/105/2017 [H3N2] - Day 57: number analyzed (Participants) | 37 | 38 | 37 | 41
  A/Kenya/105/2017 [H3N2] - Day 57 | 2.4 [1.5 to 3.8] | 1.2 [0.7 to 1.9] | 0.9 [0.6 to 1.4] | 0.9 [0.6 to 1.3]
  A/Kenya/105/2017 [H3N2] - Day 90: number analyzed (Participants) | 36 | 38 | 37 | 40
  A/Kenya/105/2017 [H3N2] - Day 90 | 2.5 [1.5 to 4.1] | 1.1 [0.7 to 1.9] | 0.9 [0.6 to 1.5] | 0.8 [0.6 to 1.3]
  A/Kenya/105/2017 [H3N2] - Day 118: number analyzed (Participants) | 30 | 34 | 32 | 34
  A/Kenya/105/2017 [H3N2] - Day 118 | 1.6 [0.9 to 2.6] | 1.1 [0.7 to 1.9] | 0.8 [0.5 to 1.4] | 0.7 [0.4 to 1.2]
  A/Louisiana/13/2017 [H3N2] - Day 1 | 2.1 [1.2 to 3.7] | 1.0 [0.6 to 1.7] | 0.8 [0.4 to 1.3] | 0.8 [0.5 to 1.3]
  A/Louisiana/13/2017 [H3N2] - Day 8 | 2.4 [1.5 to 4.0] | 1.2 [0.7 to 1.9] | 1.1 [0.7 to 1.9] | 0.9 [0.6 to 1.4]
  A/Louisiana/13/2017 [H3N2] - Day 29: number analyzed (Participants) | 36 | 39 | 37 | 41
  A/Louisiana/13/2017 [H3N2] - Day 29 | 2.4 [1.5 to 3.9] | 1.1 [0.7 to 1.9] | 0.9 [0.5 to 1.4] | 0.8 [0.5 to 1.3]
  A/Louisiana/13/2017 [H3N2] - Day 57: number analyzed (Participants) | 37 | 38 | 37 | 41
  A/Louisiana/13/2017 [H3N2] - Day 57 | 2.3 [1.4 to 3.7] | 1.2 [0.7 to 1.9] | 0.7 [0.4 to 1.2] | 0.7 [0.4 to 1.1]
  A/Louisiana/13/2017 [H3N2] - Day 90: number analyzed (Participants) | 36 | 38 | 37 | 40
  A/Louisiana/13/2017 [H3N2] - Day 90 | 2.3 [1.3 to 3.8] | 1.1 [0.6 to 1.8] | 0.7 [0.4 to 1.3] | 0.7 [0.4 to 1.2]
  A/Louisiana/13/2017 [H3N2] - Day 118: number analyzed (Participants) | 30 | 34 | 32 | 34
  A/Louisiana/13/2017 [H3N2] - Day 118 | 1.1 [0.6 to 1.9] | 1.0 [0.6 to 1.7] | 0.8 [0.4 to 1.4] | 0.5 [0.3 to 1.0]
  A/Michigan/84/2016 [H3N2] - Day 1 | 1.2 [0.7 to 1.9] | 0.8 [0.5 to 1.2] | 0.6 [0.4 to 1.0] | 0.8 [0.5 to 1.2]
  A/Michigan/84/2016 [H3N2] - Day 8 | 1.5 [1.0 to 2.2] | 0.8 [0.6 to 1.2] | 0.8 [0.5 to 1.3] | 0.8 [0.5 to 1.3]
  A/Michigan/84/2016 [H3N2] - Day 29: number analyzed (Participants) | 36 | 39 | 37 | 41
  A/Michigan/84/2016 [H3N2] - Day 29 | 1.2 [0.8 to 1.9] | 0.8 [0.5 to 1.2] | 0.6 [0.4 to 1.1] | 0.7 [0.4 to 1.2]
  A/Michigan/84/2016 [H3N2] - Day 57: number analyzed (Participants) | 37 | 38 | 37 | 41
  A/Michigan/84/2016 [H3N2] - Day 57 | 1.4 [0.9 to 2.2] | 0.8 [0.5 to 1.2] | 0.5 [0.3 to 0.9] | 0.7 [0.4 to 1.1]
  A/Michigan/84/2016 [H3N2] - Day 90: number analyzed (Participants) | 36 | 38 | 37 | 40
  A/Michigan/84/2016 [H3N2] - Day 90 | 1.4 [0.9 to 2.2] | 0.8 [0.5 to 1.3] | 0.5 [0.3 to 0.8] | 0.7 [0.4 to 1.2]
  A/Michigan/84/2016 [H3N2] - Day 118: number analyzed (Participants) | 30 | 34 | 32 | 34
  A/Michigan/84/2016 [H3N2] - Day 118 | 1.4 [0.9 to 2.4] | 0.9 [0.6 to 1.5] | 0.5 [0.3 to 0.8] | 0.6 [0.3 to 0.9]

50. Secondary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Titer Seroconversion Against Heterologous H1 and H3 Influenza Strains
Description: Blood was collected for HAI assay which was conducted with the heterologous H1 and H3 influenza viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. HAI seroconversion was defined as either a pre-vaccination titer < 1:10 and a post-vaccination titer >= 1:40 or a pre-vaccination titer >= 1:10 and a minimum four-fold rise in post-vaccination antibody titer.
Time Frame: Day 8, Day 29, Day 57, Day 90, Day 118
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 41 | 38 | 42
percentage of participants
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 8 | 44 [28 to 60] | 38 [22 to 55] | 33 [19 to 49] | 27 [14 to 43] | 50 [33 to 67] | 48 [32 to 64]
  A/Aksaray/4048/2016 [H3N2] - Day 8 | 27 [14 to 43] | 30 [16 to 47] | 30 [17 to 47] | 29 [16 to 46] | 47 [31 to 64] | 40 [26 to 57]
  A/Kenya/105/2017 [H3N2] - Day 8 | 32 [18 to 48] | 38 [22 to 55] | 35 [21 to 52] | 32 [18 to 48] | 58 [41 to 74] | 57 [41 to 72]
  A/Louisiana/13/2017 [H3N2] - Day 8 | 39 [24 to 55] | 41 [25 to 58] | 45 [29 to 62] | 29 [16 to 46] | 47 [31 to 64] | 40 [26 to 57]
  A/Michigan/84/2016 [H3N2] - Day 8 | 10 [3 to 23] | 11 [3 to 25] | 10 [3 to 24] | 5 [NA to 17] — Value is NA because it's >0 but <1 | 11 [3 to 25] | 7 [1 to 19]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 29 | 37 [22 to 53] | 31 [16 to 48] | 36 [21 to 53] | 55 [38 to 71] | 57 [39 to 73] | 63 [47 to 78]
  A/Aksaray/4048/2016 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Aksaray/4048/2016 [H3N2] - Day 29 | 27 [14 to 43] | 31 [16 to 48] | 31 [17 to 48] | 48 [32 to 64] | 57 [39 to 73] | 59 [42 to 74]
  A/Kenya/105/2017 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Kenya/105/2017 [H3N2] - Day 29 | 51 [35 to 67] | 56 [38 to 72] | 51 [35 to 68] | 65 [48 to 79] | 78 [62 to 90] | 78 [62 to 89]
  A/Louisiana/13/2017 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Louisiana/13/2017 [H3N2] - Day 29 | 41 [26 to 58] | 53 [35 to 70] | 56 [40 to 72] | 53 [36 to 68] | 73 [56 to 86] | 59 [42 to 74]
  A/Michigan/84/2016 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Michigan/84/2016 [H3N2] - Day 29 | 5 [NA to 17] — Value is NA because it's >0 but <1 | 8 [2 to 22] | 8 [2 to 21] | 10 [3 to 24] | 16 [6 to 32] | 12 [4 to 26]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 57 | 18 [7 to 33] | 24 [12 to 41] | 26 [13 to 43] | 40 [25 to 57] | 49 [32 to 66] | 46 [31 to 63]
  A/Aksaray/4048/2016 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Aksaray/4048/2016 [H3N2] - Day 57 | 23 [11 to 38] | 27 [14 to 44] | 29 [15 to 46] | 40 [25 to 57] | 57 [39 to 73] | 51 [35 to 67]
  A/Kenya/105/2017 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Kenya/105/2017 [H3N2] - Day 57 | 23 [11 to 38] | 35 [20 to 53] | 39 [24 to 57] | 50 [34 to 66] | 62 [45 to 78] | 66 [49 to 80]
  A/Louisiana/13/2017 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Louisiana/13/2017 [H3N2] - Day 57 | 25 [13 to 41] | 30 [16 to 47] | 32 [18 to 49] | 45 [29 to 62] | 46 [29 to 63] | 44 [28 to 60]
  A/Michigan/84/2016 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Michigan/84/2016 [H3N2] - Day 57 | 3 [NA to 13] — Value is NA because it's >0 but <1 | 8 [2 to 22] | 5 [NA to 18] — Value is NA because it's >0 but <1 | 8 [2 to 20] | 11 [3 to 25] | 10 [3 to 23]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 90 | 20 [9 to 35] | 19 [8 to 36] | 24 [11 to 40] | 38 [23 to 55] | 38 [22 to 55] | 45 [29 to 62]
  A/Aksaray/4048/2016 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Aksaray/4048/2016 [H3N2] - Day 90 | 20 [9 to 35] | 19 [8 to 36] | 24 [11 to 40] | 38 [23 to 55] | 41 [25 to 58] | 45 [29 to 62]
  A/Kenya/105/2017 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Kenya/105/2017 [H3N2] - Day 90 | 34 [20 to 51] | 36 [21 to 54] | 39 [24 to 57] | 59 [42 to 74] | 62 [45 to 78] | 65 [48 to 79]
  A/Louisiana/13/2017 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Louisiana/13/2017 [H3N2] - Day 90 | 27 [14 to 43] | 22 [10 to 39] | 24 [11 to 40] | 46 [30 to 63] | 43 [27 to 61] | 48 [32 to 64]
  A/Michigan/84/2016 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Michigan/84/2016 [H3N2] - Day 90 | 2 [NA to 13] — Value is NA because it's >0 but <1 | 6 [NA to 19] — Value is NA because it's >0 but <1 | 5 [NA to 18] — Value is NA because it's >0 but <1 | 8 [2 to 21] | 14 [5 to 29] | 13 [4 to 27]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 118 | 53 [35 to 70] | 33 [17 to 53] | 47 [30 to 65] | 71 [53 to 85] | 69 [50 to 84] | 79 [62 to 91]
  A/Aksaray/4048/2016 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Aksaray/4048/2016 [H3N2] - Day 118 | 58 [41 to 74] | 37 [20 to 56] | 62 [44 to 78] | 79 [62 to 91] | 75 [57 to 89] | 76 [59 to 89]
  A/Kenya/105/2017 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Kenya/105/2017 [H3N2] - Day 118 | 56 [38 to 72] | 30 [15 to 49] | 62 [44 to 78] | 74 [56 to 87] | 88 [71 to 96] | 82 [65 to 93]
  A/Louisiana/13/2017 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Louisiana/13/2017 [H3N2] - Day 118 | 78 [61 to 90] | 47 [28 to 66] | 82 [65 to 93] | 85 [69 to 95] | 91 [75 to 98] | 91 [76 to 98]
  A/Michigan/84/2016 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Michigan/84/2016 [H3N2] - Day 118 | 11 [3 to 26] | 13 [4 to 31] | 15 [5 to 31] | 38 [22 to 56] | 38 [21 to 56] | 26 [13 to 44]

51. Secondary Outcome: Percentage of Participants With Hemagglutination Inhibition (HAI) Titer of 1:40 or Greater Against Heterologous H1 and H3 Influenza Strains
Description: Blood was collected for HAI assay which was conducted with the heterologous H1 and H3 influenza viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result.
Time Frame: Day 1, Day 8, Day 29, Day 57, Day 90, Day 118
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 41 | 38 | 42
percentage of participants
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 1 | 78 [62 to 89] | 78 [62 to 90] | 73 [56 to 85] | 71 [54 to 84] | 71 [54 to 85] | 69 [53 to 82]
  A/Aksaray/4048/2016 [H3N2] - Day 1 | 78 [62 to 89] | 81 [65 to 92] | 70 [53 to 83] | 80 [65 to 91] | 71 [54 to 85] | 81 [66 to 91]
  A/Kenya/105/2017 [H3N2] - Day 1 | 78 [62 to 89] | 86 [71 to 95] | 70 [53 to 83] | 90 [77 to 97] | 74 [57 to 87] | 86 [71 to 95]
  A/Louisiana/13/2017 [H3N2] - Day 1 | 54 [37 to 69] | 68 [50 to 82] | 43 [27 to 59] | 56 [40 to 72] | 47 [31 to 64] | 52 [36 to 68]
  A/Michigan/84/2016 [H3N2] - Day 1 | 78 [62 to 89] | 81 [65 to 92] | 68 [51 to 81] | 80 [65 to 91] | 66 [49 to 80] | 83 [69 to 93]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 8 | 98 [87 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 100 [91 to 100] | 93 [80 to 98] | 92 [79 to 98] | 100 [92 to 100]
  A/Aksaray/4048/2016 [H3N2] - Day 8 | 98 [87 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 98 [87 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 97 [86 to NA] — Value is NA because it's >99 but <100 | 100 [92 to 100]
  A/Kenya/105/2017 [H3N2] - Day 8 | 98 [87 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 98 [87 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 97 [86 to NA] — Value is NA because it's >99 but <100 | 100 [92 to 100]
  A/Louisiana/13/2017 [H3N2] - Day 8 | 88 [74 to 96] | 95 [82 to NA] — Value is NA because it's >99 but <100 | 88 [73 to 96] | 88 [74 to 96] | 89 [75 to 97] | 86 [71 to 95]
  A/Michigan/84/2016 [H3N2] - Day 8 | 93 [80 to 98] | 92 [78 to 98] | 93 [80 to 98] | 88 [74 to 96] | 79 [63 to 90] | 93 [81 to 99]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 29 | 95 [83 to NA] — Value is NA because it's >99 but <100 | 100 [90 to 100] | 97 [87 to NA] — Value is NA because it's >99 but <100 | 98 [87 to NA] — Value is NA because it's >99 but <100 | 95 [82 to NA] — Value is NA because it's >99 but <100 | 98 [87 to NA] — Value is NA because it's >99 but <100
  A/Aksaray/4048/2016 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Aksaray/4048/2016 [H3N2] - Day 29 | 95 [83 to NA] — Value is NA because it's >99 but <100 | 100 [90 to 100] | 97 [87 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100]
  A/Kenya/105/2017 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Kenya/105/2017 [H3N2] - Day 29 | 98 [87 to NA] — Value is NA because it's >99 but <100 | 100 [90 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100]
  A/Louisiana/13/2017 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Louisiana/13/2017 [H3N2] - Day 29 | 90 [77 to 97] | 97 [85 to NA] — Value is NA because it's >99 but <100 | 95 [83 to NA] — Value is NA because it's >99 but <100 | 95 [83 to NA] — Value is NA because it's >99 but <100 | 97 [86 to NA] — Value is NA because it's >99 but <100 | 95 [83 to NA] — Value is NA because it's >99 but <100
  A/Michigan/84/2016 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Michigan/84/2016 [H3N2] - Day 29 | 98 [87 to NA] — Value is NA because it's >99 but <100 | 94 [81 to NA] — Value is NA because it's >99 but <100 | 87 [73 to 96] | 90 [76 to 97] | 78 [62 to 90] | 90 [77 to 97]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 57 | 83 [67 to 93] | 100 [91 to 100] | 92 [79 to 98] | 95 [83 to NA] — Value is NA because it's >99 but <100 | 95 [82 to NA] — Value is NA because it's >99 but <100 | 95 [83 to NA] — Value is NA because it's >99 but <100
  A/Aksaray/4048/2016 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Aksaray/4048/2016 [H3N2] - Day 57 | 90 [76 to 97] | 100 [91 to 100] | 97 [86 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 97 [86 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100]
  A/Kenya/105/2017 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Kenya/105/2017 [H3N2] - Day 57 | 95 [83 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 95 [82 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100]
  A/Louisiana/13/2017 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Louisiana/13/2017 [H3N2] - Day 57 | 78 [62 to 89] | 95 [82 to NA] — Value is NA because it's >99 but <100 | 82 [66 to 92] | 95 [83 to NA] — Value is NA because it's >99 but <100 | 92 [78 to 98] | 90 [77 to 97]
  A/Michigan/84/2016 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Michigan/84/2016 [H3N2] - Day 57 | 83 [67 to 93] | 89 [75 to 97] | 82 [66 to 92] | 88 [73 to 96] | 76 [59 to 88] | 88 [74 to 96]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 90 | 85 [71 to 94] | 100 [90 to 100] | 92 [79 to 98] | 97 [87 to NA] — Value is NA because it's >99 but <100 | 95 [82 to NA] — Value is NA because it's >99 but <100 | 95 [83 to NA] — Value is NA because it's >99 but <100
  A/Aksaray/4048/2016 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Aksaray/4048/2016 [H3N2] - Day 90 | 90 [77 to 97] | 100 [90 to 100] | 92 [79 to 98] | 100 [91 to 100] | 97 [86 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100]
  A/Kenya/105/2017 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Kenya/105/2017 [H3N2] - Day 90 | 95 [83 to NA] — Value is NA because it's >99 but <100 | 100 [90 to 100] | 95 [82 to NA] — Value is NA because it's >99 but <100 | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100]
  A/Louisiana/13/2017 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Louisiana/13/2017 [H3N2] - Day 90 | 78 [62 to 89] | 94 [81 to NA] — Value is NA because it's >99 but <100 | 74 [57 to 87] | 97 [87 to NA] — Value is NA because it's >99 but <100 | 89 [75 to 97] | 93 [80 to 98]
  A/Michigan/84/2016 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Michigan/84/2016 [H3N2] - Day 90 | 83 [68 to 93] | 89 [74 to 97] | 79 [63 to 90] | 95 [83 to NA] — Value is NA because it's >99 but <100 | 76 [59 to 88] | 85 [70 to 94]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 118 | 94 [81 to NA] — Value is NA because it's >99 but <100 | 100 [88 to 100] | 94 [80 to NA] — Value is NA because it's >99 but <100 | 100 [90 to 100] | 97 [84 to NA] — Value is NA because it's >99 but <100 | 100 [90 to 100]
  A/Aksaray/4048/2016 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Aksaray/4048/2016 [H3N2] - Day 118 | 100 [90 to 100] | 100 [88 to 100] | 94 [80 to NA] — Value is NA because it's >99 but <100 | 100 [90 to 100] | 100 [89 to 100] | 100 [90 to 100]
  A/Kenya/105/2017 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Kenya/105/2017 [H3N2] - Day 118 | 100 [90 to 100] | 100 [88 to 100] | 97 [85 to NA] — Value is NA because it's >99 but <100 | 100 [90 to 100] | 100 [89 to 100] | 100 [90 to 100]
  A/Louisiana/13/2017 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Louisiana/13/2017 [H3N2] - Day 118 | 97 [85 to NA] — Value is NA because it's >99 but <100 | 97 [83 to NA] — Value is NA because it's >99 but <100 | 94 [80 to NA] — Value is NA because it's >99 but <100 | 100 [90 to 100] | 97 [84 to NA] — Value is NA because it's >99 but <100 | 100 [90 to 100]
  A/Michigan/84/2016 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Michigan/84/2016 [H3N2] - Day 118 | 94 [81 to NA] — Value is NA because it's >99 but <100 | 93 [78 to NA] — Value is NA because it's >99 but <100 | 88 [73 to 97] | 97 [85 to NA] — Value is NA because it's >99 but <100 | 84 [67 to 95] | 91 [76 to 98]

52. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in Hemagglutination Inhibition (HAI) Titers Against Heterologous H1 and H3 Influenza Strains
Description: Blood was collected for HAI assay which was conducted with the heterologous H1 and H3 influenza viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. Fold-rises from baseline were calculated as the Day 8 (or Day 29, Day 57, Day 90, Day 118) titer divided by the baseline titers for each participant. The geometric mean of these fold rises was then calculated to obtain the GMFR.
Time Frame: Day 8, Day 29, Day 57, Day 90, Day 118
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 41 | 38 | 42
fold rise
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 8 | 3.2 [2.2 to 4.6] | 3.9 [2.5 to 6.0] | 4.2 [2.6 to 6.8] | 3.0 [2.1 to 4.3] | 4.5 [2.9 to 7.1] | 4.7 [3.1 to 7.2]
  A/Aksaray/4048/2016 [H3N2] - Day 8 | 2.4 [1.8 to 3.4] | 3.2 [2.1 to 5.0] | 3.4 [2.2 to 5.2] | 2.8 [2.0 to 4.0] | 4.9 [3.2 to 7.7] | 3.9 [2.7 to 5.5]
  A/Kenya/105/2017 [H3N2] - Day 8 | 2.9 [2.1 to 4.1] | 3.9 [2.6 to 6.0] | 3.7 [2.4 to 5.7] | 3.0 [2.1 to 4.1] | 5.8 [3.8 to 9.0] | 4.8 [3.4 to 6.7]
  A/Louisiana/13/2017 [H3N2] - Day 8 | 3.5 [2.5 to 4.8] | 4.0 [2.8 to 5.8] | 4.1 [2.8 to 5.9] | 3.0 [2.2 to 4.1] | 4.5 [3.2 to 6.4] | 3.4 [2.4 to 4.7]
  A/Michigan/84/2016 [H3N2] - Day 8 | 1.4 [1.2 to 1.7] | 1.7 [1.4 to 2.1] | 1.5 [1.3 to 1.9] | 1.3 [1.1 to 1.5] | 1.7 [1.3 to 2.4] | 1.4 [1.2 to 1.7]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 29 | 3.1 [2.2 to 4.5] | 3.4 [2.2 to 5.2] | 4.2 [2.7 to 6.6] | 4.6 [3.1 to 6.7] | 5.2 [3.6 to 7.6] | 5.5 [3.7 to 8.3]
  A/Aksaray/4048/2016 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Aksaray/4048/2016 [H3N2] - Day 29 | 2.4 [1.7 to 3.3] | 2.7 [1.8 to 4.0] | 3.1 [2.1 to 4.5] | 3.8 [2.6 to 5.5] | 5.3 [3.5 to 8.0] | 4.4 [3.0 to 6.5]
  A/Kenya/105/2017 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Kenya/105/2017 [H3N2] - Day 29 | 4.2 [2.9 to 5.9] | 4.8 [3.2 to 7.2] | 4.9 [3.3 to 7.1] | 6.1 [4.2 to 8.8] | 9.5 [6.2 to 14.5] | 8.1 [5.8 to 11.2]
  A/Louisiana/13/2017 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Louisiana/13/2017 [H3N2] - Day 29 | 3.8 [2.8 to 5.1] | 4.2 [3.0 to 5.9] | 4.6 [3.4 to 6.3] | 5.0 [3.6 to 7.0] | 5.7 [4.1 to 7.8] | 5.1 [3.6 to 7.3]
  A/Michigan/84/2016 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Michigan/84/2016 [H3N2] - Day 29 | 1.5 [1.3 to 1.8] | 1.6 [1.3 to 1.9] | 1.5 [1.3 to 1.7] | 1.7 [1.3 to 2.1] | 1.8 [1.3 to 2.4] | 1.6 [1.3 to 2.0]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 57 | 2.0 [1.4 to 2.8] | 2.4 [1.6 to 3.5] | 2.6 [1.7 to 4.0] | 3.6 [2.5 to 5.1] | 3.9 [2.7 to 5.6] | 4.2 [2.9 to 6.3]
  A/Aksaray/4048/2016 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Aksaray/4048/2016 [H3N2] - Day 57 | 2.0 [1.5 to 2.8] | 2.4 [1.6 to 3.6] | 2.7 [1.9 to 3.9] | 3.6 [2.5 to 5.1] | 5.1 [3.3 to 7.6] | 4.0 [2.8 to 5.6]
  A/Kenya/105/2017 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Kenya/105/2017 [H3N2] - Day 57 | 2.9 [2.2 to 3.9] | 3.5 [2.5 to 5.0] | 3.6 [2.5 to 5.1] | 4.2 [3.0 to 5.9] | 5.8 [3.9 to 8.6] | 5.0 [3.7 to 6.9]
  A/Louisiana/13/2017 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Louisiana/13/2017 [H3N2] - Day 57 | 2.6 [2.0 to 3.4] | 2.8 [2.0 to 3.8] | 3.3 [2.4 to 4.5] | 3.9 [3.0 to 5.2] | 4.0 [3.0 to 5.3] | 3.6 [2.7 to 4.9]
  A/Michigan/84/2016 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Michigan/84/2016 [H3N2] - Day 57 | 1.2 [1.0 to 1.3] | 1.3 [1.1 to 1.7] | 1.2 [1.1 to 1.4] | 1.5 [1.2 to 1.9] | 1.4 [1.1 to 1.8] | 1.4 [1.1 to 1.8]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 90 | 1.9 [1.4 to 2.5] | 2.1 [1.5 to 3.1] | 2.4 [1.7 to 3.5] | 3.1 [2.3 to 4.4] | 3.5 [2.5 to 5.1] | 3.6 [2.5 to 5.3]
  A/Aksaray/4048/2016 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Aksaray/4048/2016 [H3N2] - Day 90 | 1.9 [1.5 to 2.6] | 1.9 [1.4 to 2.7] | 2.3 [1.6 to 3.2] | 2.9 [2.1 to 4.0] | 3.9 [2.6 to 5.7] | 3.2 [2.3 to 4.4]
  A/Kenya/105/2017 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Kenya/105/2017 [H3N2] - Day 90 | 3.2 [2.4 to 4.2] | 3.8 [2.6 to 5.4] | 3.8 [2.6 to 5.4] | 5.1 [3.6 to 7.1] | 7.1 [4.8 to 10.6] | 5.7 [4.1 to 7.9]
  A/Louisiana/13/2017 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Louisiana/13/2017 [H3N2] - Day 90 | 2.4 [1.9 to 3.1] | 2.5 [1.9 to 3.4] | 2.9 [2.2 to 3.9] | 3.8 [2.9 to 4.8] | 3.9 [2.9 to 5.2] | 3.5 [2.5 to 4.8]
  A/Michigan/84/2016 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Michigan/84/2016 [H3N2] - Day 90 | 1.2 [1.1 to 1.4] | 1.4 [1.2 to 1.7] | 1.3 [1.1 to 1.5] | 1.6 [1.3 to 1.9] | 1.4 [1.1 to 1.7] | 1.5 [1.2 to 1.9]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 118 | 4.1 [2.9 to 5.9] | 2.8 [1.9 to 4.1] | 4.9 [3.2 to 7.3] | 6.8 [4.3 to 10.7] | 8.1 [5.1 to 12.9] | 6.6 [4.5 to 9.6]
  A/Aksaray/4048/2016 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Aksaray/4048/2016 [H3N2] - Day 118 | 5.1 [3.5 to 7.4] | 3.1 [2.2 to 4.5] | 6.5 [4.3 to 9.8] | 8.1 [5.4 to 12.0] | 11.0 [6.6 to 18.1] | 6.9 [4.9 to 9.6]
  A/Kenya/105/2017 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Kenya/105/2017 [H3N2] - Day 118 | 4.8 [3.4 to 6.9] | 3.1 [2.2 to 4.2] | 5.2 [3.4 to 7.8] | 7.8 [5.1 to 12.0] | 10.4 [6.8 to 15.9] | 7.5 [5.4 to 10.6]
  A/Louisiana/13/2017 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Louisiana/13/2017 [H3N2] - Day 118 | 9.8 [6.2 to 15.5] | 4.1 [2.8 to 6.0] | 9.7 [6.5 to 14.6] | 15.5 [9.5 to 25.4] | 16.5 [10.2 to 26.7] | 11.1 [7.7 to 15.9]
  A/Michigan/84/2016 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Michigan/84/2016 [H3N2] - Day 118 | 1.7 [1.4 to 2.0] | 1.6 [1.3 to 2.1] | 2.0 [1.6 to 2.4] | 2.9 [2.2 to 3.7] | 2.8 [1.9 to 4.0] | 2.4 [1.9 to 3.0]

53. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Neuraminidase Inhibition (NAI) Against Heterologous N1 and N2 Neuraminidase (NA) Antigens for the Fluzone Study Arms
Description: Blood was collected for NAI assay which was conducted with the heterologous N1 and N2 NA viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at Day 1, Day 8, Day 29, Day 57, Day 90, and Day 118 Post first study vaccination.
Time Frame: Day 1, Day 8, Day 29, Day 57, Day 90, Day 118
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55
Number analyzed (Participants) | 41 | 37 | 40
titer
  A/Townsville/51/2016 H6N2 - Day 1 | 16.6 [12.8 to 21.5] | 20.2 [15.5 to 26.3] | 14.5 [10.7 to 19.6]
  A/Townsville/51/2016 H6N2 - Day 8 | 34.1 [27.3 to 42.5] | 49.6 [39.8 to 61.8] | 35.1 [27.8 to 44.4]
  A/Townsville/51/2016 H6N2 - Day 29: number analyzed (Participants) | 41 | 36 | 39
  A/Townsville/51/2016 H6N2 - Day 29 | 21.9 [17.8 to 27.1] | 35.6 [27.5 to 46.1] | 23.3 [17.6 to 30.7]
  A/Townsville/51/2016 H6N2 - Day 57: number analyzed (Participants) | 40 | 37 | 38
  A/Townsville/51/2016 H6N2 - Day 57 | 26.2 [20.7 to 33.1] | 37.1 [29.0 to 47.4] | 24.2 [17.9 to 32.7]
  A/Townsville/51/2016 H6N2 - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Townsville/51/2016 H6N2 - Day 90 | 22.7 [17.9 to 28.8] | 34.6 [25.9 to 46.2] | 24.0 [17.4 to 33.1]
  A/Townsville/51/2016 H6N2 - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Townsville/51/2016 H6N2 - Day 118 | 32.4 [24.7 to 42.4] | 39.1 [29.3 to 52.1] | 29.5 [21.3 to 40.8]
  A/Cameroon/9766/2017 H6N1 - Day 1 | 48.2 [33.0 to 70.4] | 47.3 [33.5 to 67.0] | 40.0 [26.7 to 59.8]
  A/Cameroon/9766/2017 H6N1 - Day 8 | 104.0 [79.2 to 136.5] | 117.5 [91.0 to 151.6] | 91.1 [66.5 to 124.7]
  A/Cameroon/9766/2017 H6N1 - Day 29: number analyzed (Participants) | 41 | 36 | 39
  A/Cameroon/9766/2017 H6N1 - Day 29 | 80.7 [60.4 to 107.8] | 95.1 [69.6 to 130.1] | 68.2 [49.9 to 93.1]
  A/Cameroon/9766/2017 H6N1 - Day 57: number analyzed (Participants) | 40 | 37 | 38
  A/Cameroon/9766/2017 H6N1 - Day 57 | 76.6 [55.3 to 106.1] | 76.3 [55.2 to 105.6] | 53.6 [37.0 to 77.6]
  A/Cameroon/9766/2017 H6N1 - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Cameroon/9766/2017 H6N1 - Day 90 | 69.3 [49.7 to 96.6] | 66.6 [47.0 to 94.5] | 48.9 [33.9 to 70.4]
  A/Cameroon/9766/2017 H6N1 - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Cameroon/9766/2017 H6N1 - Day 118 | 83.1 [58.2 to 118.8] | 81.9 [56.1 to 119.5] | 62.0 [42.9 to 89.6]
  A/Hubeiwujiagang/SWL310/2013 - Day 1 | 108.5 [73.7 to 159.7] | 105.0 [74.1 to 148.6] | 92.7 [60.6 to 141.7]
  A/Hubeiwujiagang/SWL310/2013 - Day 8 | 197.7 [147.4 to 265.0] | 191.2 [141.7 to 257.8] | 167.1 [120.8 to 231.1]
  A/Hubeiwujiagang/SWL310/2013 - Day 29: number analyzed (Participants) | 41 | 36 | 39
  A/Hubeiwujiagang/SWL310/2013 - Day 29 | 143.3 [104.2 to 197.3] | 161.5 [112.3 to 232.4] | 128.1 [91.0 to 180.4]
  A/Hubeiwujiagang/SWL310/2013 - Day 57: number analyzed (Participants) | 40 | 37 | 38
  A/Hubeiwujiagang/SWL310/2013 - Day 57 | 144.2 [103.7 to 200.5] | 151.3 [105.8 to 216.3] | 117.3 [80.0 to 172.7]
  A/Hubeiwujiagang/SWL310/2013 - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Hubeiwujiagang/SWL310/2013 - Day 90 | 139.8 [99.2 to 196.8] | 145.3 [100.2 to 210.7] | 113.1 [76.9 to 166.5]
  A/Hubeiwujiagang/SWL310/2013 - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Hubeiwujiagang/SWL310/2013 - Day 118 | 141.2 [98.8 to 201.7] | 160.0 [108.1 to 236.8] | 130.5 [90.0 to 189.3]
  A/Oman/5532/2017 H6N1 - Day 1 | 37.7 [26.4 to 53.9] | 35.1 [25.1 to 49.0] | 31.7 [20.9 to 48.0]
  A/Oman/5532/2017 H6N1 - Day 8 | 80.7 [59.6 to 109.2] | 100.2 [75.3 to 133.3] | 75.3 [55.8 to 101.5]
  A/Oman/5532/2017 H6N1 - Day 29: number analyzed (Participants) | 41 | 36 | 39
  A/Oman/5532/2017 H6N1 - Day 29 | 65.9 [49.7 to 87.3] | 74.8 [55.4 to 101.0] | 54.1 [39.5 to 74.1]
  A/Oman/5532/2017 H6N1 - Day 57: number analyzed (Participants) | 40 | 37 | 38
  A/Oman/5532/2017 H6N1 - Day 57 | 63.3 [45.8 to 87.6] | 62.1 [44.2 to 87.4] | 48.4 [33.0 to 71.2]
  A/Oman/5532/2017 H6N1 - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Oman/5532/2017 H6N1 - Day 90 | 57.5 [40.1 to 82.6] | 53.9 [38.1 to 76.3] | 40.4 [27.7 to 58.9]
  A/Oman/5532/2017 H6N1 - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Oman/5532/2017 H6N1 - Day 118 | 72.7 [51.1 to 103.3] | 70.5 [47.6 to 104.2] | 54.9 [38.0 to 79.2]
  A/Aksaray/4048/2016 H6N2 - Day 1 | 33.2 [23.7 to 46.5] | 45.2 [32.7 to 62.4] | 28.5 [19.3 to 42.2]
  A/Aksaray/4048/2016 H6N2 - Day 8 | 72.9 [57.1 to 93.1] | 117.5 [93.9 to 147.0] | 81.4 [62.4 to 106.2]
  A/Aksaray/4048/2016 H6N2 - Day 29: number analyzed (Participants) | 41 | 36 | 39
  A/Aksaray/4048/2016 H6N2 - Day 29 | 59.5 [47.2 to 75.1] | 102.8 [79.6 to 132.6] | 62.9 [47.2 to 84.0]
  A/Aksaray/4048/2016 H6N2 - Day 57: number analyzed (Participants) | 40 | 37 | 38
  A/Aksaray/4048/2016 H6N2 - Day 57 | 51.9 [39.6 to 67.9] | 90.4 [70.9 to 115.1] | 56.6 [40.6 to 78.7]
  A/Aksaray/4048/2016 H6N2 - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Aksaray/4048/2016 H6N2 - Day 90 | 60.0 [45.2 to 79.7] | 96.1 [74.8 to 123.3] | 63.1 [43.8 to 90.8]
  A/Aksaray/4048/2016 H6N2 - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Aksaray/4048/2016 H6N2 - Day 118 | 69.9 [52.3 to 93.5] | 91.9 [69.4 to 121.8] | 68.0 [48.4 to 95.3]
  A/Louisiana/13/2017 H6N2 - Day 1 | 124.2 [94.1 to 163.8] | 154.1 [109.9 to 216.0] | 126.6 [86.8 to 184.7]
  A/Louisiana/13/2017 H6N2 - Day 8 | 181.6 [137.6 to 239.7] | 317.0 [247.9 to 405.4] | 216.7 [161.8 to 290.1]
  A/Louisiana/13/2017 H6N2 - Day 29: number analyzed (Participants) | 41 | 36 | 39
  A/Louisiana/13/2017 H6N2 - Day 29 | 181.6 [140.7 to 234.4] | 305.0 [230.0 to 404.3] | 201.6 [149.2 to 272.4]
  A/Louisiana/13/2017 H6N2 - Day 57: number analyzed (Participants) | 40 | 37 | 38
  A/Louisiana/13/2017 H6N2 - Day 57 | 153.2 [117.4 to 199.9] | 250.8 [188.1 to 334.6] | 183.5 [131.6 to 225.8]
  A/Louisiana/13/2017 H6N2 - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Louisiana/13/2017 H6N2 - Day 90 | 144.6 [111.8 to 186.9] | 215.6 [162.7 to 285.9] | 157.1 [113.3 to 217.8]
  A/Louisiana/13/2017 H6N2 - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Louisiana/13/2017 H6N2 - Day 118 | 167.9 [127.2 to 221.6] | 266.0 [198.3 to 356.8] | 212.8 [142.8 to 317.2]

54. Secondary Outcome: Ratio of Geometric Mean Titers (GMTs) of Serum Neuraminidase Inhibition (NAI) Against Heterologous N1 and N2 Neuraminidase (NA) Antigens Between Adjuvanted and Unadjuvanted Study Arms for the Fluzone Study Arms
Description: Blood was collected for NAI assay which was conducted with the heterologous N1 and N2 NA viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at Day 1, Day 8, Day 29, Day 57, Day 90, and Day 118 Post first study vaccination and the ratio of these GMTs between adjuvanted and unadjuvanted study arms were calculated.
  The unadjuvanted Fluzone study arm is considered a reference group for the analysis of ratio of GMTs.
  Ratio of GMTs is defined as the ratio of the GMT from the adjuvanted group divided by the GMT from the corresponding unadjuvanted group.
Time Frame: Day 1, Day 8, Day 29, Day 57, Day 90, Day 118
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: ratio of GMT
Arm/Group | Fluzone + AF03 | Fluzone + CpG55
Number analyzed (Participants) | 37 | 40
ratio of GMT
  A/Townsville/51/2016 H6N2 - Day 1 | 1.2 [0.8 to 1.7] | 0.9 [0.6 to 1.3]
  A/Cameroon/9766/2017 H6N1 - Day 1 | 1.0 [0.6 to 1.6] | 0.8 [0.5 to 1.4]
  A/Hubeiwujiagang/SWL310/2013 - Day 1 | 1.0 [0.6 to 1.6] | 0.9 [0.5 to 1.5]
  A/Oman/5532/2017 H6N1 - Day 1 | 0.9 [0.6 to 1.5] | 0.8 [0.5 to 1.4]
  A/Aksaray/4048/2016 H6N2 - Day 1 | 1.4 [0.9 to 2.2] | 0.9 [0.5 to 1.4]
  A/Townsville/51/2016 H6N2 - Day 8 | 1.5 [1.1 to 2.0] | 1.0 [0.8 to 1.4]
  A/Cameroon/9766/2017 H6N1 - Day 8 | 1.1 [0.8 to 1.6] | 0.9 [0.6 to 1.3]
  A/Hubeiwujiagang/SWL310/2013 - Day 8 | 1.0 [0.6 to 1.5] | 0.8 [0.5 to 1.3]
  A/Oman/5532/2017 H6N1 - Day 8 | 1.2 [0.8 to 1.9] | 0.9 [0.6 to 1.4]
  A/Aksaray/4048/2016 H6N2 - Day 8 | 1.6 [1.2 to 2.2] | 1.1 [0.8 to 1.6]
  A/Townsville/51/2016 H6N2 - Day 29: number analyzed (Participants) | 36 | 39
  A/Townsville/51/2016 H6N2 - Day 29 | 1.6 [1.2 to 2.3] | 1.1 [0.8 to 1.5]
  A/Cameroon/9766/2017 H6N1 - Day 29: number analyzed (Participants) | 36 | 39
  A/Cameroon/9766/2017 H6N1 - Day 29 | 1.2 [0.8 to 1.8] | 0.8 [0.6 to 1.3]
  A/Hubeiwujiagang/SWL310/2013 - Day 29: number analyzed (Participants) | 36 | 39
  A/Hubeiwujiagang/SWL310/2013 - Day 29 | 1.1 [0.7 to 1.8] | 0.9 [0.6 to 1.4]
  A/Oman/5532/2017 H6N1 - Day 29: number analyzed (Participants) | 36 | 39
  A/Oman/5532/2017 H6N1 - Day 29 | 1.1 [0.8 to 1.7] | 0.8 [0.5 to 1.2]
  A/Aksaray/4048/2016 H6N2 - Day 29: number analyzed (Participants) | 36 | 39
  A/Aksaray/4048/2016 H6N2 - Day 29 | 1.7 [1.2 to 2.4] | 1.1 [0.7 to 1.5]
  A/Townsville/51/2016 H6N2 - Day 57: number analyzed (Participants) | 37 | 38
  A/Townsville/51/2016 H6N2 - Day 57 | 1.4 [1.0 to 2.0] | 0.9 [0.6 to 1.3]
  A/Cameroon/9766/2017 H6N1 - Day 57: number analyzed (Participants) | 37 | 38
  A/Cameroon/9766/2017 H6N1 - Day 57 | 1.0 [0.6 to 1.6] | 0.7 [0.4 to 1.1]
  A/Hubeiwujiagang/SWL310/2013 - Day 57: number analyzed (Participants) | 37 | 38
  A/Hubeiwujiagang/SWL310/2013 - Day 57 | 1.0 [0.7 to 1.7] | 0.8 [0.5 to 1.3]
  A/Oman/5532/2017 H6N1 - Day 57: number analyzed (Participants) | 37 | 38
  A/Oman/5532/2017 H6N1 - Day 57 | 1.0 [0.6 to 1.6] | 0.8 [0.5 to 1.3]
  A/Aksaray/4048/2016 H6N2 - Day 57: number analyzed (Participants) | 37 | 38
  A/Aksaray/4048/2016 H6N2 - Day 57 | 1.7 [1.2 to 2.5] | 1.1 [0.7 to 1.7]
  A/Townsville/51/2016 H6N2 - Day 90: number analyzed (Participants) | 36 | 38
  A/Townsville/51/2016 H6N2 - Day 90 | 1.5 [1.1 to 2.2] | 1.1 [0.7 to 1.6]
  A/Cameroon/9766/2017 H6N1 - Day 90: number analyzed (Participants) | 36 | 38
  A/Cameroon/9766/2017 H6N1 - Day 90 | 1.0 [0.6 to 1.5] | 0.7 [0.4 to 1.1]
  A/Hubeiwujiagang/SWL310/2013 - Day 90: number analyzed (Participants) | 36 | 38
  A/Hubeiwujiagang/SWL310/2013 - Day 90 | 1.0 [0.6 to 1.7] | 0.8 [0.5 to 1.3]
  A/Oman/5532/2017 H6N1 - Day 90: number analyzed (Participants) | 36 | 38
  A/Oman/5532/2017 H6N1 - Day 90 | 0.9 [0.6 to 1.5] | 0.7 [0.4 to 1.2]
  A/Aksaray/4048/2016 H6N2 - Day 90: number analyzed (Participants) | 36 | 38
  A/Aksaray/4048/2016 H6N2 - Day 90 | 1.6 [1.1 to 2.3] | 1.1 [0.7 to 1.7]
  A/Townsville/51/2016 H6N2 - Day 118: number analyzed (Participants) | 30 | 34
  A/Townsville/51/2016 H6N2 - Day 118 | 1.2 [0.8 to 1.8] | 0.9 [0.6 to 1.4]
  A/Cameroon/9766/2017 H6N1 - Day 118: number analyzed (Participants) | 30 | 34
  A/Cameroon/9766/2017 H6N1 - Day 118 | 1.0 [0.6 to 1.6] | 0.7 [0.5 to 1.2]
  A/Hubeiwujiagang/SWL310/2013 - Day 118: number analyzed (Participants) | 30 | 34
  A/Hubeiwujiagang/SWL310/2013 - Day 118 | 1.1 [0.7 to 1.9] | 0.9 [0.6 to 1.5]
  A/Oman/5532/2017 H6N1 - Day 118: number analyzed (Participants) | 30 | 30
  A/Oman/5532/2017 H6N1 - Day 118 | 1.0 [0.6 to 1.6] | 0.8 [0.5 to 1.2]
  A/Aksaray/4048/2016 H6N2 - Day 118: number analyzed (Participants) | 30 | 34
  A/Aksaray/4048/2016 H6N2 - Day 118 | 1.3 [0.9 to 2.0] | 1.0 [0.6 to 1.5]
  A/Louisiana/13/2017 H6N2 - Day 1 | 1.2 [0.8 to 1.9] | 1.0 [0.6 to 1.6]
  A/Louisiana/13/2017 H6N2 - Day 8 | 1.7 [1.2 to 2.5] | 1.2 [0.8 to 1.8]
  A/Louisiana/13/2017 H6N2 - Day 29: number analyzed (Participants) | 36 | 39
  A/Louisiana/13/2017 H6N2 - Day 29 | 1.7 [1.2 to 2.4] | 1.1 [0.8 to 1.6]
  A/Louisiana/13/2017 H6N2 - Day 57: number analyzed (Participants) | 37 | 38
  A/Louisiana/13/2017 H6N2 - Day 57 | 1.6 [1.1 to 2.4] | 1.2 [0.8 to 1.8]
  A/Louisiana/13/2017 H6N2 - Day 90: number analyzed (Participants) | 36 | 38
  A/Louisiana/13/2017 H6N2 - Day 90 | 1.5 [1.0 to 2.2] | 1.1 [0.7 to 1.6]
  A/Louisiana/13/2017 H6N2 - Day 118: number analyzed (Participants) | 30 | 34
  A/Louisiana/13/2017 H6N2 - Day 118 | 1.6 [1.1 to 2.4] | 1.3 [0.8 to 2.0]

55. Secondary Outcome: Percentage of Participants Achieving Neuraminidase Inhibition (NAI) Titer Seroconversion Against Heterologous N1 and N2 Neuraminidase (NA) Antigens for the Fluzone Study Arms
Description: Blood was collected for NAI assay which was conducted with the heterologous N1 and N2 NA viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. NAI seroconversion was defined as >4 four-fold rise in post-vaccination antibody titer at Day 8, 29, 57, 90, and 118.
Time Frame: Day 8, Day 29, Day 57, Day 90, Day 118
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55
Number analyzed (Participants) | 41 | 37 | 40
percentage of participants
  A/Townsville/51/2016 H6N2 - Day 8 | 17 [7 to 32] | 27 [14 to 44] | 25 [13 to 41]
  A/Cameroon/9766/2017 H6N1 - Day 8 | 24 [12 to 40] | 32 [18 to 50] | 38 [23 to 54]
  A/Hubeiwujiagang/SWL310/2013 - Day 8 | 17 [7 to 32] | 14 [5 to 29] | 18 [7 to 33]
  A/Oman/5532/2017 H6N1 - Day 8 | 27 [14 to 43] | 41 [25 to 58] | 28 [15 to 44]
  A/Aksaray/4048/2016 H6N2 - Day 8 | 29 [16 to 46] | 38 [22 to 55] | 38 [23 to 54]
  A/Louisiana/13/2017 H6N2 - Day 8 | 10 [3 to 23] | 27 [14 to 44] | 10 [3 to 24]
  A/Townsville/51/2016 H6N2 - Day 29: number analyzed (Participants) | 41 | 36 | 39
  A/Townsville/51/2016 H6N2 - Day 29 | 10 [3 to 23] | 14 [5 to 29] | 5 [NA to 17] — Value is NA because it's >0 but <1
  A/Cameroon/9766/2017 H6N1 - Day 29: number analyzed (Participants) | 41 | 36 | 39
  A/Cameroon/9766/2017 H6N1 - Day 29 | 15 [6 to 29] | 22 [10 to 39] | 18 [8 to 34]
  A/Hubeiwujiagang/SWL310/2013 - Day 29: number analyzed (Participants) | 41 | 36 | 39
  A/Hubeiwujiagang/SWL310/2013 - Day 29 | 5 [NA to 17] — Value is NA because it's >0 but <1 | 14 [5 to 29] | 3 [NA to 13] — Value is NA because it's >0 but <1
  A/Oman/5532/2017 H6N1 - Day 29: number analyzed (Participants) | 41 | 36 | 39
  A/Oman/5532/2017 H6N1 - Day 29 | 17 [7 to 32] | 19 [8 to 36] | 18 [8 to 34]
  A/Aksaray/4048/2016 H6N2 - Day 29: number analyzed (Participants) | 41 | 36 | 39
  A/Aksaray/4048/2016 H6N2 - Day 29 | 17 [7 to 32] | 25 [12 to 42] | 33 [19 to 50]
  A/Louisiana/13/2017 H6N2 - Day 29: number analyzed (Participants) | 41 | 36 | 39
  A/Louisiana/13/2017 H6N2 - Day 29 | 7 [2 to 20] | 19 [8 to 36] | 13 [4 to 27]
  A/Townsville/51/2016 H6N2 - Day 57: number analyzed (Participants) | 40 | 37 | 38
  A/Townsville/51/2016 H6N2 - Day 57 | 8 [2 to 20] | 11 [3 to 25] | 5 [NA to 18] — Value is NA because it's >0 but <1
  A/Cameroon/9766/2017 H6N1 - Day 57: number analyzed (Participants) | 40 | 37 | 38
  A/Cameroon/9766/2017 H6N1 - Day 57 | 8 [2 to 20] | 11 [3 to 25] | 5 [NA to 18] — Value is NA because it's >0 but <1
  A/Hubeiwujiagang/SWL310/2013 - Day 57: number analyzed (Participants) | 40 | 37 | 38
  A/Hubeiwujiagang/SWL310/2013 - Day 57 | 0 [0 to 9] | 8 [2 to 22] | 3 [NA to 14] — Value is NA because it's >0 but <1
  A/Oman/5532/2017 H6N1 - Day 57: number analyzed (Participants) | 40 | 37 | 38
  A/Oman/5532/2017 H6N1 - Day 57 | 13 [4 to 27] | 8 [2 to 22] | 11 [3 to 25]
  A/Aksaray/4048/2016 H6N2 - Day 57: number analyzed (Participants) | 40 | 37 | 38
  A/Aksaray/4048/2016 H6N2 - Day 57 | 5 [NA to 17] — Value is NA because it's >0 but <1 | 19 [8 to 35] | 18 [8 to 34]
  A/Louisiana/13/2017 H6N2 - Day 57: number analyzed (Participants) | 41 | 37 | 38
  A/Louisiana/13/2017 H6N2 - Day 57 | 3 [NA to 13] — Value is NA because it's >0 but <1 | 11 [3 to 25] | 8 [2 to 21]
  A/Townsville/51/2016 H6N2 - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Townsville/51/2016 H6N2 - Day 90 | 2 [NA to 13] — Value is NA because it's >0 but <1 | 6 [NA to 19] — Value is NA because it's >0 but <1 | 5 [NA to 18] — Value is NA because it's >0 but <1
  A/Cameroon/9766/2017 H6N1 - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Cameroon/9766/2017 H6N1 - Day 90 | 5 [NA to 17] — Value is NA because it's >0 but <1 | 11 [3 to 26] | 3 [NA to 14] — Value is NA because it's >0 but <1
  A/Hubeiwujiagang/SWL310/2013 - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Hubeiwujiagang/SWL310/2013 - Day 90 | 5 [NA to 17] — Value is NA because it's >0 but <1 | 11 [3 to 26] | 3 [NA to 14] — Value is NA because it's >0 but <1
  A/Oman/5532/2017 H6N1 - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Oman/5532/2017 H6N1 - Day 90 | 10 [3 to 23] | 6 [NA to 19] — Value is NA because it's >0 but <1 | 5 [NA to 18] — Value is NA because it's >0 but <1
  A/Aksaray/4048/2016 H6N2 - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Aksaray/4048/2016 H6N2 - Day 90 | 7 [2 to 20] | 17 [6 to 33] | 24 [11 to 40]
  A/Louisiana/13/2017 H6N2 - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Louisiana/13/2017 H6N2 - Day 90 | 2 [NA to 13] — Value is NA because it's >0 but <1 | 6 [NA to 19] — Value is NA because it's >0 but <1 | 3 [NA to 14] — Value is NA because it's >0 but <1
  A/Townsville/51/2016 H6N2 - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Townsville/51/2016 H6N2 - Day 118 | 22 [10 to 39] | 10 [2 to 27] | 18 [7 to 35]
  A/Cameroon/9766/2017 H6N1 - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Cameroon/9766/2017 H6N1 - Day 118 | 8 [2 to 22] | 13 [4 to 31] | 15 [5 to 31]
  A/Hubeiwujiagang/SWL310/2013 - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Hubeiwujiagang/SWL310/2013 - Day 118 | 11 [3 to 26] | 10 [2 to 27] | 15 [5 to 31]
  A/Oman/5532/2017 H6N1 - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Oman/5532/2017 H6N1 - Day 118 | 19 [8 to 36] | 17 [6 to 35] | 18 [7 to 35]
  A/Aksaray/4048/2016 H6N2 - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Aksaray/4048/2016 H6N2 - Day 118 | 25 [12 to 42] | 17 [6 to 35] | 32 [17 to 51]
  A/Louisiana/13/2017 H6N2 - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Louisiana/13/2017 H6N2 - Day 118 | 8 [2 to 22] | 10 [2 to 27] | 18 [7 to 35]

56. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in Neuraminidase Inhibition (NAI) Titers Against Heterologous N1 and N2 Neuraminidase (NA) Antigens for the Fluzone Study Arms
Description: Blood was collected for NAI assay which was conducted with the heterologous N1 and N2 NA viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. Fold-rises from baseline were calculated as the Day 8 (or Day 29, Day 57, Day 90, Day 118) titer divided by the baseline titers for each participant. The geometric mean of these fold rises was then calculated to obtain the GMFR.
Time Frame: Day 8, Day 29, Day 57, Day 90, Day 118
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55
Number analyzed (Participants) | 41 | 37 | 40
fold rise
  A/Townsville/51/2016 H6N2 - Day 8 | 2.1 [1.7 to 2.4] | 2.5 [2.0 to 3.1] | 2.4 [2.0 to 2.9]
  A/Cameroon/9766/2017 H6N1 - Day 8 | 2.2 [1.7 to 2.8] | 2.5 [2.0 to 3.1] | 2.3 [1.8 to 3.0]
  A/Hubeiwujiagang/SWL310/2013 - Day 8 | 1.8 [1.5 to 2.3] | 1.8 [1.5 to 2.2] | 1.8 [1.5 to 2.2]
  A/Oman/5532/2017 H6N1 - Day 8 | 2.1 [1.6 to 2.8] | 2.9 [2.3 to 3.6] | 2.4 [1.8 to 3.1]
  A/Aksaray/4048/2016 H6N2 - Day 8 | 2.2 [1.8 to 2.7] | 2.6 [2.0 to 3.4] | 2.9 [2.3 to 3.6]
  A/Louisiana/13/2017 H6N2 - Day 8 | 1.5 [1.2 to 1.8] | 2.1 [1.6 to 2.7] | 1.7 [1.4 to 2.1]
  A/Townsville/51/2016 H6N2 - Day 29: number analyzed (Participants) | 41 | 36 | 39
  A/Townsville/51/2016 H6N2 - Day 29 | 1.3 [1.1 to 1.5] | 1.7 [1.4 to 2.1] | 1.6 [1.4 to 1.9]
  A/Cameroon/9766/2017 H6N1 - Day 29: number analyzed (Participants) | 41 | 36 | 39
  A/Cameroon/9766/2017 H6N1 - Day 29 | 1.7 [1.4 to 2.1] | 2.0 [1.6 to 2.5] | 1.8 [1.5 to 2.2]
  A/Hubeiwujiagang/SWL310/2013 - Day 29: number analyzed (Participants) | 41 | 36 | 39
  A/Hubeiwujiagang/SWL310/2013 - Day 29 | 1.3 [1.1 to 1.5] | 1.6 [1.3 to 1.9] | 1.5 [1.3 to 1.7]
  A/Oman/5532/2017 H6N1 - Day 29: number analyzed (Participants) | 41 | 36 | 39
  A/Oman/5532/2017 H6N1 - Day 29 | 1.7 [1.4 to 2.1] | 2.1 [1.8 to 2.6] | 1.8 [1.5 to 2.2]
  A/Aksaray/4048/2016 H6N2 - Day 29: number analyzed (Participants) | 41 | 36 | 39
  A/Aksaray/4048/2016 H6N2 - Day 29 | 1.8 [1.5 to 2.1] | 2.2 [1.7 to 2.7] | 2.3 [1.9 to 2.8]
  A/Louisiana/13/2017 H6N2 - Day 29: number analyzed (Participants) | 41 | 36 | 39
  A/Louisiana/13/2017 H6N2 - Day 29 | 1.5 [1.3 to 1.7] | 1.9 [1.5 to 2.4] | 1.6 [1.4 to 1.9]
  A/Townsville/51/2016 H6N2 - Day 57: number analyzed (Participants) | 40 | 37 | 38
  A/Townsville/51/2016 H6N2 - Day 57 | 1.6 [1.4 to 1.9] | 1.8 [1.5 to 2.2] | 1.7 [1.5 to 2.0]
  A/Cameroon/9766/2017 H6N1 - Day 57: number analyzed (Participants) | 40 | 37 | 38
  A/Cameroon/9766/2017 H6N1 - Day 57 | 1.5 [1.3 to 1.8] | 1.6 [1.3 to 1.9] | 1.5 [1.2 to 1.7]
  A/Hubeiwujiagang/SWL310/2013 - Day 57: number analyzed (Participants) | 40 | 37 | 38
  A/Hubeiwujiagang/SWL310/2013 - Day 57 | 1.3 [1.1 to 1.5] | 1.4 [1.2 to 1.7] | 1.4 [1.2 to 1.6]
  A/Oman/5532/2017 H6N1 - Day 57: number analyzed (Participants) | 40 | 37 | 38
  A/Oman/5532/2017 H6N1 - Day 57 | 1.6 [1.4 to 1.9] | 1.8 [1.5 to 2.1] | 1.7 [1.4 to 2.0]
  A/Aksaray/4048/2016 H6N2 - Day 57: number analyzed (Participants) | 40 | 37 | 38
  A/Aksaray/4048/2016 H6N2 - Day 57 | 1.6 [1.4 to 1.8] | 2.0 [1.6 to 2.5] | 2.0 [1.7 to 2.3]
  A/Louisiana/13/2017 H6N2 - Day 57: number analyzed (Participants) | 40 | 37 | 38
  A/Louisiana/13/2017 H6N2 - Day 57 | 1.3 [1.1 to 1.5] | 1.6 [1.3 to 2.0] | 1.5 [1.3 to 1.8]
  A/Townsville/51/2016 H6N2 - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Townsville/51/2016 H6N2 - Day 90 | 1.4 [1.2 to 1.5] | 1.6 [1.4 to 1.9] | 1.7 [1.5 to 1.9]
  A/Cameroon/9766/2017 H6N1 - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Cameroon/9766/2017 H6N1 - Day 90 | 1.4 [1.2 to 1.7] | 1.4 [1.2 to 1.7] | 1.3 [1.1 to 1.5]
  A/Hubeiwujiagang/SWL310/2013 - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Hubeiwujiagang/SWL310/2013 - Day 90 | 1.3 [1.1 to 1.5] | 1.4 [1.2 to 1.7] | 1.3 [1.2 to 1.5]
  A/Oman/5532/2017 H6N1 - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Oman/5532/2017 H6N1 - Day 90 | 1.5 [1.3 to 1.8] | 1.5 [1.3 to 1.8] | 1.4 [1.2 to 1.6]
  A/Aksaray/4048/2016 H6N2 - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Aksaray/4048/2016 H6N2 - Day 90 | 1.8 [1.6 to 2.0] | 2.0 [1.6 to 2.5] | 2.2 [1.9 to 2.6]
  A/Louisiana/13/2017 H6N2 - Day 90: number analyzed (Participants) | 41 | 36 | 38
  A/Louisiana/13/2017 H6N2 - Day 90 | 1.2 [1.0 to 1.3] | 1.3 [1.1 to 1.7] | 1.3 [1.1 to 1.5]
  A/Townsville/51/2016 H6N2 - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Townsville/51/2016 H6N2 - Day 118 | 2.1 [1.7 to 2.7] | 2.0 [1.6 to 2.4] | 2.1 [1.8 to 2.5]
  A/Cameroon/9766/2017 H6N1 - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Cameroon/9766/2017 H6N1 - Day 118 | 1.8 [1.5 to 2.3] | 1.7 [1.3 to 2.1] | 2.0 [1.7 to 2.4]
  A/Hubeiwujiagang/SWL310/2013 - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Hubeiwujiagang/SWL310/2013 - Day 118 | 1.4 [1.1 to 1.7] | 1.6 [1.2 to 2.0] | 1.7 [1.4 to 2.1]
  A/Oman/5532/2017 H6N1 - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Oman/5532/2017 H6N1 - Day 118 | 2.0 [1.6 to 2.5] | 2.0 [1.6 to 2.5] | 2.2 [1.8 to 2.7]
  A/Aksaray/4048/2016 H6N2 - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Aksaray/4048/2016 H6N2 - Day 118 | 2.4 [1.9 to 2.9] | 2.0 [1.6 to 2.6] | 2.4 [1.9 to 3.0]
  A/Louisiana/13/2017 H6N2 - Day 118: number analyzed (Participants) | 36 | 30 | 34
  A/Louisiana/13/2017 H6N2 - Day 118 | 1.5 [1.2 to 1.9] | 1.7 [1.4 to 2.2] | 1.7 [1.4 to 2.1]

57. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Neutralizing (Neut) Titers Against Heterologous H1 and H3 Influenza Strains
Description: Blood was collected for Neut assay which was conducted with the heterologous H1 and H3 influenza viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, but only one result which a geometric mean titer of the replicates was reported by the lab. The geometric mean titer was calculated for each study arm from the available results at Day 1, Day 8, Day 29, Day 57, Day 90, and Day 118 Post first study vaccination.
Time Frame: Day 1, Day 8, Day 29, Day 57, Day 90, Day 118
Population: as for outcome 18
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 41 | 38 | 42
titer
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 1 | 293.5 [177.4 to 485.3] | 535.4 [308.2 to 930.0] | 348.3 [204.3 to 593.9] | 412.1 [240.7 to 705.3] | 388.6 [219.7 to 687.4] | 307.9 [189.9 to 499.4]
  A/Aksaray/4048/2016 [H3N2] - Day 1 | 34.2 [27.9 to 42.0] | 46.7 [34.5 to 63.3] | 40.5 [32.0 to 51.3] | 47.1 [36.3 to 61.2] | 40.3 [32.6 to 49.9] | 40.9 [33.1 to 50.6]
  A/Kenya/105/2017 [H3N2] - Day 1 | 183.2 [135.0 to 248.5] | 294.8 [212.0 to 410.0] | 218.7 [162.1 to 295.1] | 226.8 [171.6 to 299.8] | 232.4 [174.5 to 309.5] | 217.9 [170.6 to 278.3]
  A/Michigan/84/2016 [H3N2] - Day 1 | 858.5 [602.9 to 1222.5] | 852.9 [590.6 to 1231.8] | 616.3 [438.6 to 866.0] | 736.5 [520.1 to 1042.8] | 667.0 [483.7 to 919.9] | 624.2 [455.1 to 856.2]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 8 | 830.8 [534.9 to 1290.4] | 2284.7 [1470.2 to 3550.6] | 1656.1 [1098.6 to 2496.5] | 1212.0 [783.0 to 1876.0] | 1795.8 [1069.5 to 3015.4] | 1425.2 [913.7 to 2222.9]
  A/Aksaray/4048/2016 [H3N2] - Day 8 | 45.4 [33.8 to 61.0] | 101.3 [71.1 to 144.4] | 65.8 [46.4 to 93.2] | 88.2 [64.1 to 121.5] | 121.5 [81.1 to 182.2] | 86.9 [60.8 to 124.0]
  A/Kenya/105/2017 [H3N2] - Day 8 | 267.6 [191.5 to 374.1] | 486.9 [362.5 to 654.0] | 312.8 [231.4 to 422.9] | 431.4 [332.7 to 559.6] | 559.0 [377.8 to 827.1] | 505.9 [384.6 to 665.2]
  A/Michigan/84/2016 [H3N2] - Day 8 | 1237.6 [972.5 to 1574.9] | 1798.5 [1329.9 to 2432.3] | 1088.9 [833.9 to 1421.9] | 1051.7 [802.0 to 1379.2] | 852.0 [591.9 to 1226.5] | 882.3 [652.2 to 1193.5]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 29 | 819.1 [531.4 to 1262.6] | 2083.9 [1428.1 to 3041.0] | 1416.0 [928.8 to 2158.7] | 1940.2 [1267.2 to 2970.8] | 2359.5 [1437.0 to 3874.2] | 1922.4 [1287.1 to 2871.3]
  A/Aksaray/4048/2016 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Aksaray/4048/2016 [H3N2] - Day 29 | 43.3 [35.1 to 53.5] | 70.9 [53.4 to 94.0] | 48.9 [40.2 to 59.6] | 82.0 [63.0 to 106.7] | 107.0 [73.8 to 155.1] | 81.4 [59.0 to 112.4]
  A/Kenya/105/2017 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Kenya/105/2017 [H3N2] - Day 29 | 344.4 [247.5 to 479.3] | 698.1 [498.6 to 977.6] | 421.4 [303.5 to 585.2] | 821.9 [618.7 to 1091.7] | 983.9 [672.0 to 1440.4] | 790.8 [597.1 to 1047.2]
  A/Michigan/84/2016 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Michigan/84/2016 [H3N2] - Day 29 | 1232.8 [936.8 to 1622.3] | 1541.8 [1141.7 to 2082.1] | 1032.4 [782.2 to 1362.6] | 1424.0 [1017.3 to 1993.5] | 1020.1 [669.5 to 1554.2] | 1054.4 [724.7 to 1534.0]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 57 | 396.0 [245.2 to 639.7] | 1000.2 [630.6 to 1586.5] | 720.2 [448.3 to 1157.0] | 1086.0 [692.4 to 1703.1] | 1208.6 [710.9 to 2054.8] | 1032.9 [659.4 to 1618.0]
  A/Aksaray/4048/2016 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Aksaray/4048/2016 [H3N2] - Day 57 | 53.7 [36.9 to 78.0] | 117.6 [83.2 to 166.2] | 61.8 [42.4 to 90.0] | 151.8 [111.0 to 207.6] | 156.5 [110.1 to 222.5] | 140.0 [101.3 to 193.4]
  A/Kenya/105/2017 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Kenya/105/2017 [H3N2] - Day 57 | 237.7 [168.6 to 335.2] | 469.4 [338.5 to 650.9] | 283.7 [187.6 to 429.0] | 634.0 [467.3 to 860.1] | 688.0 [478.2 to 989.7] | 517.7 [364.7 to 735.1]
  A/Michigan/84/2016 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Michigan/84/2016 [H3N2] - Day 57 | 1071.2 [844.9 to 1358.2] | 1602.1 [1174.2 to 2186.0] | 946.6 [701.5 to 1277.2] | 1533.4 [1127.0 to 2086.4] | 904.9 [631.5 to 1296.8] | 1158.3 [829.3 to 1617.9]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 90 | 556.7 [338.1 to 916.8] | 1501.0 [927.7 to 2316.6] | 946.6 [567.5 to 1579.1] | 1331.6 [812.5 to 2182.4] | 1563.9 [898.7 to 2721.5] | 1268.5 [799.6 to 2012.6]
  A/Aksaray/4048/2016 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Aksaray/4048/2016 [H3N2] - Day 90 | 62.4 [41.3 to 94.2] | 111.0 [77.1 to 159.6] | 64.7 [44.7 to 93.6] | 149.1 [110.6 to 201.0] | 147.2 [104.2 to 208.0] | 129.6 [91.8 to 183.1]
  A/Kenya/105/2017 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Kenya/105/2017 [H3N2] - Day 90 | 151.6 [107.9 to 212.9] | 315.4 [220.1 to 452.1] | 200.1 [130.8 to 306.1] | 431.5 [300.0 to 620.7] | 444.3 [297.7 to 663.0] | 385.5 [270.5 to 549.4]
  A/Michigan/84/2016 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Michigan/84/2016 [H3N2] - Day 90 | 841.2 [627.1 to 1128.5] | 1268.8 [907.6 to 1773.7] | 778.8 [576.1 to 1052.8] | 1297.0 [905.5 to 1857.7] | 733.5 [488.2 to 1102.1] | 905.2 [611.5 to 1340.1]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 118 | 1128.1 [631.8 to 2014.4] | 1723.8 [1046.1 to 2840.8] | 1631.8 [995.5 to 2674.9] | 2739.4 [1472.3 to 5096.9] | 3672.3 [2051.3 to 6574.1] | 2233.2 [1295.2 to 3850.4]
  A/Aksaray/4048/2016 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Aksaray/4048/2016 [H3N2] - Day 118 | 94.6 [66.8 to 134.1] | 139.0 [89.9 to 215.1] | 150.1 [103.6 to 217.3] | 326.1 [213.5 to 498.3] | 296.5 [200.9 to 437.6] | 241.3 [149.0 to 390.9]
  A/Kenya/105/2017 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Kenya/105/2017 [H3N2] - Day 118 | 300.7 [210.5 to 429.5] | 400.6 [253.2 to 633.8] | 369.1 [235.3 to 538.0] | 936.6 [636.7 to 1377.7] | 965.5 [623.9 to 1494.3] | 733.9 [478.8 to 1125.0]
  A/Michigan/84/2016 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Michigan/84/2016 [H3N2] - Day 118 | 1382.3 [1083.1 to 1764.2] | 1785.2 [1201.1 to 2653.4] | 1487.2 [1108.4 to 1996.6] | 2572.0 [1842.0 to 3591.3] | 1537.3 [1005.4 to 2350.7] | 1641.9 [1095.4 to 2461.0]

58. Secondary Outcome: Ratio of Serum Neutralizing (Neut) Geometric Mean Titers (GMT) Against Heterologous H1 and H3 Influenza Strains Between Adjuvanted and Unadjuvanted Study Arms
Description: Blood was collected for Neut assay which was conducted with the heterologous H1 and H3 influenza viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, but only one result which a geometric mean titer of the replicates was reported by the lab. The geometric mean titer was calculated for each study arm from the available results at Day 1, Day 8, Day 29, Day 57, Day 90, and Day 118 Post first study vaccination and the ratio of these GMTs between adjuvanted and unadjuvanted study arms were calculated.
  Unadjuvanted Fluzone and Flublok study arms are considered as reference groups for the analysis of ratio of GMTs.
  Ratio of GMTs is defined as the ratio of the GMT from the adjuvanted group divided by the GMT from the corresponding unadjuvanted group.
Time Frame: Day 1, Day 8, Day 29, Day 57, Day 90, Day 118
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: ratio of GMT
Arm/Group | Fluzone + AF03 | Fluzone + CpG55 | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 37 | 40 | 38 | 42
ratio of GMT
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 1 | 1.8 [0.9 to 3.8] | 1.2 [0.6 to 2.4] | 0.9 [0.4 to 2.0] | 0.7 [0.4 to 1.5]
  A/Aksaray/4048/2016 [H3N2] - Day 1 | 1.4 [1.0 to 2.0] | 1.2 [0.9 to 1.6] | 0.9 [0.6 to 1.2] | 0.9 [0.6 to 1.2]
  A/Kenya/105/2017 [H3N2] - Day 1 | 1.6 [1.0 to 2.5] | 1.2 [0.8 to 1.8] | 1.0 [0.7 to 1.5] | 1.0 [0.7 to 1.4]
  A/Michigan/84/2016 [H3N2] - Day 1 | 1.0 [0.6 to 1.6] | 0.7 [0.4 to 1.2] | 0.9 [0.6 to 1.4] | 0.8 [0.5 to 1.3]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 8 | 2.7 [1.5 to 5.1] | 2.0 [1.1 to 3.6] | 1.5 [0.8 to 2.9] | 1.2 [0.6 to 2.2]
  A/Aksaray/4048/2016 [H3N2] - Day 8 | 2.2 [1.4 to 3.5] | 1.4 [0.9 to 2.3] | 1.4 [0.8 to 2.3] | 1.0 [0.6 to 1.6]
  A/Kenya/105/2017 [H3N2] - Day 8 | 1.8 [1.2 to 2.8] | 1.2 [0.8 to 1.8] | 1.3 [0.8 to 2.1] | 1.2 [0.8 to 1.7]
  A/Michigan/84/2016 [H3N2] - Day 8 | 1.5 [1.0 to 2.1] | 0.9 [0.6 to 1.3] | 0.8 [0.5 to 1.3] | 0.8 [0.6 to 1.3]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 29: number analyzed (Participants) | 36 | 39 | 37 | 41
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 29 | 2.5 [1.4 to 4.5] | 1.7 [1.0 to 3.1] | 1.2 [0.6 to 2.3] | 1.0 [0.6 to 1.8]
  A/Aksaray/4048/2016 [H3N2] - Day 29: number analyzed (Participants) | 36 | 39 | 37 | 41
  A/Aksaray/4048/2016 [H3N2] - Day 29 | 1.6 [1.2 to 2.3] | 1.1 [0.8 to 1.5] | 1.3 [0.8 to 2.0] | 1.0 [0.7 to 1.5]
  A/Kenya/105/2017 [H3N2] - Day 29: number analyzed (Participants) | 36 | 39 | 37 | 41
  A/Kenya/105/2017 [H3N2] - Day 29 | 2.0 [1.3 to 3.2] | 1.2 [0.8 to 1.9] | 1.2 [0.7 to 1.9] | 1.0 [0.6 to 1.4]
  A/Michigan/84/2016 [H3N2] - Day 29: number analyzed (Participants) | 36 | 39 | 37 | 41
  A/Michigan/84/2016 [H3N2] - Day 29 | 1.3 [0.8 to 1.9] | 0.8 [0.6 to 1.2] | 0.7 [0.4 to 1.2] | 0.7 [0.5 to 1.2]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 57: number analyzed (Participants) | 37 | 38 | 37 | 41
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 57 | 2.5 [1.3 to 4.9] | 1.8 [0.9 to 3.5] | 1.1 [0.6 to 2.2] | 1.0 [0.5 to 1.8]
  A/Aksaray/4048/2016 [H3N2] - Day 57: number analyzed (Participants) | 37 | 38 | 37 | 41
  A/Aksaray/4048/2016 [H3N2] - Day 57 | 2.2 [1.3 to 3.6] | 1.2 [0.7 to 1.9] | 1.0 [0.6 to 1.6] | 0.9 [0.6 to 1.4]
  A/Kenya/105/2017 [H3N2] - Day 57: number analyzed (Participants) | 37 | 38 | 37 | 41
  A/Kenya/105/2017 [H3N2] - Day 57 | 2.0 [1.2 to 3.1] | 1.2 [0.7 to 2.0] | 1.1 [0.7 to 1.7] | 0.8 [0.5 to 1.3]
  A/Michigan/84/2016 [H3N2] - Day 57: number analyzed (Participants) | 37 | 38 | 37 | 41
  A/Michigan/84/2016 [H3N2] - Day 57 | 1.5 [1.0 to 2.2] | 0.9 [0.6 to 1.3] | 0.6 [0.4 to 0.9] | 0.8 [0.5 to 1.2]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 90: number analyzed (Participants) | 36 | 38 | 37 | 40
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 90 | 2.7 [1.4 to 5.2] | 1.7 [0.8 to 3.4] | 1.2 [0.6 to 2.4] | 1.0 [0.5 to 1.9]
  A/Aksaray/4048/2016 [H3N2] - Day 90: number analyzed (Participants) | 36 | 38 | 37 | 40
  A/Aksaray/4048/2016 [H3N2] - Day 90 | 1.8 [1.0 to 3.1] | 1.0 [0.6 to 1.8] | 1.0 [0.6 to 1.5] | 0.9 [0.6 to 1.4]
  A/Kenya/105/2017 [H3N2] - Day 90: number analyzed (Participants) | 36 | 38 | 37 | 40
  A/Kenya/105/2017 [H3N2] - Day 90 | 2.1 [1.3 to 3.4] | 1.3 [0.8 to 2.3] | 1.0 [0.6 to 1.8] | 0.9 [0.5 to 1.5]
  A/Michigan/84/2016 [H3N2] - Day 90: number analyzed (Participants) | 36 | 38 | 37 | 40
  A/Michigan/84/2016 [H3N2] - Day 90 | 1.5 [1.0 to 2.3] | 0.9 [0.6 to 1.4] | 0.6 [0.3 to 1.0] | 0.7 [0.4 to 1.2]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 118: number analyzed (Participants) | 30 | 34 | 32 | 34
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 118 | 1.5 [0.7 to 3.2] | 1.4 [0.7 to 3.1] | 1.3 [0.6 to 3.1] | 0.8 [0.4 to 1.8]
  A/Aksaray/4048/2016 [H3N2] - Day 118: number analyzed (Participants) | 30 | 34 | 32 | 34
  A/Aksaray/4048/2016 [H3N2] - Day 118 | 1.5 [0.8 to 2.5] | 1.6 [1.0 to 2.6] | 0.9 [0.5 to 1.6] | 0.7 [0.4 to 1.4]
  A/Kenya/105/2017 [H3N2] - Day 118: number analyzed (Participants) | 30 | 34 | 32 | 34
  A/Kenya/105/2017 [H3N2] - Day 118 | 1.3 [0.8 to 2.4] | 1.2 [0.7 to 2.0] | 1.0 [0.6 to 1.8] | 0.8 [0.4 to 1.4]
  A/Michigan/84/2016 [H3N2] - Day 118: number analyzed (Participants) | 30 | 34 | 32 | 34
  A/Michigan/84/2016 [H3N2] - Day 118 | 1.3 [0.8 to 2.0] | 1.1 [0.7 to 1.6] | 0.6 [0.4 to 1.0] | 0.6 [0.4 to 1.1]

59. Secondary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Titer Seroconversion Against Heterologous H1 and H3 Influenza Strains
Description: Blood was collected for Neut assay which was conducted with the heterologous H1 and H3 influenza viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, but only one result which a geometric mean titer of the replicates was reported by the lab. Neut seroconversion was defined as either a pre-vaccination titer < 1:10 and a post-vaccination titer >= 1:40 or a pre-vaccination titer >= 1:10 and a minimum four-fold rise in post-vaccination antibody titer.
Time Frame: Day 8, Day 29, Day 57, Day 90, Day 118
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 41 | 38 | 42
percentage of participants
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 8 | 24 [12 to 40] | 32 [18 to 50] | 33 [19 to 49] | 27 [14 to 43] | 42 [26 to 59] | 45 [30 to 61]
  A/Aksaray/4048/2016 [H3N2] - Day 8 | 7 [2 to 20] | 16 [6 to 32] | 13 [4 to 27] | 20 [9 to 35] | 34 [20 to 51] | 21 [10 to 37]
  A/Kenya/105/2017 [H3N2] - Day 8 | 12 [4 to 26] | 16 [6 to 32] | 15 [6 to 30] | 15 [6 to 29] | 24 [11 to 40] | 24 [12 to 39]
  A/Michigan/84/2016 [H3N2] - Day 8 | 12 [4 to 26] | 19 [8 to 35] | 13 [4 to 27] | 10 [3 to 23] | 8 [2 to 21] | 12 [4 to 26]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 29 | 34 [20 to 51] | 33 [19 to 51] | 31 [17 to 48] | 55 [38 to 71] | 51 [34 to 68] | 49 [33 to 65]
  A/Aksaray/4048/2016 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Aksaray/4048/2016 [H3N2] - Day 29 | 7 [2 to 20] | 11 [3 to 26] | 5 [NA to 17] — Value is NA because it's >0 but <1 | 10 [3 to 24] | 24 [12 to 41] | 17 [7 to 32]
  A/Kenya/105/2017 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Kenya/105/2017 [H3N2] - Day 29 | 15 [6 to 29] | 22 [10 to 39] | 21 [9 to 36] | 35 [21 to 52] | 43 [27 to 61] | 39 [24 to 55]
  A/Michigan/84/2016 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Michigan/84/2016 [H3N2] - Day 29 | 12 [4 to 26] | 17 [6 to 33] | 10 [3 to 24] | 15 [6 to 30] | 11 [3 to 25] | 12 [4 to 26]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 57: number analyzed (Participants) | 41 | 37 | 38 | 40 | 37 | 41
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 57 | 15 [6 to 30] | 16 [6 to 32] | 26 [13 to 43] | 33 [19 to 49] | 35 [20 to 53] | 32 [18 to 48]
  A/Aksaray/4048/2016 [H3N2] - Day 57: number analyzed (Participants) | 41 | 37 | 38 | 40 | 37 | 41
  A/Aksaray/4048/2016 [H3N2] - Day 57 | 13 [4 to 27] | 14 [5 to 29] | 11 [3 to 25] | 38 [23 to 54] | 49 [32 to 66] | 37 [22 to 53]
  A/Kenya/105/2017 [H3N2] - Day 57: number analyzed (Participants) | 41 | 37 | 38 | 40 | 37 | 41
  A/Kenya/105/2017 [H3N2] - Day 57 | 8 [2 to 20] | 19 [8 to 35] | 16 [6 to 31] | 30 [17 to 47] | 32 [18 to 50] | 29 [16 to 46]
  A/Michigan/84/2016 [H3N2] - Day 57: number analyzed (Participants) | 41 | 37 | 38 | 40 | 37 | 42
  A/Michigan/84/2016 [H3N2] - Day 57 | 13 [4 to 27] | 16 [6 to 32] | 3 [NA to 14] — Value is NA because it's >0 but <1 | 13 [4 to 27] | 8 [2 to 22] | 12 [4 to 26]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 90 | 20 [9 to 35] | 25 [12 to 42] | 24 [11 to 40] | 33 [19 to 50] | 41 [25 to 58] | 40 [25 to 57]
  A/Aksaray/4048/2016 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Aksaray/4048/2016 [H3N2] - Day 90 | 17 [7 to 32] | 17 [6 to 33] | 11 [3 to 25] | 33 [19 to 50] | 49 [32 to 66] | 30 [17 to 47]
  A/Kenya/105/2017 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Kenya/105/2017 [H3N2] - Day 90 | 5 [NA to 17] — Value is NA because it's >0 but <1 | 8 [2 to 22] | 8 [2 to 21] | 18 [8 to 34] | 22 [10 to 38] | 18 [7 to 33]
  A/Michigan/84/2016 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Michigan/84/2016 [H3N2] - Day 90 | 0 [0 to 9] | 8 [2 to 22] | 3 [NA to 14] — Value is NA because it's >0 but <1 | 10 [3 to 24] | 8 [2 to 22] | 8 [2 to 20]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 118 | 47 [30 to 65] | 33 [17 to 53] | 44 [27 to 62] | 56 [38 to 73] | 72 [53 to 86] | 68 [49 to 83]
  A/Aksaray/4048/2016 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Aksaray/4048/2016 [H3N2] - Day 118 | 33 [19 to 51] | 27 [12 to 46] | 35 [20 to 54] | 79 [62 to 91] | 69 [50 to 84] | 62 [44 to 78]
  A/Kenya/105/2017 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Kenya/105/2017 [H3N2] - Day 118 | 19 [8 to 36] | 10 [2 to 27] | 21 [9 to 38] | 44 [27 to 62] | 44 [26 to 62] | 38 [22 to 56]
  A/Michigan/84/2016 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Michigan/84/2016 [H3N2] - Day 118 | 19 [8 to 36] | 17 [6 to 35] | 18 [7 to 35] | 32 [17 to 51] | 22 [9 to 40] | 35 [20 to 54]

60. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in Neutralizing (Neut) Titers Against Heterologous H1 and H3 Influenza Strains
Description: Blood was collected for Neut assay which was conducted with the heterologous H1 and H3 influenza viruses as the antigens. Each sample was tested twice per antigen per the laboratory's standard operating procedure, but only one result which a geometric mean titer of the replicates was reported by the lab. Fold-rises from baseline were calculated as the Day 8 (or Day 29, Day 57, Day 90, Day 118) titer divided by the baseline titers for each participant. The geometric mean of these fold rises was then calculated to obtain the GMFR.
Time Frame: Day 8, Day 29, Day 57, Day 90, Day 118
Population: as for outcome 18
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
Number analyzed (Participants) | 41 | 37 | 40 | 41 | 38 | 42
fold rise
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 8 | 2.8 [1.8 to 4.4] | 4.3 [2.6 to 7.0] | 4.8 [2.9 to 7.7] | 2.9 [2.0 to 4.3] | 4.6 [2.8 to 7.7] | 4.6 [2.8 to 7.7]
  A/Aksaray/4048/2016 [H3N2] - Day 8 | 1.3 [1.0 to 1.7] | 2.2 [1.6 to 3.0] | 1.6 [1.2 to 2.2] | 1.9 [1.4 to 2.5] | 3.0 [2.1 to 4.3] | 2.1 [1.5 to 3.0]
  A/Kenya/105/2017 [H3N2] - Day 8 | 1.5 [1.1 to 2.0] | 1.7 [1.2 to 2.3] | 1.4 [1.1 to 1.9] | 1.9 [1.5 to 2.5] | 2.4 [1.7 to 3.5] | 2.3 [1.7 to 3.1]
  A/Michigan/84/2016 [H3N2] - Day 8 | 1.4 [1.1 to 1.9] | 2.1 [1.5 to 2.9] | 1.8 [1.3 to 2.3] | 1.4 [1.2 to 1.8] | 1.3 [1.0 to 1.7] | 1.4 [1.1 to 1.8]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 29 | 2.8 [1.8 to 4.3] | 3.4 [2.1 to 5.5] | 4.3 [2.6 to 7.1] | 4.7 [3.1 to 7.2] | 5.5 [3.5 to 8.5] | 5.9 [3.6 to 9.7]
  A/Aksaray/4048/2016 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Aksaray/4048/2016 [H3N2] - Day 29 | 1.3 [1.0 to 1.5] | 1.5 [1.1 to 2.0] | 1.2 [1.0 to 1.5] | 1.7 [1.3 to 2.3] | 2.6 [1.8 to 3.7] | 2.0 [1.4 to 2.8]
  A/Kenya/105/2017 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Kenya/105/2017 [H3N2] - Day 29 | 1.9 [1.4 to 2.5] | 2.3 [1.6 to 3.2] | 1.9 [1.4 to 2.7] | 3.6 [2.6 to 4.8] | 4.1 [2.9 to 5.8] | 3.5 [2.6 to 4.8]
  A/Michigan/84/2016 [H3N2] - Day 29: number analyzed (Participants) | 41 | 36 | 39 | 40 | 37 | 41
  A/Michigan/84/2016 [H3N2] - Day 29 | 1.4 [1.1 to 1.8] | 1.8 [1.3 to 2.3] | 1.6 [1.4 to 1.9] | 1.9 [1.4 to 2.5] | 1.5 [1.2 to 1.9] | 1.7 [1.3 to 2.2]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 57 | 1.4 [0.9 to 2.1] | 1.9 [1.2 to 2.9] | 2.3 [1.4 to 3.6] | 2.6 [1.8 to 3.9] | 3.0 [1.9 to 4.7] | 3.2 [2.0 to 5.2]
  A/Aksaray/4048/2016 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Aksaray/4048/2016 [H3N2] - Day 57 | 1.6 [1.2 to 2.1] | 2.5 [1.9 to 3.4] | 1.6 [1.2 to 2.1] | 3.2 [2.4 to 4.2] | 3.8 [2.7 to 5.2] | 3.4 [2.4 to 4.7]
  A/Kenya/105/2017 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Kenya/105/2017 [H3N2] - Day 57 | 1.3 [1.0 to 1.8] | 1.6 [1.1 to 2.3] | 1.3 [0.9 to 1.9] | 2.7 [2.0 to 3.7] | 2.9 [2.2 to 3.9] | 2.3 [1.6 to 3.3]
  A/Michigan/84/2016 [H3N2] - Day 57: number analyzed (Participants) | 40 | 37 | 38 | 40 | 37 | 41
  A/Michigan/84/2016 [H3N2] - Day 57 | 1.3 [1.0 to 1.6] | 1.9 [1.4 to 2.5] | 1.5 [1.3 to 1.8] | 2.0 [1.5 to 2.6] | 1.4 [1.1 to 1.7] | 1.8 [1.4 to 2.4]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 90 | 1.9 [1.3 to 2.7] | 2.5 [1.5 to 4.0] | 3.0 [2.0 to 4.6] | 3.3 [2.3 to 4.8] | 3.8 [2.4 to 6.0] | 3.8 [2.4 to 6.1]
  A/Aksaray/4048/2016 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Aksaray/4048/2016 [H3N2] - Day 90 | 1.8 [1.3 to 2.5] | 2.3 [1.8 to 3.0] | 1.6 [1.3 to 2.1] | 3.1 [2.4 to 4.1] | 3.5 [2.6 to 4.8] | 3.1 [2.3 to 4.3]
  A/Kenya/105/2017 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Kenya/105/2017 [H3N2] - Day 90 | 0.8 [0.6 to 1.1] | 1.0 [0.7 to 1.4] | 0.9 [0.7 to 1.3] | 1.9 [1.4 to 2.6] | 1.9 [1.3 to 2.7] | 1.7 [1.3 to 2.3]
  A/Michigan/84/2016 [H3N2] - Day 90: number analyzed (Participants) | 41 | 36 | 38 | 39 | 37 | 40
  A/Michigan/84/2016 [H3N2] - Day 90 | 1.0 [0.8 to 1.2] | 1.5 [1.1 to 1.9] | 1.3 [1.0 to 1.5] | 1.7 [1.3 to 2.2] | 1.1 [0.8 to 1.4] | 1.4 [1.1 to 1.9]
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Shandonglaicheng/1763/2016 [H3N2] - Day 118 | 4.6 [2.9 to 7.3] | 2.8 [1.8 to 4.3] | 5.7 [3.5 to 9.4] | 6.8 [4.2 to 11.0] | 9.9 [5.8 to 16.8] | 7.8 [4.7 to 12.8]
  A/Aksaray/4048/2016 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Aksaray/4048/2016 [H3N2] - Day 118 | 3.0 [2.2 to 4.1] | 2.9 [2.0 to 4.1] | 3.7 [2.6 to 5.3] | 6.9 [4.8 to 9.9] | 7.3 [5.0 to 10.6] | 6.1 [4.0 to 9.5]
  A/Kenya/105/2017 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Kenya/105/2017 [H3N2] - Day 118 | 1.8 [1.3 to 2.6] | 1.2 [0.9 to 1.7] | 1.8 [1.3 to 2.4] | 4.2 [3.0 to 6.0] | 4.2 [2.9 to 6.2] | 3.5 [2.5 to 4.9]
  A/Michigan/84/2016 [H3N2] - Day 118: number analyzed (Participants) | 36 | 30 | 34 | 34 | 32 | 34
  A/Michigan/84/2016 [H3N2] - Day 118 | 1.7 [1.3 to 2.3] | 1.8 [1.4 to 2.3] | 2.4 [1.9 to 3.0] | 3.2 [2.3 to 4.3] | 2.3 [1.7 to 3.1] | 2.6 [1.9 to 3.7]

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs), AESIs (including protocol-specified AESIs, MAAEs, NOCMCs and PIMMCs) were collected from the time of first study vaccination through approximately 12 months following first study vaccination. Solicited Adverse Events (AEs) and clinical safety laboratory AEs were collected from the time of first study vaccination through Day 7. Non-serious, unsolicited AEs were collected from the time of first study vaccination through approximately Day 29.
Description: Solicited AEs include injection site reactions and systemic reactions. Injection site reactions include pruritus, ecchymosis, erythema, induration, edema, pain, and tenderness. Systemic reactions include fever, feverishness, fatigue, malaise, myalgia, arthralgia, headache, and nausea.
Arm/Group | Fluzone | Fluzone + AF03 | Fluzone + CpG55 | Flublok | Flublok + AF03 | Flublok + CpG55
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/37 | 0/40 | 0/42 | 0/37 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/41 | 1/37 | 0/40 | 0/42 | 0/37 | 1/43
Other Adverse Events (participants affected / at risk) | 37/41 | 36/37 | 40/40 | 36/42 | 34/37 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluzone (N=41) | Fluzone + AF03 (N=37) | Fluzone + CpG55 (N=40) | Flublok (N=42) | Flublok + AF03 (N=37) | Flublok + CpG55 (N=43)
Chronic Left Knee Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium Difficile Colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluzone (N=41) | Fluzone + AF03 (N=37) | Fluzone + CpG55 (N=40) | Flublok (N=42) | Flublok + AF03 (N=37) | Flublok + CpG55 (N=43)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (3) | 5 (5) | 5 (5) | 6 (6)
Fatigue (General disorders) | 13 (13) | 16 (16) | 14 (14) | 13 (13) | 14 (14) | 15 (15)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 9 (9) | 11 (11) | 8 (8) | 6 (6) | 8 (8) | 5 (5)
Pyrexia (General disorders) | 3 (3) | 4 (4) | 6 (6) | 5 (5) | 5 (5) | 4 (4)
Vaccination site bruising (General disorders) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 4 (4)
Vaccination site erythema (General disorders) | 8 (8) | 9 (9) | 16 (16) | 6 (6) | 7 (7) | 12 (12)
Vaccination site induration (General disorders) | 12 (12) | 4 (4) | 13 (13) | 6 (6) | 6 (6) | 13 (13)
Vaccination site pain (General disorders) | 12 (12) | 22 (22) | 26 (26) | 7 (7) | 21 (21) | 27 (27)
Vaccination site pain (tenderness) (General disorders) | 29 (29) | 35 (35) | 38 (38) | 30 (30) | 30 (30) | 41 (41)
Vaccination site pruritus (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (2)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1) | 2 (3) | 4 (6) | 0 (0) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (8) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 6 (6) | 3 (3) | 3 (3) | 2 (2) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (11) | 15 (15) | 12 (12) | 6 (6) | 9 (9) | 11 (11)
Headache (Nervous system disorders) | 11 (12) | 21 (21) | 10 (10) | 13 (13) | 11 (11) | 10 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT03945825/Prot_001.pdf
  • Statistical Analysis Plan (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/25/NCT03945825/SAP_002.pdf
  • Informed Consent Form (2019-06-04): https://cdn.clinicaltrials.gov/large-docs/25/NCT03945825/ICF_000.pdf